

## The world's childhood cancer experts



October 28, 2022

# PPD

**RE:** Request for Amendments with FDA requested language for Pediatric MATCH consents

Dear PPD

The study committee thanks CTEP for forwarding the Amendment Request dated October 17, 2022. In response to the request, please see attached Amendment #6 to APEC1621D. The complete list of changes can be found below.

Please contact us if you have any further questions.

Sincerely,





#### **SUMMARY OF CHANGES: PROTOCOL**

In accordance with the above discussion, the following specific revisions have been made to the protocol.

Additions are in boldfaced font and deletions in strikethrough font.

| # | Section | Page(s) | Change |
|---|---|---|---|
| 1. | General | - | Updated protocol version date in the footer. |
| 2. | Cover Page | 1 | Updated version date and amendment number. |
| 3. | Contact<br>Information | 2 | Cancer Trials Support Unit (CTSU)information updated with email address CTSURegHelp@coccg.org |
| 4. | <u>Table of</u><br><u>Contents</u> | 3-5 | Updated for re-pagination. |
| 5. | Study Committee | 7 | Deleted PPD and added PPD as Protocol Coordinator |

ii



CHILDREN'S

**ONCOLOGY** 

GROUP

ncer experts APEC1621D

Activated: July 31, 2017 Version Date: 10/28/2022

Closed: Amendment: 6

#### **CHILDREN'S ONCOLOGY GROUP**

#### APEC1621D

## NCI-COG PEDIATRIC MATCH (MOLECULAR ANALYSIS FOR THERAPY CHOICE)PHASE 2 SUBPROTOCOL OF LY3023414 IN PATIENTS WITH SOLID TUMORS

#### Open to COG Member Institutions in the USA

THIS PROTOCOL IS FOR RESEARCH PURPOSES ONLY, AND SHOULD NOT BE COPIED, REDISTRIBUTED OR USED FOR ANY OTHER PURPOSE. MEDICAL AND SCIENTIFIC INFORMATION CONTAINED WITHIN THIS PROTOCOL IS NOT INCLUDED TO AUTHORIZE OR FACILITATE THE PRACTICE OF MEDICINE BY ANY PERSON OR ENTITY. RESEARCH MEANS A SYSTEMATIC INVESTIGATION, INCLUDING RESEARCH DEVELOPMENT, TESTING AND EVALUATION, DESIGNED TO DEVELOP OR CONTRIBUTE TO GENERALIZABLE KNOWLEDGE. THIS PROTOCOL IS THE RESEARCH PLAN DEVELOPED BY THE CHILDREN'S ONCOLOGY GROUP TO INVESTIGATE A PARTICULAR STUDY QUESTION OR SET OF STUDY QUESTIONS AND SHOULD NOT BE USED TO DIRECT THE PRACTICE OF MEDICINE BY ANY PERSON OR TO PROVIDE INDIVIDUALIZED MEDICAL CARE, TREATMENT, OR ADVICE TO ANY PATIENT OR STUDY SUBJECT. THE PROCEDURES IN THIS PROTOCOL ARE INTENDED ONLY FOR USE BY CLINICAL ONCOLOGISTS IN CAREFULLY STRUCTURED SETTINGS, AND MAY NOT PROVE TO BE MORE EFFECTIVE THAN STANDARD TREATMENT. ANY PERSON WHO REQUIRES MEDICAL CARE IS URGED TO CONSULT WITH HIS OR HER PERSONAL PHYSICIAN OR TREATING PHYSICIAN OR VISIT THE NEAREST LOCAL HOSPITAL OR HEALTHCARE INSTITUTION.





| CONTACT INFORMATION | | |
|---|---|---|
| For Regulatory Requirements | For patient enrollments: | For Data Submission |
| Regulatory documentation must be submitted to the Cancer Trials Support Unit (CTSU) via the Regulatory Submission Portal. (Sign in at <a href="https://www.ctsu.org">www.ctsu.org</a> , and select the Regulatory > Regulatory Submission.) Institutions with patients waiting that are unable to use the Portal should alert the CTSU Regulatory Office immediately by phone or email: 1-866-651-CTSU (2878), or <a href="https://creativecommons.org/ctsuregHelp@coccg.org">CTSURegHelp@coccg.org</a> to receive further instruction and support. Contact the CTSU Regulatory Help | Please refer to the patient enrollment section of the protocol for instructions on using the Oncology Patient Enrollment Network (OPEN). OPEN is accessed at <a href="https://www.ctsu.org/OPEN_SYSTEM/">https://www.ctsu.org/OPEN_SYSTEM/</a> or <a href="https://open.ctsu.org">https://open.ctsu.org</a> . Contact the CTSU Help Desk with any OPEN-related questions by phone or email: 1-888-823-5923, or <a href="mailto:ctsucontact@westat.com">ctsucontact@westat.com</a> . | Data collection for this study will be done exclusively through Medidata Rave. Please see the Data Submission Schedule in the CRF packet for further instructions. |
| should alert the CTSU Regulatory Office immediately by phone or email: 1-866-651-CTSU (2878), or CTSURegHelp@coccg.org to receive further instruction and | | |

The most current version of the **study protocol** must be downloaded from the protocol-specific page located on the CTSU members' website (<a href="https://www.ctsu.org">https://www.ctsu.org</a>). Access to the CTSU members' website is managed through the Cancer Therapy and Evaluation Program - Identity and Access Management (CTEP-IAM) registration system and requires log in with a CTEP-IAM username and password. Permission to view and download this protocol and its supporting documents is restricted and is based on person and site roster assignment housed in the CTSU Regulatory Support System (RSS).

#### For clinical questions (ie, patient eligibility or treatment-related)

Contact the Study PI of the Lead Protocol Organization.

#### For non-clinical questions (ie, unrelated to patient eligibility, treatment, or clinical data submission)

Contact the CTSU Help Desk by phone or e-mail:

CTSU General Information Line -1-888-823-5923, or <u>ctsucontact@westat.com</u>. All calls and correspondence will be triaged to the appropriate CTSU representative.

The CTSU Website is located at https://www.ctsu.org.



#### TABLE OF CONTENTS

| SECTIO | <u>N</u> | <u>PAGE</u> |
|---|---|---|
| CHILDRI | EN'S ONCOLOGY GROUP | 1 |
| TABLE C | OF CONTENTS | 3 |
| STUDY ( | COMMITTEE | 6 |
| STUDY O | COMMITTEE, CONT. | 7 |
| ABSTRA | CT | 8 |
| EXPERIN | MENTAL DESIGN SCHEMA | 8 |
| 1. | 2 Secondary Aims | 9<br>9<br>9<br>9 |
| 2.<br>2.<br>2. | <ul> <li>2 Preclinical Studies</li> <li>3 Adult Studies</li> <li>4 Pediatric Studies</li> </ul> | 10<br>10<br>10<br>13<br>15<br>17 |
| 3.0 So 3. | <ul> <li>Informed Consent/Assent</li> <li>Screening Procedures</li> <li>Eligibility Checklist</li> <li>Study Enrollment</li> <li>Institutional Pathology Report</li> </ul> | 19<br>19<br>22<br>22<br>22<br>22<br>22<br>22 |
| 4.0 P. 4. 4. 4. | | 23<br>23<br>27 |
| 5.0 T<br>5.<br>5.<br>5. | <ul><li>2 Criteria for Starting Subsequent Cycles</li><li>3 Grading of Adverse Events</li></ul> | 28<br>28<br>30<br>30<br>30 |
| 6.0 D<br>6. | | 32<br>32<br>32 |
| 7.0 Si 7. 7. 7. 7. 7. | <ul><li>Investigational Agents</li><li>Supportive Care</li></ul> | 33<br>33<br>33<br>33<br>35 |



| CHILDREN'S |
|------------|
| ONCOLOGY |
| GROUP |

| | 7.5 | Concomitant Medications | 35 |
|---|---|---|---|
| 8.0 | EVAL | UATIONS/MATERIAL AND DATA TO BE ACCESSIONED | 36 |
| | 8.1 | Required Clinical, Laboratory and Disease Evaluation | 36 |
| | 8.2 | Radiology Studies | 37 |
| | 8.3 | Pharmacology (optional) | 38 |
| | 8.4 | Circulating Tumor DNA Study (optional) | 39 |
| 9.0 | AGEN | NT INFORMATION | 41 |
| | 9.1 | LY3023414 | 41 |
| | 9.2 | Agent Ordering and Agent Accountability | 45 |
| | 9.3 | Clinical Drug Request and Investigator Brochure Availability | 45 |
| | 9.4 | Agent Inventory Records | 45 |
| 10.0 | CRITI | CRITERIA FOR REMOVAL FROM PROTOCOL THERAPY AND OFF STUDY CRITERIA | |
| | 10.1 | Criteria for Removal from Protocol Therapy | 46<br>46 |
| | 10.1 | Follow-Up Data Submission and APEC1621SC Off Study Criteria | 46 |
| | | • | |
| 11.0 | | ISTICAL AND ETHICAL CONSIDERATIONS | 47 |
| | 11.1 | Sample Size and Study Duration | 47 |
| | 11.2 | Dosing Considerations | 47 |
| | 11.3 | Study Design | 48 |
| | 11.4<br>11.5 | Methods of Analysis Evaluability for Response | 51<br>51 |
| | 11.5 | Evaluability for Toxicity | 51 |
| | 11.7 | Progression free survival (PFS) | 51 |
| | 11.8 | Correlative Studies | 52 |
| | 11.9 | Gender and Minority Accrual Estimates | 52 |
| 12.0 | EVAL | UATION CRITERIA | 53 |
| | 12.1 | Common Terminology Criteria for Adverse Events (CTCAE) | 53 |
| | 12.2 | Progression-Free Survival | 53 |
| | 12.3 | Response Criteria for Patients with Solid Tumors | 53 |
| | 12.4 | Response Criteria for Patients with Solid Tumor and Measurable Disease | 56 |
| | 12.5 | Response Criteria for Neuroblastoma Patients with MIBG Positive Lesions | 59 |
| | 12.6 | Response Criteria for Neuroblastoma Patients with Bone Marrow Involvement | 61 |
| | 12.7 | Response Criteria for Patients with CNS Tumors | 61 |
| | 12.8 | Response Criteria for Patients with non-Hodgkin Lymphoma/Histiocytosis | 63 |
| | 12.9 | Best Response | 65 |
| 13.0 | | ERSE EVENT REPORTING REQUIREMENTS | 67 |
| | 13.1 | Expedited Reporting Requirements – Serious Adverse Events (SAEs) | 67 |
| | 13.2 | Steps to Determine If an Adverse Event Is To Be Reported In an Expedited Manner | 68 |
| | 13.3 | Exceptions to CTEP-AERS Expedited Reporting Requirements: | 70 |
| | 13.4<br>13.5 | Definition of Onset and Resolution of Adverse Events Other Propinions of Adverse Event Property | 70<br>71 |
| | 13.5 | Other Recipients of Adverse Event Reports Specific Examples for Expedited Reporting | 71 |
| 140 | | | |
| 14.0 | 14.1 | ORDS, REPORTING, AND DATA AND SAFETY MONITORING PLAN Categories of Research Records | 73<br>73 |
| | 14.1 | CDUS | 73 |
| | 14.3 | CRADA/CTA/CSA | 73 |
| | 14.4 | Data and Safety Monitoring Plan | 75 |
| | | $\mathcal{L}$ | |

CHILDREN'S ONCOLOGY GROUP



| REFERENCES | 76 |
|---|---|
| APPENDIX I: PERFORMANCE STATUS SCALES/SCORES | 80 |
| APPENDIX II: CYP3A4 SUBSTRATES, INDUCERS AND INHIBITORS | 81 |
| APPENDIX III-A: MEDICATION DIARY FOR LY3023414 | 84 |
| APPENDIX III-B: PATIENT DRUG INFORMATION HANDOUT AND WALLET CARE | ) |
| APPENDIX IV: LY3023414 DOSING NOMOGRAM | 90 |
| APPENDIX V: CORRELATIVE STUDIES GUIDE | 91 |
| APPENDIX VI: APEC1621D THERAPY DELIVERY MAP All Subsequent Cycles | 92<br>94 |
| APPENDIX VII-A: EXAMPLES OF ACTIONABLE MUTATIONS OF INTEREST FOR APEC COHORT A (TSC) | C1621D<br>96 |
| APPENDIX VII-B: EXAMPLES OF ACTIONABLE MUTATIONS OF INTEREST FOR APEC<br>COHORT B (PI3K) | C1621D<br>108 |
| APPENDIX VIII: TARGET HISTOLOGIES FOR APEC1621D EXPANSION COHORTS | 123 |
| APPENDIX IX: YOUTH INFORMATION SHEETS | 124 |
| APPENDIX X: CTEP AND CTSU REGISTRATION PROCEDURES | 126 |
| APPENDIX XI: TOXICITY-SPECIFIC GRADING | 130 |



#### **STUDY COMMITTEE**





Version Date: 10/28/2022

#### STUDY COMMITTEE, CONT.





PD



The Children's Oncology Group has received a Certificate of Confidentiality from the federal government, which will help us protect the privacy of our research subjects. The Certificate protects against the involuntary release of information about subjects collected during the course of our covered studies. The researchers involved in the studies cannot be forced to disclose the identity or any information collected in the study in any legal proceedings at the federal, state, or local level, regardless of whether they are criminal, administrative, or legislative proceedings. However, the subject or the researcher may choose to voluntarily disclose the protected information under certain circumstances. For example, if the subject or his/her guardian requests the release of information in writing, the Certificate does not protect against that voluntary disclosure. Furthermore, federal agencies may review our records under limited circumstances, such as a DHHS request for information for an audit or program evaluation or an FDA request under the Food, Drug and Cosmetics Act.

The Certificate of Confidentiality will not protect against mandatory disclosure by the researchers of information on suspected child abuse, reportable communicable diseases, and/or possible threat of harm to self or others.

#### **ABSTRACT**

This subprotocol is a component of the NCI-COG Pediatric MATCH trial APEC1621. The APEC1621SC screening protocol details the process used to identify actionable mutations in patient tumor samples which will determine eligibility for this subprotocol. This is a Phase 2 trial of LY3023414 in children with recurrent or refractory solid tumors, CNS tumors, and non-Hodgkin lymphomas harboring specified activating mutations of the PI3K/MTOR pathway. LY3023414 is a potent orally bioavailable small molecule inhibitor of class 1 PI3K isoforms, MTOR, and DNAPK. LY3023414 will be given twice daily continuously for 28-day cycles. Because the pediatric dose of LY3023414 has not been established, there will be a limited dose finding phase consisting of the first 12 evaluable patients enrolled on study. The primary endpoint will be objective response rate as determined by RECIST. Progression free survival (PFS) will be assessed as a secondary endpoint. In addition, toxicity will be assessed and the pharmacokinetics of LY3023414 in children will be evaluated.

#### EXPERIMENTAL DESIGN SCHEMA

| Day 1-28 | Day 28 |
|------------------------|------------|
| <b>LY3023414</b> (BID) | Evaluation |

Patients will receive LY3023414 twice daily for 28-day cycles. Evaluations will occur at the end of every other cycle.

Therapy will be discontinued if there is evidence of progressive disease or drug related dose-limiting toxicity that requires removal from therapy (Section 6.0). Therapy may otherwise continue for up to 6 cycles (approximately 6 months) provided the patient meets the criteria for starting subsequent cycles (Section 5.2) and does not meet any of the criteria for removal from protocol therapy criteria (Section 10.0).



#### 1.0 GOALS AND OBJECTIVES (SCIENTIFIC AIMS)

#### 1.1 Primary Aims

1.1.1 To determine the objective response rate (ORR; complete response + partial response) in pediatric patients treated with LY3023414 with advanced solid tumors, non-Hodgkin lymphomas or CNS tumors that harbor TSC loss of function mutations, and/or other PI3K/MTOR activating mutations.

#### 1.2 Secondary Aims

- 1.2.1 To estimate the progression free survival in pediatric patients treated with LY3023414 with advanced solid tumors, non-Hodgkin lymphomas or CNS tumors that harbor TSC loss of function mutations, and/or other PI3K/MTOR activating mutations.
- 1.2.2 To obtain information about the tolerability of LY3023414 in children with relapsed or refractory cancer.
- 1.2.3 To characterize the pharmacokinetics of LY3023414 in children with recurrent or refractory cancer.

#### 1.3 Exploratory Aims

- 1.3.1 To increase knowledge of the genomic landscape of relapsed pediatric solid tumors and lymphomas and identify potential predictive biomarkers (other than the genomic alteration for which study treatment was assigned) using additional genomic, transcriptomic, and proteomic testing platforms.
- 1.3.2 To explore approaches to profiling changes in tumor genomics over time through evaluation of circulating tumor DNA
- 1.3.3 To evaluate the frequency and mechanism of biallelic loss of function, and evaluate the expression of TSC1, TSC2, and PTEN in subjects who enroll with a loss of function mutation in one of these genes.



#### 2.0 BACKGROUND

#### 2.1 Introduction/Rationale for Development PI3K/MTOR pathway:

Phosphoinositide 3-kinases (PI3Ks) function downstream of receptor tyrosine kinases (RTKs) and G-protein coupled receptors (GPCRs) to stimulate a number of pro-growth and anti-apoptotic pathways within tumor cells. PI3Ks consist of a catalytic subunit (PIK3CA, PIK3CB, or PIK3CD) and a regulatory subunit (including PIK3R1). Mechanistically, PI3Ks phosphorylate phosphatidylinositol 4,5-bisphosphate (PIP2) to phosphatidyl 3,4,5-triphosphate (PIP3). Phosphatase and tensin homolog (PTEN) catalyzes the reverse reaction and thus negatively regulates this pathway. PIP3 allows the activation of protein kinase B (AKT) which in turn phosphorylates and inactivates Tuberous Sclerosis Complex 2 (TSC2). With TSC1, TSC2 normally inhibits the function of Ras homolog enriched in brain (RHEB), which stimulates mechanistic target of rapamycin (MTOR) activity. Thus, by inhibiting TSC1-TSC2, PI3K and AKT signaling stimulates MTOR activity to activate pro-growth and anti-apoptotic pathways in tumor cells.

#### PIK3/MTOR pathway mutations occur across a broad spectrum of pediatric cancers:

Histology specific sequencing efforts have demonstrated that activating mutations of the PI3K/MTOR pathway are present in a wide variety of pediatric solid tumors including osteosarcoma (24% of patients,) embryonal rhabdomyosarcoma (7.4% with PIK3CA mutation, rare patients with PTEN loss,) and diffuse intrinsic pontine gliomas (DIPG, 15% with PIK3CA mutation.)<sup>1-4</sup> While these studies can provide a suggestion of the frequency of mutations in patients eligible for the pediatric MATCH study, the precise frequency of mutations in this population as a whole is unknown. The best estimates likely come from cross-sectional studies of next generation sequencing of pediatric solid tumors and publically disclosed sequencing data released by Foundation Medicine, in which 1-10% of subjects had identified mutations in the PI3K/MTOR pathway.<sup>5,6</sup>

In the Foundation Medicine dataset, panel based sequencing of solid tumors from 981 pediatric patients detected the following mutations deemed to activate the PI3K/MTOR pathway:

- 42 PIK3CA mutations (including 26 brain tumors and 11 sarcomas)
- 4 PIK3R1 mutations (including 3 brain tumors and 1 sarcoma)
- 26 PTEN deletions or truncations (including 12 brain tumors, 10 sarcomas)
- 6 PTEN point mutations (including 4 brain tumors, 2 sarcomas)
- 8 TSC1 truncations or deletions (including 6 brain tumors)
- 6 TSC2 truncations or deletions (including 3 brain tumors and 2 sarcomas)
- 6 TSC2 point mutations (including 3 sarcomas and 3 extracranial embryonal tumors)
- 2 point mutations in MTOR (both in extracranial embryonal tumors)

Thus, activating PI3K/MTOR pathway alterations occurred in 10% of pediatric solid tumors, with the majority (55%) occurring in brain tumors and 31% occurring in sarcomas. However, not all of the variants reported by Foundation Medicine may be considered actionable for pediatric MATCH. As an example, the TSC2 A607T variant was observed 3 times and is reported as likely activating by the Foundation Medicine. However, a report studying the biochemical effects of TSC1 and TSC2 variants concluded that the variant was likely neutral. Conversely, none of these cross-sectional sequencing studies evaluated PTEN loss by IHC, which has been selected as an variant eligible for inclusion in this arm of pediatric MATCH. Thus, we estimate that in total between 2-5% of subjects enrolled on the pediatric MATCH protocol will have one of the defined PI3K/MTOR pathway



activating lesions eligible for this arm.

#### PI3K/MTOR pathway mutations may confer sensitivity to PI3K/MTOR inhibitors:

Multiple lines of evidence point to activating mutations of the PI3K/MTOR pathway as biomarkers of response to targeted PI3K and MTOR inhibitors. In preclinical studies in breast cancer, activating mutations of PIK3CA have been shown to confer sensitivity to PI3K inhibitors, AKT inhibitors, allosteric MTOR inhibitors, TORC1/2 inhibitors, and PI3K/MTOR inhibitors. These findings have been extended to other PIK3CA mutant tumor models including melanoma, lung, ovarian, prostate, and endometrial cancer. In preclinical studies, the relationship between PTEN deficiency and sensitivity to PI3K pathway inhibitors has been less clear. Some studies have found that some PTEN deficient cell lines are sensitive to PI3K inhibitors, I1,13,15 but others have found that PTEN deficient cells are preferentially resistant to PI3K/MTOR inhibitors. Recent studies have suggested that PTEN deficient tumors are specifically dependent on the beta rather than the alpha isoform of PI3K, and thus are sensitive to inhibitors of PIK3CB (which is inhibited by LY3023414). On the state of the present studies are sensitive by LY3023414).

In clinical trials, evidence also suggests that PI3K pathway mutations may confer sensitivity to MTOR inhibitors. The strongest evidence links TSC mutations to sensitivity. Everolimus was studied in a randomized phase 3 trial in patients with subependymal giant cell astrocytomas (SEGA) and a clinical diagnosis of TSC, most of whom are predicted to have loss of function mutations in TSC1 or TSC2. 35% of everolimus treated patients had at least 50% reduction in SEGA volume, and 53% of everolimus treated patients had at least 50% reduction in the volume of their concurrent angiomyolipomas vs none in placebo treated patients. Further, a retrospective study of patients with metastatic renal cell carcinoma found that mutations in MTOR, TSC1 or TSC2 were more common in patients who responded to rapalogs than those who did not respond. Patients with other tumors harboring TSC mutations have experienced extraordinatory responses to MTOR inhibition: two patients with metastatic RCC and biallelic inactivation of TSC1 experienced >24 month disease control with temsirolimus, and a patient metastatic bladder cancer with TSC1 and NF2 mutations experienced a >24 month complete response to everolimus.

There is also clinical evidence of response to MTOR inhibitors for mutations of other genes in this pathway including PIK3CA, PTEN, PIK3R1, and MTOR itself. PIK3CA mutation or PTEN loss of function mutations have correlated with response to allosteric MTOR inhibitors in several studies, although some studies have shown similar efficacy in both biomarker positive and biomarker negative patients. 10,28-32 As examples, of 258 adult patients with advanced cancers treated at a single institution on phase 1 studies that included various inhibitors of the PI3K/MTOR pathway, 35% (6 of 17) of patients with PIK3CA mutations achieved a partial response vs 6% of patients who did not have a PIK3CA mutation.<sup>28</sup> Similarly, of 23 patients with PIK3CA mutant breast, cervical, endometrial, and ovarian cancer treated on various phase 1 studies of PI3K/MTOR pathway inhibitors at a single institution, 30% had a partial response compared to 10% of patients with the same disease types lacking PIK3CA mutations.<sup>33</sup> An adult subject with an endometrial cancer harboring a PIK3R1 X448 Y452 deletion experienced a PR to LY3023414 in the phase 1 study of this agent. Several small case series have reported extraordinary responses to allosteric MTOR inhibitors in patients with activating mutations of the MTOR gene itself, including a 14-month complete remission to the combination of everolimus and pazopanib in a patient biallelic activating mutations in MTOR. 27,32,34



#### RAS pathway mutations are biomarkers of resistance to PI3K/MTOR inhibitors:

Preclinical studies in a number of cancer types have demonstrated that mutations in the RAS/MAPK pathway confir resistance to PI3K/MTOR pathway inhibitors.<sup>9,35-38</sup> While concurrent PIK3CA mutations and RAS pathway mutations are rare in breast cancer, these mutations co-exist with high frequency in a number of other adult malignancies, including colorectal and ovarian cancer.<sup>39</sup> Similarly, in the Foundation Medicine pediatric dataset, 20% of pediatric patients with TSC1/2 mutations, and 28% of pediatric patients with other PI3K pathway mutaions harbor concurrent RAS pathway mutations (Figure 1).

In preclinical studies, RAS pathway mutations confer resistance to PI3K/MTOR pathway inhibitors even when there is a concurrent activating mutation of the PI3K/MTOR pathway.<sup>36</sup> While the number of patients treated is small, retrospective analyses of early phase clinical trials also suggest that RAS pathway mutations are biomarkers of resistance, even for patients with PI3K/MTOR pathway activating mutations. Among 18 patients with PTEN negative tumors treated on phase I/II studies of everolimus at a single institution, 6 patients were found to have concurrent BRAF or KRAS mutations, and all had progressive disease as their best response. Among the 12 patients without these muations, there was 1 partial response, 7 patients with stable disease, and 4 patients with progressive disease as the best response. 10 Therefore, we will exclude patients with mutations that activate the RAS from APEC1621D.

## PI3K/MTOR inhibitors in biomarker negative patients:

While activating mutations in the PI3K/MTOR



Figure 1: Percentage of pediatric tumors with TSC1/2, other PI3K pathway, and RAS pathway mutations, excluding amplification, and their overlap. From Foundation Medicine pediatric data.

pathway correlate with response to PI3K/MTOR inhibitors, PI3K/MTOR inhibitors have also demonstrated efficacy against tumors without identified PI3K/MTOR pathway mutations both preclinically and in clinical trials. Several inhibitors of this pathway have been studied against pediatric cancer xenografts in the pediatric preclinical testing program (PPTP). Rapamycin, an allosteric MTOR inhibitor, had intermediate or high activity against 14 of 31 evaluable solid tumor xenografts, including partial responses in a rhabdoid tumor, two rhabdomyosarcomas, and a maintained CR in an osteosarcoma. A PI3K inhibitor (XL147) demonstrated significant tumor growth delay in 79% of solid tumor xenografts, and two MTOR kinase inhibitors (AZD8055 and MON1028) induced significant tumor growth delay in the majority to solid tumors xenografts studied (55.6% and 77%, respectively.) While the correlation between mutational status and response in these models is unknown, the percentage of xenografts with tumor growth delay is much higher than the percentage predicted to have genetic alterations in this pathway.

Clinically, an analysis of 724 women with advanced hormone receptor-positive breast cancer randomly assigned to treatment with exemestane with or without everolimus demonstrated that the efficacy of everolimus was largely independent of mutations in the



PI3K/MTOR pathway, the exception of a small group of patients with MTOR mutations for whom there may have been increased efficacy.<sup>32</sup> In this study, everolimus was associated with a hazard ratio of 0.37 (95% CI 0.25-0.55) for disease progression in patients without identified mutations in PIK3CA, PTEN, AKT, PIK3R1, or low PTEN expression by IHC. Clinical trials in adults with colorectal cancer have also shown that patients lacking PIK3CA and PTEN mutations can respond.<sup>29</sup>

In pediatric patients, the allosteric MTOR inhibitor temsirolimus demonstrated improved EFS compared to bevacizumab in a COG randomized phase 2 trial in recurrent rhabdomyosarcoma in combination with vinorelbine/cyclophosphamide. 44 This population was not biomarker selected. Evaluation for activating mutations in the PI3K/MTOR pathway in these subjects has not been completed. However, activating mutations in the PI3K/MTOR pathway are rare in rhabdomyosarcoma, occurring in less than 10% of patients.4

#### Other biomarkers of PI3K/MTOR response:

There are other potential biomarkers of efficacy of MTOR inhibitors including PI3K/MTOR pathway biochemical activity as assessed by phosphorylation of target proteins. In preclinical studies, response of breast cancer cell lines has been correlated with baseline phosphorylation of both AKT and S6K. 45,46 In clinical trials, response to MTOR inhibitors has also been correlated with phosphorylation of both AKT1 and S6RP in tumor cells as measured by IHC. 47-52 As examples, elevated baseline phospho-AKT levels were predictors of progression free survival in 40 NSCLC patients treated with everolimus.<sup>53</sup> Similarly, among 44 patients with glioblastoma treated with temsirolimus, baseline phosphorylation of S6K was associated with response to therapy. <sup>49</sup> However, other studies have not found a correlation between these biomarkers and response. 52,54

#### LY3023414:

LY3023414 is an orally bioavailable small molecule inhibitor of class 1 PI3K isoforms, MTOR, and DNAPK that has low nM potency, inhibiting PI3K isoforms at concentrations ranging from 6-78 nM, MTOR at 165 nM and DNAPK at 4 uM.55 LY3023414 was selected for the PI3K/MTOR arm of the pediatric MATCH study as a broadly active inhibitor of the PI3K/MTOR pathway with an available recommended phase 2 dose in adult patients. Due to its broad activity within this pathway, LY3023414 is appropriate to study across the range of alterations in the PI3K/MTOR pathway seen in pediatric cancers.

#### 2.2 **Preclinical Studies**

#### 2.2.1 **Antitumor Activity**

In vitro, LY3023414 inhibits purified class I isoforms, PI3Kalpha, PI3Kbeta, PI3Kdelta, and PI3Kgamma with IC50 values of 0.006 micromolar, 0.078 micromolar, 0.038 micromolar, and 0.024 micromolar, respectively. LY3023414 inhibits MTOR and DNA-PK with IC50 values of 0.165 micromolar and 0.004 micromolar in a cell lysate assay. LY3023414 is highly selective against a panel of 101 kinase enzymes and 200 kinases in a cell lysate assay system. LY3023414 demonstrates inhibitory activity against PI3K and MTOR and antiproliferative activity in a variety of cultured cancer cells.<sup>55</sup>

In studies of in vivo activity, LY3023414 as a single agent inhibits the growth of multiple tumor models with activating mutations in the PI3K/MTOR pathway, specifically the PTEN-deficient U87MG glioblastoma and 786-O renal carcinoma

This protocol is for research purposes only, see page 1 for usage policy. APEC1621D

models, the PIK3CA mutant NCI-H1975 non-small cell lung cancer (NSCLC) model, and a leukemia model driven by oncogenic Myc and mutant PIK3CA E545K. LY3023414 demonstrated equivalent tumor growth inhibition at doses of 15 mg/kg dosed twice daily or 30 mg/kg dosed daily in the U87MG xenograft model. <sup>55</sup>

In these preclinical studies, tumor growth inhibition is associated with pharmacodynamic markers of pathway inhibition. Phosphorylation of the PIK3CA and MTOR downstream targets AKT, S6K, S6RP, and 4E-BP1 was inhibited by LY3023414 in a dose-dependent and time-dependent manner in the U87MG xenograft model. Maximum inhibition of pAKT, pS6K, and p4E-BP1 was observed 30 minutes after oral dosing, while S6RP was maximally inhibited 2 to 3 hours or 4 to 6 hours after oral dosing for pS235/236 and pS240/244 S6RP, respectively.<sup>55</sup>

#### 2.2.2 Animal Toxicology

LY3023414 has been evaluated in nonclinical toxicology studies of 1 and 3 months in duration using daily oral dosing in rats and dogs.

Early deaths in the 1- and 3-month toxicology studies occurred in rats treated with daily doses  $\geq 15$  mg/kg and dogs treated with  $\geq 9$  mg/kg. The deaths in rats and dogs were preceded by premonitory clinical signs of deteriorating physical condition and moribundity. A single cause of death could not be established for the rat and dog mortalities, but indications of toxicity were present in multiple organs, including lymphoid tissue, the GI tract, and bone marrow.

Notable toxicities observed at non-lethal doses in the preclinical toxicology studies included dose related decreases in lymphocyte count and decreased or absent antibody response to keyhole limpet hemocyanin challenge in rats and dogs. Gastrointestinal toxicity was observed in both rats and dogs in a dose related manner. These included ulceration, epithelial atrophy, and villous blunting. Gastrointestinal toxicities were seen only in rats treated at doses  $\geq 10$  mg/kg and dogs treated at doses  $\geq 6$  mg/kg. Bone marrow hypocellularity was observed in animals treated above the MTD. In rats treated with doses  $\leq 15$  mg/kg and dogs treated with doses  $\leq 6$  mg/kg, there were no or only minimal bone marrow findings. Rats were noted to develop crusted skin and sores with both 1 and 3 month treatment, which were reversible when treatment was stopped. No effects on skin were seen in dogs. Hypospermia was observed in both rats and dogs treated with LY3023414 and was reversible in the 3 month dog study.

In dogs, blood insulin and glucose concentrations increased at doses of  $\geq 3$  mg/kg within 30 minutes of dosing and generally peaked at 1 to 2 hours after dosing. At doses  $\geq 9$  mg/kg, these changes were marked. At all doses, these increases returned to normal approximately 4 hours or 8 hours after dosing. Increased QT and QTc intervals were observed on Day 25 at the 6 mg/kg and 9 mg/kg doses in dogs. At 6 mg/kg, an increase of 4 msec to 16 msec was observed postdose and was reversible. At 9 mg/kg (a dose that exceeded the MTD based on clinical observations) increased QTc intervals were observed up to 19 hours postdose, with peak increases (37 msec) observed at approximately 3 hours postdose.

Effects on glucose metabolism are an expected pharmacologic effect based on the

role that PI3K and MTOR pathways play in glucose metabolism. Consistent with what has been observed with LY3023414, other small molecule inhibitors of the PI3K/MTOR pathway cause similar changes to glucose metabolism.<sup>56</sup>

The genotoxic potential of LY3023414 was evaluated in a test battery that included a bacterial mutagenicity test ("Ames assay"), an in vitro chromosome aberrations assay in Chinese hamster ovary (CHO) cells, and an in vivo rat bone marrow micronucleus test. Collectively, the genetic toxicology results (negative for gene mutations in bacteria, negative for clastogenic activity in CHO cells, and positive for micronucleus induction in rat bone marrow erythrocytes) provide the weight of evidence to support the conclusion that LY3023414 has an ugenic activity. The positive micronucleus results with LY3023414 were consistently observed in rats at acute doses ≥ 30 mg/kg, while negative results were obtained at 20 mg/kg. The exposure (Cmax) associated with a 30 mg/kg dose following the first day of dosing in the 4-week repeat-dose toxicology study was 2400 ng/mL (for males). Assuming dose-proportionality of the rat exposures in the 4-week study, the Cmax value associated with an acute 20 mg/kg dose can be estimated to be 1600 ng/mL. Because dose-response curves for aneugens are well-known to have a threshold, human exposures to LY3023414 at levels below the 1600-ng/mL threshold are not expected to be accompanied by any aneugenic risks.

In an enhanced pilot embryo-fetal developmental study of LY3023414 in rats, embryo-fetal lethality was seen along with an increase in fetal and litter incidence of external, visceral, and skeletal malformations. These consisted primarily of cranial, abdominal wall, cardiovascular, vertebral, rib, and sternebrae dysmorphologies when female Sprague-Dawley rats were administered 15 mg/kg (90 mg/m²) LY3023414 orally on gestation days 6 through 17. There were no compound-related changes in embryo-fetal survival; fetal weight; or external, visceral, or skeletal morphology at  $\leq 2$  mg/kg (12 mg/m²).

In conclusion, the nonclinical toxicology findings with LY3023414 are consistent with the known toxicity profile of inhibution of the PI3K/MTOR signaling pathway. Inhibitors of the PI3K/MTOR pathway are well-characterized both clinically and nonclinically, with the predominant target organs for toxicity in nonclinical species being the GI tract, hematopoietic system, lymphoid tissues, and reproductive tissues. Additional target organs for toxicity include the kidney, skin, and the cardiovascular system. These toxicities are anticipated to be reversible. <sup>57</sup>

#### 2.3 Adult Studies

#### 2.3.1 Phase 1 Studies

The recommended phase 2 dose of LY3023414 in adult subjects with advanced cancer has been determined in a phase 1 study (NCT01655225). As of the cut-off date (08 June 2016), a total of 110 patients have received LY3023414 on this study. A total of 25 patients were enrolled in the dose-escalation portion (Part A) investigating continuous QD administration of LY3023414. Patients received LY3023414 at 7 dose levels ranging 20 mg to 450 mg daily. A dose of 325 mg once daily was determined to the maximum tolerated dose based on dose limiting toxicities (DLTs) observed in 3 of 3 patients treated at 450 mg once daily. These DLTs consisted of thrombocytopenia (Grade 4), hypotension (Grade 3), and hyperkalemia (Grade 3).

This protocol is for research purposes only, see page 1 for usage policy. APEC1621D

Following Part A, a second dose-escalation phase (Part A2) was initiated to investigate BID oral administration of LY3023414. Part A2 was completed with a total of 13 patients who received LY3023414 BID at dose levels ranging from 150 mg to 250 mg twice daily. A dose of 200 mg twice daily was determined to be the MTD based on DLTs observed in 3 of 4 patients treated at 250 mg twice daily. These DLTs consisted of hypophosphatemia (Grade 4), fatigue, and mucositis (Grade 3; all n = 1). At the 200 mg twice daily dose level, 1 of 6 patients experienced a DLT in the form of grade 2 nausea.

Part B of this study is ongoing enrolling patients into tumor-specific cohorts (B1 through B6) at the recommended phase 2 dose of 200 mg BID. As of the data cut-off date (08 June 2016), a total of 56 patients received 200 mg BID LY3023414 monotherapy; 9 patients received 200 mg BID LY3023414 in combination with fulvestrant; and 7 patients received 100-200 mg BID of LY3023414 with cisplatin and pemetrexed.

An additional phase 1 study of LY3023414 is now enrolling in Japanese patients with advanced malignancies with 11 of 12 planned subjects enrolled as of 8 June 2016.

#### 2.3.2 Phase 2 Studies

No phase 2 studies of LY3023414 have been completed to date. A phase 2 double blind, placebo controlled study of enzalutamide with or without 200 mg BID of LY3023414 is currently enrolling men with castration-resistant prostate cancer (NCT02407054). As of 8 June 2016, 13 subjects have been enrolled to the open-label safety lead-in phase and enrollment to the randomized double-blind, placebo-controlled treatment part is ongoing with 6 of 132 subjects enrolled. A second phase 2 single arm study of LY3023414 with necitumumab is currently enrolled men with advanced or metastatic squamous non-small cell carcinoma of the lung (NCT02443337). 22 of 48 planned patients have been enrolled as of 8 June 2016.

#### 2.3.3 Pharmacology/Pharmacokinetics/Correlative and Biological Studies

#### 2.3.3.1 Pharmacology:

In vitro human microsomal data indicated possible time-dependent inhibition of CYP3A4 by LY3023414. To investigate this, one objective of the now completed Part B1 cohort in the phase 1 study of LY3023414 was to investigate whether LY3023414 impacts (decreases) the metabolic clearance of drugs that are metabolized through CYP3A4, such as midazolam. The results indicate that LY3023414 increases the exposure (AUC∞) of midazolam by a geometric mean ratio of 1.46 (90% CI 1.21-1.76). Therefore, LY3023414 is classified as a weak CYP3A4 inhibitor because it leads to less than a 2-fold increase in exposure of the enzyme substrate drug.

Extensive PK time-matched central ECGs were collected in parts A and A2 of the adult phase 1 study of LY3023414 at doses up to 450 mg. Despite changes in the QT interval in preclinical studies in dogs, LY3023414 did not lead to clinically and/or statistically significant

THIS PROTOCOL IS FOR RESEARCH PURPOSES ONLY, SEE PAGE 1 FOR USAGE POLICY. APEC1621D

changes in QTcF in humans.

#### 2.3.3.2 Pharmacokinetics:

The world's childhood

The pharmacokinetics of LY3023414 in adults with advanced malignancies is available from subjects treated on the phase 1 study. Following oral administration, LY3023414 concentrations reach a maximum value at approximately 1 to 2 hours postdose. Cmax and AUC $\infty$  increase approximately dose-proportionally from 20 to 325 mg; however, Cmax and AUC $\infty$  at the dose of 450 mg show a greater than dose proportional increase.

A single 200 mg dose of LY3023414 resulted in a geometric mean Cmax value of 863 ng/mL. Cmax and AUC<sub>0-12 hr</sub> at steady state on Day 15 were 884 ng/mL and 2950 ng·h/mL for the 200 mg twice daily dose.

LY3023414 has a geometric mean half-life ( $t_{1/2}$ ) of 1.87 hours for all doses of 20 mg to 325 mg. Mean apparent clearance (CL/F) and mean apparent volume of distribution (Vz/F) were calculated to be 74.3 L/hr and 200 L, respectively, across the 20- mg to 325-mg dose range.

Based on the short terminal  $t_{1/2}$ , steady state is anticipated to be reached after 1 dose of LY3023414. In adult subjects, there is limited accumulation of LY3023414 with a geometric mean exposure ratio (Day 15: Day 1) of 1.28 with BID dosing. This small/moderate ratio indicates a slight decrease in LY3023414 CL/F after repeated dosing between Day 1 and Day 15 (in particular for doses  $\geq$  150 mg). However, once steady state is stabilized, LY3023414 CL/F, and hence exposure (AUC), is stable.

#### 2.3.3.3 Pharmacodynamics:

Inhibition of phosphorylation of the MTOR target 4EBP1 was evaluated in 35 patients treated with LY302314 in Parts A and A2 of the phase 1 study. At doses above 150 mg daily, LY3023414 inhibits phosphorylation of 4EBP1 in PBMCs by  $\geq$  90%.

#### 2.3.3.4 Response:

As of 08 June 2016, limited data are available for only a preliminary evaluation of clinical activity of LY3023414 in the ongoing adult phase 1 study. Most notably, in the dose-escalation part of this study, a woman with an endometrial cancer bearing PIK3R1 and PTEN mutations experienced a durable PR with 50% reduction in tumor volume. In the tumor-specific expansion cohorts, a partial response was observed in 5 patients (out of 74 patients enrolled).

#### 2.4 Pediatric Studies

There have been no prior studies of LY3023414 in children.

#### 2.5 Overview of Proposed Pediatric Study

This subprotocol is a component of the Pediatric MATCH trial. The APEC1621SC screening protocol details the assay used for the integral genomic profiling which will determine eligibility for this arm. This is a phase 2 trial of LY3023414 in children with recurrent or refractory solid tumors, CNS tumors, and non-Hodgkin lymphomas harboring

This protocol is for research purposes only, see page 1 for usage policy. APEC1621D

specified activating mutations of the PI3K/MTOR pathway.

Because the pediatric dose of LY3023414 has not been established, there will be a limited dose finding phase consisting of the first 12 evaluable patients enrolled on study. Patients will receive LY3023414 twice daily for 28-day cycles. The first 6 evaluable patients will be enrolled at a dose of 80 mg/m<sup>2</sup>/dose BID, equivalent to 70% of the maximum tolerated dose (MTD) in adults. There will be a single dose escalation to 115 mg/m<sup>2</sup>/dose BID (100% of the adult MTD) or de-escalation to 55 mg/m<sup>2</sup>/dose BID (50% of the adult MTD) for the next six subjects. Following the first 12 evaluable patients, all subsequent patients will be enrolled at the highest dose level not exceeding the pediatric MTD. Patients enrolled in the dose escalation component will be included in the analysis of efficacy.

The primary aim of this trial will be to establish the objective response rate to LY3023414 in patients with inactivating mutations in TSC1/2 and/or other specified PI3K/MTOR activating mutations.

Key secondary objectives include evaluating the tolerability and pharmacokinetics of LY3023414 in pediatric patients as no pediatric studies of LY3023414 have been conducted to date. Toxicity will be assessed using CTCAE V5.0. Imaging for disease evaluation will occur every other cycle. Disease response will be assessed according to RECIST v1.1 criteria for solid tumors and 2-dimensional measurement for CNS tumors.



#### 3.0 SCREENING AND STUDY ENROLLMENT PROCEDURES

#### 3.1 Study Enrollment

The world's childhood

Patient enrollment for this study will be facilitated using the Oncology Patient Enrollment Network (OPEN), a web-based registration system available on a 24/7 basis. It is integrated with the NCI Cancer Trials Support Unit (CTSU) Enterprise System for regulatory and roster data and, upon enrollment, initializes the patient position in the RAVE database.

#### 3.1.1 Access requirements for OPEN:

Patient enrollment for this study will be facilitated using the Oncology Patient Enrollment Network (OPEN), a web-based registration system available on a 24/7 basis. OPEN is integrated with CTSU regulatory and roster data and with the Lead Protocol Organization (LPOs) registration/randomization systems or Theradex Interactive Web Response System (IWRS) for retrieval of patient registration/randomization assignment. OPEN will populate the patient enrollment data in NCI's clinical data management system, Medidata Rave.

#### **Requirements for OPEN access:**

- A valid CTEP-IAM account;
- To perform enrollments: Be on a LPO roster, ETCTN Corresponding roster, or PO roster with the role of Registrar. Registrars must hold a minimum of an AP registration type;
- Have an approved site registration for a protocol prior to patient enrollment.

To assign an Investigator (IVR) or Non-Physician Investigator (NPIVR) as the treating, crediting, consenting, drug shipment (IVR only), or receiving investigator for a patient transfer in OPEN, the IVR or NPIVR must list the IRB number used on the site's IRB approval on their Form FDA 1572 in RCR.

Prior to accessing OPEN, site staff should verify the following:

- Patient has met all eligibility criteria within the protocol stated timeframes;
   and
- All patients have signed an appropriate consent form and HIPAA authorization form (if applicable).

Note: The OPEN system will provide the site with a printable confirmation of registration and treatment information. Please print this confirmation for your records.

Access OPEN at <a href="https://open.ctsu.org">https://open.ctsu.org</a> or from the OPEN link on the CTSU members' website. Further instructional information is in the OPEN section of the CTSU website at <a href="https://www.ctsu.org">https://open.ctsu.org</a>. For any additional questions, contact the CTSU Help Desk at 1-888-823-5923 or <a href="mailto:ctsu.org">ctsu.org</a>. at 1-888-823-5923 or <a href="mailto:ctsu.org">ctsu.org</a>.

Please see Appendix X for detailed CTEP and CTSU Registration Procedures including: registration in Registration and Credential Repository (RCR),

This protocol is for research purposes only, see page 1 for usage policy. APEC1621D

requirements for site registration, submission of regulatory documents and how to check your site's registration status.

#### 3.1.2 IRB Approval

The world's childhood

Each investigator or group of investigators at a clinical site must obtain IRB approval for this protocol and submit IRB approval and supporting documentation to the CTSU Regulatory Office before they can be approved to enroll patients. For CTEP and Division of Cancer Prevention (DCP) studies open to the National Clinical Trials Network (NCTN) and NCI Community Oncology Research Program (NCORP) Research Bases after March 1, 2019, all U.S.-based sites must be members of the NCI Central Institutional Review Board (NCI CIRB). In addition, U.S.-based sites must accept the NCI CIRB review to activate new studies at the site after March 1, 2019. Local IRB review will continue to be accepted for studies that are not reviewed by the CIRB, or if the study was previously open at the site under the local IRB. International sites should continue to submit Research Ethics Board (REB) approval to the CTSU Regulatory Office following country-specific regulations.

Sites participating with the NCI CIRB must submit the Study Specific Worksheet for Local Context (SSW) to the CIRB using IRBManager to indicate their intent to open the study locally. The NCI CIRB's approval of the SSW is automatically communicated to the CTSU Regulatory Office, but sites are required to contact the CTSU Regulatory Office at <a href="https://creativecommons.org/creat

Sites using their local IRB or REB, must submit their approval to the CTSU Regulatory Office using the Regulatory Submission Portal located in the Regulatory section of the CTSU website. Acceptable documentation of local IRB/REB approval includes:

- Local IRB documentation;
- IRB-signed CTSU IRB Certification Form; and/or
- Protocol of Human Subjects Assurance Identification/IRB Certification/Declaration of Exemption Form.

In addition, the Site-Protocol Principal Investigator (PI) (i.e. the investigator on the IRB/REB approval) must meet the following criteria in order for the processing of the IRB/REB approval record to be completed:

- Holds an active CTEP status;
- Rostered at the site on the IRB/REB approval (applies to US and Canadian sites only) and on at least one participating roster;
- If using NCI CIRB, rostered on the NCI CIRB Signatory record;
- Includes the IRB number of the IRB providing approval in the Form FDA 1572 in the RCR profile; and
- Holds the appropriate CTEP registration type for the protocol.

THIS PROTOCOL IS FOR RESEARCH PURPOSES ONLY, SEE PAGE 1 FOR USAGE POLICY. APEC 1621D

#### **Additional Requirements**

Additional requirements to obtain an approved site registration status include:

- An active Federal Wide Assurance (FWA) number;
- An active roster affiliation with the Lead Protocol Organization (LPO) or a Participating Organization (PO); and
- Compliance with all protocol-specific requirements (PSRs).

For information about the submission of IRB/REB approval documents and other regulatory documents as well as checking the status of study center registration packets, please see Appendix X.

Institutions with patients waiting that are unable to use the Portal should alert the CTSU Regulatory Office immediately at 1-866-651-2878 in order to receive further instruction and support. For general (non-regulatory) questions call the CTSU General Helpdesk at: 1-888-823-5923.

Note: Sites participating on the NCI CIRB initiative and accepting CIRB approval for the study are not required to submit separate IRB approval documentation to the CTSU Regulatory Office for initial, continuing or amendment review.

Investigators and site staff will need to be registered with CTEP and have a valid and active Cancer Therapy Evaluation Program-Identity and Access Management (CTEP-IAM) account (check at < <a href="https://eapps-ctep.nci.nih.gov/iam/index.jsp">https://eapps-ctep.nci.nih.gov/iam/index.jsp</a>). This is the same account (user id and password) used for credentialing in the CTSU members' web site. To perform registrations in OPEN, the site user must have been assigned the 'Registrar' role on the relevant Group or CTSU roster. OPEN can be accessed at <a href="https://www.ctsu.org">https://www.ctsu.org</a> or from the OPEN tab on the CTSU members' side of the website at <a href="https://www.ctsu.org">https://www.ctsu.org</a>.

#### 3.1.3 Genetic Screening Procedures for Eligibility

Patient enrollment onto the APEC1621SC screening protocol is required. In Stage 2 of Pediatric MATCH (effective with Amendment #4A of APEC1621SC for patients enrolling on screening protocol) tumor genomic testing results from a CAP/CLIA-certified laboratory will be reviewed by the APEC1621SC Molecular Review Committee after APEC1621SC screening protocol enrollment to confirm the identification of an actionable Mutation of Interest (aMOI) for which a MATCH treatment subprotocol is available. Questions regarding interpretation of tumor testing results for potential APEC1621D study patients (such as whether a specific mutation would be considered actionable for the study) should be directed to the APEC1621SC and APEC1621D study chairs.

The treatment assignment to a MATCH subprotocol (if a relevant aMOI is detected) will be communicated to the enrolling institution via the COG treatment assignment mechanism, upon which a reservation to APEC1621D will be secured by COG. Reservations should be withdrawn by the institution if at any point the patient indicates they do NOT intend to consent to participation or the site investigator indicates the patient will never be eligible for APEC1621D.



#### 3.2 Informed Consent/Assent

The investigational nature and objectives of the trial, the procedures and treatments involved and their attendant risks and discomforts, and potential alternative therapies will be carefully explained to the patient or the patient's parents or guardian if the patient is a child, and a signed informed consent and assent will be obtained according to institutional guidelines.

#### 3.3 Screening Procedures

Diagnostic or laboratory studies performed exclusively to determine eligibility for this trial must only be done after obtaining written informed consent. This can be accomplished through the study-specific protocol. Documentation of the informed consent for screening will be maintained in the patient's research chart. Studies or procedures that were performed for clinical indications (not exclusively to determine eligibility) may be used for baseline values even if the studies were done before informed consent was obtained.

#### 3.4 Eligibility Checklist

Before the patient can be enrolled, the responsible institutional investigator must sign and date the completed eligibility checklist. A signed copy of the checklist will be uploaded into RAVE immediately following enrollment.

#### 3.5 Study Enrollment

Following a MATCH treatment assignment to a protocol, patients may be enrolled on the study once all eligibility requirements for the study have been met. Before enrolling a patient on study, the Study Chair or Vice Chair should be notified. Patients who give informed consent for the protocol in order to undergo screening for eligibility are not considered enrolled and should not be enrolled until the screening is completed and they are determined to meet all eligibility criteria. Study enrollment in Stage 2 of Pediatric MATCH (effective with Amendment #4A of APEC1621SC for patients enrolling on screening protocol) is outlined in Section 3.1.3.

Patients must be enrolled within 2 weeks (14 days) of treatment assignment. The date protocol therapy is projected to start must be no later than 7 calendar days after the date of enrollment. Patients enrolling onto APEC1621D will have a COG ID obtained through their prior enrollment onto the screening protocol or from a prior COG study. Patients who are started on protocol therapy prior to study enrollment will be considered ineligible.

All clinical and laboratory studies to determine eligibility must be performed within 7 days prior to enrollment unless otherwise indicated in the eligibility section below.

Note: No starter supplies will be provided. Drug orders of LY3023414 should be placed with CTEP after enrollment and treatment assignment to APEC1621D with consideration for timing of processing and shipping to ensure receipt of drug supply prior to start of protocol therapy.

#### 3.6 Institutional Pathology Report

The institutional pathology report from the tumor specimen submitted for sequencing will have been uploaded into RAVE immediately following enrollment on the APEC1621SC screening protocol.

#### 3.7 **Dose Assignment**

The dose level will be assigned via OPEN at the time of study enrollment.



#### 4.0 **PATIENT ELIGIBILITY**

All clinical and laboratory studies to determine eligibility must be performed within 7 days prior to enrollment unless otherwise indicated. Laboratory values used to assess eligibility must be no older than seven (7) days at the start of therapy. Laboratory tests need **not** be repeated if therapy starts **within** seven (7) days of obtaining labs to assess eligibility. If a post-enrollment lab value is outside the limits of eligibility, or laboratory values are older than 7 days, then the following laboratory evaluations must be re-checked within 48 hours prior to initiating therapy: CBC with differential, bilirubin, ALT (SGPT) and serum creatinine. If the recheck is outside the limits of eligibility, the patient may not receive protocol therapy and will be considered off protocol therapy. Imaging studies, bone marrow biopsy and/or aspirate (when applicable) must be obtained within 14 days prior to start of protocol therapy (repeat the tumor imaging if necessary).

<u>Clarification in timing when counting days</u>: As an example, please note that if the patient's last day of prior therapy is September 1<sup>st</sup>, and the protocol requires waiting <u>at least</u> 7 days for that type of prior therapy, then that patient cannot be enrolled until September 8<sup>th</sup>.

<u>Important note</u>: The eligibility criteria listed below are interpreted literally and cannot be waived. All clinical and laboratory data required for determining eligibility of a patient enrolled on this trial must be available in the patient's medical or research record which will serve as the source document for verification at the time of audit.

#### 4.1 Inclusion Criteria

4.1.1 APEC1621SC: Patient must have enrolled onto APEC1621SC and must have been given a treatment assignment to MATCH to APEC1621D based on the presence of an actionable mutation as defined in APEC1621SC. Examples of actionable mutations for APEC1621D are listed in <a href="Appendix VII-A">Appendix VII-A</a> and <a href="Appendix VII-B">Appendix VII-B</a>.

Note that treatment assignment may be to primary cohort A for patients with TSC1 or TSC2 loss of function mutations or primary cohort B for patients with other PI3K/MTOR pathway mutations (see <a href="section 11.3.1">section 11.3.1</a>).

- 4.1.2 Age: Patients must be  $\geq$  than 12 months and  $\leq$  21 years of age at the time of study enrollment.
- 4.1.3 <u>BSA</u>: Patients accruing to Dose Level 1 must have a body surface area  $\geq 0.52$  m<sup>2</sup> at the time of study enrollment. Patients accruing to Dose Level 2 must have a body surface area  $\geq 0.37$  m<sup>2</sup> at the time of study enrollment. Patients accruing to Dose Level -1 must have a body surface area  $\geq 0.75$  m<sup>2</sup> at the time of study enrollment.

#### 4.1.4 Disease Status:

Patients must have radiographically **measurable** disease (See <u>section 12.0</u>) at the time of study enrollment. Patients with neuroblastoma who do not have measurable disease but have MIBG+ evaluable disease are eligible. Measurable disease in patients with CNS involvement is defined as any lesion that is at minimum 10 mm in one dimension on standard MRI or CT.

Note: The following do not qualify as measurable disease:

THIS PROTOCOL IS FOR RESEARCH PURPOSES ONLY. SEE PAGE 1 FOR USAGE POLICY. APEC1621D

- malignant fluid collections (e.g., ascites, pleural effusions)
- bone marrow infiltration except that detected by MIBG scan for neuroblastoma
- lesions only detected by nuclear medicine studies (e.g., bone, gallium or PET scans) except as noted for neuroblastoma
- elevated tumor markers in plasma or CSF
- previously radiated lesions that have not demonstrated clear progression post radiation
- leptomeningeal lesions that do not meet the measurement requirements for RECIST 1.1.
- bone lesions without an associated soft tissue mass  $\geq 10$  mm in greatest diameter. Bone lesions with an associated soft tissue mass  $\geq 10$  mm in greatest diameter imaged by CT or MRI are considered measurable.
- 4.1.5 Performance Level: Karnofsky ≥ 50% for patients > 16 years of age and Lansky ≥ 50 for patients ≤ 16 years of age (See Appendix I). Note: Neurologic deficits in patients with CNS tumors must have been stable for at least 7 days prior to study enrollment. Patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.

#### 4.1.6 Prior Therapy

- 4.1.6.1 Patients must have fully recovered from the acute toxic effects of all prior anti-cancer therapy and must meet the following minimum duration from prior anti-cancer directed therapy prior to enrollment. If after the required timeframe, the numerical eligibility criteria are met, e.g. blood count criteria, the patient is considered to have recovered adequately.
  - a. Cytotoxic chemotherapy or other anti-cancer agents known to be myelosuppressive.

See

https://www.cogmembers.org/Site/Disc/DevTherapeutics/Default.aspx#ToolsReferenceMaterials for commercial and Phase 1 investigational agent classifications. For agents not listed, the duration of this interval must be discussed with the study chair and the study-assigned Research Coordinator prior to enrollment.

- i.  $\geq 21$  days after the last dose of cytotoxic or myelosuppressive chemotherapy (42 days if prior nitrosourea).
- b. Anti-cancer agents not known to be myelosuppressive (e.g. not associated with reduced platelet or ANC counts): ≥ 7 days after the last dose of agent.

See

https://www.cogmembers.org/Site/Disc/DevTherapeutics/Default.aspx#ToolsReferenceMaterials for commercial and Phase 1 investigational agent classifications. For agents not listed, the duration of this interval must be discussed with the study chair and the study-assigned Research Coordinator prior to enrollment.

This protocol is for research purposes only. See page 1 for usage policy. APEC1621D

- c. Antibodies:  $\geq 21$  days must have elapsed from infusion of last dose of antibody, and toxicity related to prior antibody therapy must be recovered to Grade  $\leq 1$ .
- d. <u>Corticosteroids</u>: See <u>Section 4.2.2.1</u>. If used to modify <u>immune</u> <u>adverse events</u> related to prior therapy, ≥ 14 days must have elapsed since last dose of corticosteroid.
- e. <u>Hematopoietic growth factors</u>: ≥ 14 days after the last dose of a longacting growth factor (e.g. pegfilgrastim) or 7 days for short-acting growth factor. For growth factors that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur. The duration of this interval must be discussed with the study chair and the study-assigned Research Coordinator.
- f. Interleukins, Interferons and Cytokines (other than hematopoetic growth factors): ≥ 21 days after the completion of interleukins, interferon or cytokines (other than hematopoetic growth factors)
- g. Stem cell Infusions (with or without TBI):
  - Allogeneic (non-autologous) bone marrow or stem cell transplant, or any stem cell infusion including DLI or boost infusion: ≥ 84 days after infusion and no evidence of GVHD.
  - Autologous stem cell infusion including boost infusion:  $\geq 42$  days.
- h. <u>Cellular Therapy</u>: ≥ 42 days after the completion of any type of cellular therapy (e.g. modified T cells, NK cells, dendritic cells, etc.)
- i. XRT/External Beam Irradiation including Protons:  $\geq$  14 days after local XRT;  $\geq$  150 days after TBI, craniospinal XRT or if radiation to  $\geq$  50% of the pelvis;  $\geq$  42 days if other substantial BM radiation.
  - Note: Radiation may not be delivered to "measurable disease" tumor site(s) being used to follow response to subprotocol treatment.
- j. <u>Radiopharmaceutical therapy</u> (e.g., radiolabeled antibody, 131I-MIBG): ≥ 42 days after systemically administered radiopharmaceutical therapy.
- k. Patients must not have received prior exposure to LY3023414.
- 1. Patients must not have received prior exposure to an agent specifically directed at the PI3K/MTOR pathway (a PI3K inhibitor, an AKT inhibitor, an MTOR inhibitor, including rapalogs, or a combined PI3K/MTOR inhibitor).



#### 4.1.7 **Organ Function Requirements**

#### 4.1.7.1 Adequate Bone Marrow Function Defined as:

- a. For patients with solid tumors without known bone marrow involvement:
  - Peripheral absolute neutrophil count (ANC) ≥ 1000/mm<sup>3</sup>
  - Platelet count ≥ 100,000/mm<sup>3</sup> (transfusion independent, defined as not receiving platelet transfusions for at least 7 days prior to enrollment)
- Patients with known bone marrow metastatic disease will be b. eligible for study provided they meet the blood counts in Section 4.1.7.1.a (may receive transfusions provided they are not known to be refractory to red cell or platelet transfusions). These patients will not be evaluable for hematologic toxicity.

#### 4.1.7.2 Adequate Renal Function Defined as:

- Creatinine clearance or radioisotope GFR  $\geq$  70ml/min/1.73 m<sup>2</sup> or
- A serum creatinine based on age/gender as follows:

| Age | Maximum Serum<br>Creatinine (mg/dL) | |
|------------------|-------------------------------------|--------|
| | Male | Female |
| 1 to < 2 years | 0.6 | 0.6 |
| 2 to < 6 years | 0.8 | 0.8 |
| 6 to < 10 years | 1 | 1 |
| 10 to < 13 years | 1.2 | 1.2 |
| 13 to < 16 years | 1.5 | 1.4 |
| ≥ 16 years | 1.7 | 1.4 |

The threshold creatinine values in this Table were derived from the Schwartz formula for estimating GFR utilizing child length and stature data published by the CDC.58

#### 4.1.7.3 Adequate Liver Function Defined as:

- Bilirubin (sum of conjugated + unconjugated)  $\leq 1.5$  x upper limit of normal (ULN) for age
- SGPT (ALT)  $\leq$  135 U/L. (For the purpose of this study, the ULN for SGPT is 45 U/L.)
- Serum albumin  $\geq 2$  g/dL.

#### 4.1.7.4 Normal blood glucose for age

Patients must have a normal blood sugar level for age. If an initial random draw (i.e. non-fasting) blood glucose value is out of range, it is acceptable to repeat this test as a fasting draw.

#### 4.1.7.5 Lipids:

Patients must have a serum triglyceride level ≤ 300 mg/dL and serum cholesterol level ≤ 300 mg/dL. If an initial random draw (i.e. nonfasting) is out of range, it is acceptable to repeat this test as a fasting draw.

#### 4.1.7.6 Adequate Neurologic Function Defined as:

Patients with seizure disorder may be enrolled if on anticonvulsants and well controlled.



- Nervous system disorders (by CTCAE V 5.0) resulting from prior therapy must be ≤ Grade 2, with the exception of decreased tendon reflex (DTR). Any grade of DTR is eligible.
- 4.1.7.7 Adequate Cardiac Function Defined as:
  - QTc interval ≤ 480 milliseconds
- 4.1.8 Patients must be able to swallow intact tablets.
- 4.1.9 <u>Informed Consent:</u> All patients and/or their parents or legally authorized representatives must sign a written informed consent. Assent, when appropriate, will be obtained according to institutional guidelines.

#### 4.2 Exclusion Criteria

#### 4.2.1 Pregnancy or Breast-Feeding

Pregnant or breast-feeding women will not be entered on this study due to risks of fetal and teratogenic adverse events as seen in animal studies. Pregnancy tests must be obtained in girls who are post-menarchal. Males or females of reproductive potential may not participate unless they have agreed to use an effective contraceptive method while receiving study treatment and for 3 months after the last dose of LY3023414.

#### 4.2.2 Concomitant Medications

- 4.2.2.1 <u>Corticosteroids</u>: Patients receiving corticosteroids who have not been on a stable or decreasing dose of corticosteroid for at least 7 days prior to enrollment are not eligible. If used to modify <u>immune adverse events</u> related to prior therapy, ≥ 14 days must have elapsed since last dose of corticosteroid (See Section 4.1.6.1.d).
- 4.2.2.2 <u>Investigational Drugs</u>: Patients who are currently receiving another investigational drug are not eligible.
- 4.2.2.3 <u>Anti-cancer Agents</u>: Patients who are currently receiving other anti-cancer agents are not eligible.
- 4.2.2.4 Anti-GVHD agents post-transplant:

Patients who are receiving cyclosporine, tacrolimus or other agents to prevent graft-versus-host disease post bone marrow transplant are not eligible for this trial.

- 4.2.3 <u>Infection</u>: Patients who have an uncontrolled infection are not eligible.
- 4.2.4 <u>Diabetes:</u> Patients who have insulin dependent diabetes are not eligible.
- 4.2.5 Patients who have received a prior solid organ transplantation are not eligible.
- 4.2.6 Patients with SubEpendymal Giant cell Astrocytomas (SEGAs) are not eligible because everolimus is approved by the FDA for this patient population.



4.2.7 Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study are not eligible.

#### 5.0 TREATMENT PROGRAM

The world's childhood

#### 5.1 Overview of Treatment Plan

| Day 1-28 | Day 28 |
|-------------------------------|------------|
| LY3023414 orally, twice daily | Evaluation |

LY3023414 will be administered orally twice daily. For patients enrolled during the dose-confirmation part of the study, the Cycle 1 Day 1 PM dose of LY3023414 will be omitted for PK sampling.

Therapy will be discontinued if there is evidence of progressive disease or drug related dose-limiting toxicity that requires removal from therapy (Section 6.0). Therapy may otherwise continue for a maximum of 6 cycles provided the patient meets the criteria for starting subsequent cycles (Section 5.2) and does not meet any of the criteria for removal from protocol therapy criteria (Section 10.0).

A cycle of therapy is considered to be 28 days. A cycle may be repeated for a maximum of 6 cycles.

Drug doses should be adjusted based on the BSA calculated from height and weight measured within 7 days prior to the beginning of each cycle, and according to the dosing nomogram (see <u>Appendix IV</u>).

LY3023414 should be taken without regards to food with a glass of water at approximately the same time each day. Patients should swallow the tablets as a whole and should not chew or crush them.

If a patient misses a dose of LY3023414, the dose should be taken as soon as possible as long as it is more than 6 hours before the next scheduled dose. If it is less than 6 hours before the next dose, then the dose should be skipped. If vomiting occurs after taking LY3023414, the patient should skip the dose and take the next dose as scheduled.

#### 5.1.1 <u>Determination of Recommended Phase 2 Dose (RP2D)/Tolerable Dose</u>

| Dose Level | Dose (mg/m <sup>2</sup> ) |
|------------|---------------------------------|
| -1 | 55 mg/m <sup>2</sup> /dose BID |
| 1* | 80 mg/m²/dose BID |
| 2 | 115 mg/m <sup>2</sup> /dose BID |

Update (Amendment 5A): There were no cycle 1 dose limiting toxicities in the patients enrolled to either dose level 1 or dose level 2 during dose determination. Therefore, the RP2D on this study has been determined to be dose level 2 (115mg/m²/dose BID), and all remaining subjects will enroll at this dose.

The DLT evaluation period for the purpose of dose escalation will be cycle 1 of therapy. Patients enrolled during the determination of the recommended phase 2

CHILDREN'S ONCOLOGY GROUP

dose who are not evaluable for toxicity during cycle 1 at a given dose level will be replaced.

The starting dose will be 80 mg/m²/dose BID (Dose Level 1), which is approximately 30% below the adult MTD. Accrual will be temporarily suspended after enrollment to the first 6 toxicity-evaluable subjects to assess for toxicity as outlined in Section 11.2.

If there are fewer than 2 DLTs in the first 6 toxicity-evaluable subjects enrolled at the starting dose, the dose will be escalated to Dose Level 2. If  $\geq$  2 of the first 6 toxicity-evaluable subjects enrolled at Dose Level 2 have DLTs, all subsequent subjects will be enrolled at the original starting dose. Otherwise, remaining subjects will continue to enroll at Dose Level 2.

If there are 2 or more DLTs during cycle 1 among the first 6 toxicity-evaluable subjects enrolled at Dose Level 1, the next cohort will enroll at Dose Level -1. If  $\geq 2$  of the first 6 toxicity-evaluable subjects enrolled at the reduced dose have DLTs, the study will be closed for toxicity. Otherwise, remaining subjects will continue to enroll at Dose Level -1.

#### **Dose escalation schema:**



#### 5.1.2 Intra-Patient Escalation

Intra-patient dose escalation is not allowed.

#### 5.1.3 Therapy Delivery Map

See Appendix VI for APEC1621D Therapy Delivery Map.



#### 5.2 Criteria for Starting Subsequent Cycles

A cycle may be repeated every 28 days if the patient has at least stable disease and has again met laboratory parameters as defined in the eligibility section, Section 4.0 with the exception of hyperglycemia, hypercholesterolemia, and hypertriglyceridemia, for which the patient may proceed to the next cycle as long as there is not an ongoing dose limiting toxicity as defined in Section 5.4.1.

#### 5.3 Grading of Adverse Events

Adverse events (toxicities) will be graded according to the current version of the NCI Common Terminology Criteria for Adverse Events (CTCAE). All appropriate treatment areas should have access to a copy of the current version of the CTCAE v5.0. A copy of the CTCAE v5.0 can be downloaded from the CTEP website (<a href="http://ctep.cancer.gov">http://ctep.cancer.gov</a>). Any suspected or confirmed dose-limiting toxicity should be reported immediately (within 24 hours) to the Study Chair.

#### 5.4 Definition of Dose-Limiting Toxicity (DLT)

DLT will be defined as any of the following events that are possibly, probably or definitely attributable to protocol therapy. Dose limiting hematological and non-hematological toxicities are defined differently.

#### 5.4.1 Non-Hematological Dose-Limiting Toxicity

- 5.4.1.1 Any Grade 4 or greater non-hematological toxicity attributable to the investigational drug with the specific exclusion of:
  - Grade 4 fever < 5 days duration.
  - Hyperglycemia >500 mg/dL (>27.8 mmol/L) that returns to fasting glucose value ≤ 250 mg/dL (13.9 mmol/L) within 24 hours of initiation of appropriate supportive care as per Section 7.3.4. The severity (grade) of hyperglycemia is based upon fasting levels. If glucose >500 mg/dL (>27.8 mmol/L) is detected when routine (non-fasting) laboratory studies are performed, the test should be repeated within 24 hours in the fasting state to permit accurate grading.
  - Grade 4 hypercholesterolemia that returns to ≤ Grade 2 within 35 days of initiation of appropriate supportive care as per Section 7.3.6. The severity (grade) of hypercholesterolemia is based upon fasting levels. If Grade 4 hypercholesterolemia is detected when routine (non-fasting) laboratory studies are performed, the test should be repeated within 3 days in the fasting state to permit accurate grading.
- 5.4.1.2 Any Grade 3 non-hematological toxicity attributable to the investigational drug with the specific exclusion of:
  - Nausea, vomiting, diarrhea, constipation, or anorexia of  $\leq 3$  days duration
  - Fatigue that resolves to  $\leq$  Grade 2 within 7 days
  - Oral or pharyngeal mucositis or stomatitis ≤ 7 days duration
  - Liver enzyme elevation, including ALT/AST/GGT that returns to levels that meet initial eligibility criteria or baseline within 7 days. See <u>Appendix X</u> for values that represent thresholds between CTCAE grades.
     <u>Note</u>: For the purposes of this study the ULN for ALT is defined as 45 U/L regardless of baseline.
  - Fever < 5 days duration.
  - Infection < 5 days duration.

- Hypophosphatemia, hypokalemia, hypocalcemia or hypomagnesemia responsive to supplementation.

- Hyperglycemia that returns to fasting glucose value ≤ 250 mg/dL (13.9 mmol/L) (with or without the use of insulin or oral diabetic agents) within 7 days of initiation of appropriate supportive care as per Section 7.3.4. The severity (grade) of hyperglycemia is based upon fasting levels. If glucose in the range >250 500 mg/dL; (>13.9 27.8 mmol/L) is detected when routine (non-fasting) laboratory studies are performed, the test should be repeated within 3 days in the fasting state to permit accurate grading.
- Hypertriglyceridemia that returns to Grade ≤ 2 within 14 days of initiation of appropriate supportive care as per Section 7.3.5. The severity (grade) of hypertriglyceridemia is based upon fasting levels. If Grade 3 triglycerides are detected when routine (non-fasting) laboratory studies are performed, the test should be repeated within 3 days in the fasting state to permit accurate grading.
- Hypercholesterolemia that returns to ≤ Grade 2 within 35 days of initiation of appropriate supportive care as per Section 7.3.6. The severity (grade) of hypercholesterolemia is based upon fasting levels. If Grade 3 hypercholesterolemia is detected when routine (non-fasting) laboratory studies are performed, the test should be repeated within 3 days in the fasting state to permit accurate grading.
- Papulopustular, acneiform, or maculo-papular rash that resolves to < Grade 2 or baseline within 14 days of appropriate supportive care as per <a href="Section 7.3.2">Section 7.3.2</a>. However, any investigational drug-related grade 3 rash that is considered intolerable by the patient or limits ADLs will be considered a DLT regardless of duration.
- 5.4.1.3 Any Grade 2 non-hematological toxicity that persists for  $\geq 7$  days and is considered sufficiently medically significant or sufficiently intolerable by patients that it requires treatment interruption.
- Note: Allergic reactions that necessitate discontinuation of study drug will not be considered a dose-limiting toxicity.

#### 5.4.2 <u>Hematological dose limiting toxicity</u>

- 5.4.2.1 Hematological dose limiting toxicity is defined as:
- a) In patients evaluable for hematological toxicity (see Section 4.1.7.1),
  - Grade 4 thrombocytopenia or neutropenia, not due to malignant infiltration.
  - Grade 3 thrombocytopenia that persists for  $\geq 7$  days
  - Grade 3 thrombocytopenia requiring a platelet transfusion on two separate days within a 7-day period
  - Grade 3 thrombocytopenia with clinically significant bleeding
  - Neutropenia or thrombocytopenia that causes a delay of > 14 days between treatment cycles.
- 5.4.2.2 <u>Note</u>: Grade 3 or 4 febrile neutropenia will not be considered a dose-limiting toxicity.



#### 6.0 **DOSE MODIFICATIONS FOR ADVERSE EVENTS**

The Study Chair must be notified of any dosage modification or use of myeloid growth factor.

#### 6.1 Dose Modifications for Hematological Toxicity

- 6.1.1 If a patient experiences hematological dose-limiting toxicity as defined in Section 5.4.2, the treatment will be held. Counts should be checked every 3-4 days for thrombocytopenia and every other day for neutropenia during this time. If the toxicity resolves to meet meet eligibility parameters within 14 days of drug discontinuation, the patient may resume treatment at a reduced dose as outlined in the dose reduction table (Appendix IV). Doses reduced for toxicity will not be re-escalated, even if there is minimal or no toxicity with the reduced dose.
- 6.1.2 If toxicity does not resolve to meet eligibility parameters within 14 days of drug discontinuation, the patient must be removed from protocol therapy.
- 6.1.3 If hematological dose-limiting toxicity recurs in a patient who has resumed treatment at the reduced dose, the patient must be removed from protocol therapy.

#### 6.2 Dose Modifications for Non-Hematological Toxicity

- 6.2.1 If a patient experiences non-hematological dose-limiting toxicity as defined in Section 5.4.1, the treatment will be held. When the toxicity resolves such that there is no ongoing DLT of hyperglycemia, hypercholesterolemia, and hypertriglyceridemia as defined in Section 5.4.1 and other laboratory values meet eligibility parameters or baseline within 14 days of drug discontinuation, the patient may resume treatment at a reduced dose as outlined in the dose reduction table (Appendix IV). Doses reduced for toxicity will not be reescalated, even if there is minimal or no toxicity with the reduced dose.
- 6.2.2 If toxicity does not resolve such that there is no ongoing DLT of hyperglycemia, hypercholesterolemia, and hypertriglyceridemia as defined in <u>Section 5.4.1</u> and other laboratory values meet eligibility parameters or baseline within 14 days of drug discontinuation, the patient must be removed from protocol therapy.
- 6.2.3 If dose-limiting toxicity recurs in a patient who has resumed treatment at the reduced dose, the patient must be removed from protocol therapy.
- 6.2.4 If a patient experiences a Grade 2 or greater allergic reaction to LY3023414, the patient will be removed from protocol therapy.



#### 7.0 SUPPORTIVE CARE AND OTHER CONCOMITANT THERAPY

#### 7.1 Concurrent Anticancer Therapy

Concurrent cancer therapy, including chemotherapy, radiation therapy, immunotherapy, or biologic therapy may NOT be administered to patients receiving study drug. If these treatments are administered the patient will be removed from protocol therapy.

#### 7.2 Investigational Agents

No other investigational agents may be given while the patient is on study.

#### 7.3 Supportive Care

Appropriate antibiotics, blood products, antiemetics, fluids, electrolytes and general supportive care are to be used as necessary. See Section 7.5 for drugs that should not be used concomitantly due to potential interactions with LY3023414. See below for recommendations on management of specific toxicities associated with LY3023414.

#### 7.3.1 Nausea and vomiting:

Nausea and vomiting has been observed frequently in adult patients treated with LY3023414. It is recommended to provide all patients a 5-HT<sub>3</sub>-Receptor blocker (eg, ondansetron or granisetron) at the start of treatment to be used as needed or prophylactically. In the event of breakthrough nausea/vomiting, additional antiemetics may be added as needed.

#### 7.3.2 **Rash**:

Rashes which can be pruritic have been observed in frequently in adult patients treated with LY3023414. For all patients, prophylactic measures should be considered including the use of sunscreen prior to any sun-exposure and application of thick emollient cream to dry areas of the body at least twice daily. For grade 1 rash, mild-moderate potency topical steroids and oral antihistamines (if pruritic) should be considered. For grade 2 rash, moderate potency topical steroids and oral antihistamines (if pruritic) are recommended. For grade 3 rash, moderate potency topical steroids should be applied at least twice daily and oral antihistamines should be used if the rash is pruritic. Patients with a grade 3 or worse rash should have a physical exam at least weekly until improvement to grade ≤ 2. As per section 5.4.1.1, any grade 3 rash that is intolerable, limiting ADLs, or that persists for > 14 days after initiation of topical steroid therapy will be considered a dose limiting toxicity. LY3023414 will be held and moderate potency topical steroids will be applied at least twice daily and a course of systemic steroid should be strongly considered with oral antihistamines given as needed for pruritis.

#### 7.3.3 **Mucositis:**

Mucositis has been observed in adult patients treated with LY3023414. For grade 1 mucositis, it is recommended to use conservative measures such as non-alcoholic mouth wash or salt water (0.9%) mouth wash several times a day until resolution. For grade  $\geq 2$  mucositis, topical analgesic mouth treatments (i.e., local anesthetics such as benzocaine, butyl aminobenzoate, tetracaine hydrochloride, menthol, or phenol) may be used with or without topical corticosteroids, such as triamcinolone oral paste 0.1% (e.g. Kenalog in Orabase®). Agents containing hydrogen peroxide, iodine, and thyme derivatives may worsen mouth ulcers and should not be used.

Systemic antifungal agents should be avoided unless a fungal infection is diagnosed.

This protocol is for research purposes only, see page 1 for usage policy. APEC1621D

In particular, systemic imidazole antifungal agents (ketoconazole, fluconazole, itraconazole, etc.) should be avoided due to their strong inhibition of CYP3A4 metabolism, therefore leading to higher LY3023414 exposure. Topical antifungal agents are preferred if an infection is diagnosed.

#### 7.3.4 **Hyperglycemia:**

The world's childhood

Hyperglycemia has been observed in adults treated with LY3023414. **Initiation of treatment for hyperglycemia should occur under the guidance of a pediatric endocrinologist at the local institution.** Metformin or other oral antihyperglycemia agent may be used per local endocrinologist's recommendations. Insulin therapy should be directed by specialists in pediatric diabetes, with the goal of normal fasting blood sugars < 126 mg/dL and HgbA1C < 8%.

For fasting glucose value ≤ 160 mg/dL (8.9 mmol/L), conservative measures are recommended (dietary modification). For fasting glucose value >160 - \le 250 mgdL  $(>8.9 - \le 13.9 \text{ mmol/L})$ , consultation with an endocrinologist and consideration of initiation of an oral anti-diabetic agent is recommended. Insulin therapy should be considered if treatment with an oral anti-diabetic is insufficient. For glucose in the range >250 - 500 mg/dL; (>13.9 - 27.8 mmol/L) or glucose >500 mg/dL (>27.8 mmol/L) persisting less than 24 hours, insulin or an oral anti-diabetic agent should be started in consultation with an endocrinologist. Patients with glucose in the range >250 - 500 mg/dL; (>13.9 - 27.8 mmol/L) or worse hyperglycemia should have fasting glucose checked at least twice weekly until resolution to less than or equal to a fasting glucose value  $\leq 250 \text{ mg/dL}$  (13.9 mmol/L). Glucose in the range  $\geq 250 \text{ --}$ 500 mg/dL; (>13.9 - 27.8 mmol/L) persisting for more than 7 days after starting an oral antidiabetic agent and glucose >500 mg/dL (>27.8 mmol/L) persisting for more than 24 hours after starting an oral antidiabetic agent are a dose limiting toxicities. LY3023414 will be held and the patient will be treated with insulin or an oral antidiabetic agent in consultation with an endocrinologist.

#### 7.3.5 **Hypertriglyceridemia:**

Hypertriglyceridemia has been observed in patients treated with mTOR inhibitors. Initiation of treatment for hypertriglyceridemia should occur under the guidance of pediatric specialists with expertise in lipid disorders at the local institution.

For grade 2 hypertriglyceridemia, consultation with a pediatric specialist with expertise in lipid disorders and consideration of initiation of an HMG-CoA reductase inhibitor is recommended. For grade 3 hypertriglyceridemia, an HMG-CoA reductase inhibitor should be started in consultation with a pediatric specialist with expertise in lipid disorders. Patients with grade 3 or worse hypertriglyceridemia should have fasting triglycerides checked at least weekly until resolution to ≤ grade 2. Grade 3 hypertriglyceridemia persisting for more than 14 days after starting an HMG-CoA reductase inhibitor and any grade 4 hypertriglyceridemia are a dose limiting toxicities. LY3023414 will be held and the patient will be treated with an HMG-CoA reductase inhibitor in consultation with a pediatric specialist with expertise in lipid disorders.

#### 7.3.6 **Hypercholesterolemia:**

Hypercholesterolemia has been observed in patients treated with mTOR inhibitors. Initiation of treatment for hypercholesterolemia should occur under the


# guidance of pediatric specialists with expertise in lipid disorders at the local institution.

For grade 2 hypercholesterolemia, consultation with a pediatric specialist with expertise in lipid disorders and consideration of initiation of an HMG-CoA reductase inhibitor is recommended. For grade 3 or 4 hypercholesterolemia, an HMG-CoA reductase inhibitor should be started in consultation with a pediatric specialist with expertise in lipid disorders. Patients with grade 3 or worse hypercholesterolemia should have fasting cholesterol checked at least every other week until resolution to  $\leq$  grade 2. Grade 3 or 4 hypercholesterolemia persisting for more than 35 days after starting an HMG-CoA reductase inhibitor is a dose limiting toxicity. LY3023414 will be held and the patient will be treated with an HMG-CoA reductase inhibitor in consultation with a pediatric specialist with expertise in lipid disorders.

#### 7.4 Growth Factors

Growth factors that support platelet or white cell number or function can only be administered for culture proven bacteremia or invasive fungal infection. The Study Chair should be notified before growth factors are initiated.

#### 7.5 Concomitant Medications

#### 7.5.1 CYP3A4 substrates, inhibitors or inducers:

In vitro data showed that LY3023414 is a substrate of CYP3A4 and CYP1A2 (to a lesser extent). Therefore, moderate to strong inducers and strong inhibitors of CYP3A4 should be substituted or avoided, if possible. (See Appendix II). However, in patients for whom there are no adequate therapeutic alternatives, CYP3A4 inducing anti-epileptic drugs and dexamethasone for CNS tumors or metastases, on a stable dose, are allowed.

LY3023414 is a weak inhibitor of CYP3A4. Monitor patients receiving drugs that are either sensitive substrates of CYP3A4 or CYP3A4 substrates with a narrow therapeutic range.

7.5.2 Strong inducers (eg., smoking) and inhibitors (eg., ciprofloxacin, enoxacin, fluvoxamine, zafirlukast) of CYP1A2 should also be avoided if possible while receiving protocol therapy.



#### 8.0 EVALUATIONS/MATERIAL AND DATA TO BE ACCESSIONED

## 8.1 Required Clinical, Laboratory and Disease Evaluation

All clinical and laboratory studies to determine eligibility must be performed within 7 days prior to enrollment unless otherwise indicated. Laboratory values used to assess eligibility (see Section 4.0) must be no older than seven (7) days at the start of therapy. Laboratory tests need **not** be repeated if therapy starts **within** seven (7) days of obtaining labs to assess eligibility. If a post-enrollment lab value is outside the limits of eligibility, or laboratory values are older than 7 days, then the following laboratory evaluations must be re-checked within 48 hours prior to initiating therapy: CBC with differential, bilirubin, ALT (SGPT) and serum creatinine. If the recheck is outside the limits of eligibility, the patient may not receive protocol therapy and will be considered off protocol therapy. Imaging studies, bone marrow aspirate and/or biopsy, must be obtained within 14 days prior to start of protocol therapy (repeat the tumor imaging if necessary).

| STUDIES TO BE OBTAINED | Pre-<br>Study | During Cycle 1 | Prior to Subsequent<br>Cycles^ |
|---|---|---|---|
| History | X | Weekly | X |
| Physical Exam with vital signs | X | Weekly | X |
| Neurologic Exam | X | Weekly | X |
| Height, weight, BSA | X | | X |
| Performance Status | X | | |
| Pregnancy Test <sup>1</sup> | X | | |
| CBC, differential, platelets | X | Twice Weekly (every 3 to 4 days) <sup>2</sup> | Weekly <sup>3</sup> |
| Urinalysis | X | | |
| Electrolytes including Ca <sup>++</sup> , PO <sub>4</sub> , Mg <sup>++</sup> | X | Weekly | X |
| Creatinine, ALT, bilirubin | X | Weekly | X |
| Glucose | X | Weekly | X |
| Albumin | X | | X |
| Total cholesterol, triglycerides | X | | X |
| Tumor Disease Evaluation <sup>4A</sup> | X | | Every other cycle <sup>4</sup> |
| Bone Marrow Aspirate and/or biopsy <sup>5,6</sup> | $X^5$ | | Every other cycle <sup>6</sup> |
| EKG | X | | |
| Medication Diary <sup>7</sup> | | Weekly | X |
| Pharmacokinetics (optional) <sup>8</sup> | X | X | |
| Circulating Tumor DNA (ctDNA- | | | Cycle 5, Day 1 and |
| optional) <sup>9</sup> | | | (for patients receiving |
| | | | $\geq$ 5 cycles only) at |
| | | | end of protocol |
| | | | therapy OR disease |
| | | | progression |

Studies may be obtained within 72 hours prior to the start of the subsequent cycle.

Women of childbearing potential require a negative pregnancy test prior to starting treatment; sexually active patients must use an acceptable method of birth control. Abstinence is an acceptable method of birth control.

<sup>&</sup>lt;sup>2</sup> If patients have Grade 4 neutropenia then CBCs should be checked at least every other day until recovery to Grade 3 or until meeting the criteria for dose limiting toxicity.

<sup>&</sup>lt;sup>3</sup> If patients develop Grade 4 neutropenia then CBCs should be checked every 3 to 4 days until recovery to Grade 3

<sup>&</sup>lt;sup>4A</sup> Neurological exam also required for CNS patients.



- Tumor Disease Evaluation should be obtained on the next consecutive cycle after initial documentation of either a PR or CR. Subsequent scans may restart 2 cycles after the confirmatory scan. If the institutional investigator determines that the patient has progressed based on clinical or laboratory evidence, he/she may opt not to confirm this finding radiographically.
- Bone marrow aspirate and/or biopsy only required in patients suspected of having bone marrow metastasis on the basis of history, symptoms, laboratory evaluation or other clinical data.
- Bone marrow aspirate and/or biopsy should only be performed on patients with known bone marrow involvement at baseline
- Patient diary (see <u>Appendix III</u>) should be reviewed after completion of each treatment cycle and uploaded into RAVE.
- 8 See Section 8.3 for details of PK studies.
- With consent, two samples will be collected on this protocol (cycle 5 Day 1; and for patients receiving ≥ 5 cycles only: at progession or end of protocol therapy) see Section 8.4 for details of the ctDNA studies. Note that a ctDNA sample is scheduled to be obtained on the APEC1621SC screening protocol prior to the intiation of treatment on this subprotocol.

## 8.2 Radiology Studies

8.2.1 <u>Central Radiology Review for Response:</u> Patients who respond (CR, PR) to therapy or have long term stable disease (SD) (6 cycles) on protocol therapy will be centrally reviewed.

## 8.2.2 Technical Details of Submission:

To ensure an adequate interpretation of FDG-PET and CT with contrast scans, scans transferred between the treating institutions and the Imaging and Radiation Oncology Core Group IROC RI (QARC) must be submitted in Digital Imaging and Communications in Medicine (DICOM) format. BMP files, JPG files, or hard copies (films) are unacceptable for adequate interpretation of PET and CT with contrast scans. Imaging studies must be submitted electronically as outlined in the following paragraph. The images will be made available to study radiologists and nuclear medicine physicians for central review.

Submission of Diagnostic Imaging data in digital format is required. Digital files must be in DICOM format. Due to the critical time constraints for submitting data for the central review of response the following methods should be used to submit imaging data, such as sFTP, Dicommunicator, or on CD (if sent by courier). Digital data submission instructions including instructions for obtaining a sFTP account, can be found at http://irocri.qarc.org. Follow the link labeled digital data. Alternatively, if submission via sFTP or Dicommunicator is not feasible, the imaging may be burned to a CD and mailed to IROC RI (QARC) at the address below. Multiple studies for the same patient may be submitted on one CD; however, please submit only one patient per CD. Sites using Dicommunicator may submit imaging via that application. Contact IROC RI (QARC) with questions or for additional information.

For FDG-PET imaging, the transferred imaging data should include uncorrected and attenuation-corrected PET projection data, as well as the reconstructed PET or PET/CT images used by the institution to achieve a response assessment. If low-dose CT was used for attenuation correction, the acquired CT images should also be submitted. The imaging data submitted for central review must allow the study to be reconstructed and displayed in transaxial, sagittal and coronal formats using



This protocol is for research purposes only, see page 1 for usage policy. APEC1621D

standard reconstruction techniques. Reconstructed MPEG clips and similar types of reconstructions will not be accepted. CT and MRI images similarly should be submitted in a format that either includes properly reconstructed multi-planar viewing formats in soft tissue and bone windows, or includes the thin-section axial acquisition data from which multi-planar reconstructions can be re-created.

Address for submission: IROC RI (QARC)

Building B, Suite 201

640 George Washington Highway Lincoln, RI 02865-4207

Phone: (401) 753-7600 (401) 753-7601 Fax: Web: http://irocri.garc.org

#### 8.3 Pharmacology (optional)

#### 8.3.1 Description of Studies and Assay

Pharmacokinetics (PK) will be performed to determine the PK of LY3023414 in children who consent to this optional study. Pharmacokinetic analysis will be conducted at a centralized laboratory using validated assays.

#### 8.3.2 Sampling Schedule

Blood samples will be obtained at the following time points for ALL patients enrolled on study who consent to optional pharmacokinetics:

<u>Day 15, Cycle 1</u>: Pre-dose (12 hours after the PM dose on Day 14, Cycle 1) and at 1-2 hours after the AM dose on Day 15.

Determination of the recommended phase 2 dose is complete. Blood samples will were obtained at the following time points ONLY for patients enrolled during the determination of the recommended phase 2 dose / tolerable dose (Section **5.1.1)** who consented to optional pharmacokinetics

- Day 1, Cycle 1: Pre-dose, and at 30 minutes, 1, 2, 4, 6-8 hours after the AM dose on Day 1. The PM dose of LY3023414 on Day 1, Cycle 1 will not be given for patients undergoing these PK studies.
- Day 2, Cycle 1: Before the AM dose on Day 2 (24 hours after the AM dose on Day 1, Cycle 1).

#### 8.3.3 Sample Collection and Handling Instructions

Blood samples (2 ml for each time point) will be collected in K<sub>2</sub>-EDTA (lavender top) tubes for pharmacokinetic evaluation. Record the exact time that the sample is drawn along with the exact time that the drug is administered.

Sites are expected to use their own standard materials for PK sample collection as kits will not be provided for the PK samples for this study.

#### 8.3.4 Sample Processing

Following collection, the sample will be immediately gently mixed by inversion 8-10 times. The sample will be stored on wet ice until centrifugation. The sample will be centrifuged at 1500 x g for 15 minutes at 4° C within 60 minutes



after the sample is drawn. The plasma will be transferred to a cryovial, ensuring no RBC contamination, and frozen as soon as possible at -80° C. If a -80° C freezer is not immediately available, the cryovial may be stored on dry ice for short term storage, but must be placed in the appropriate freezer within 24 hours of the draw-time.

## 8.3.5 Sample Labeling

Each sample must be labeled with the patient's study registration number, the study I.D# (APEC1621D), and the date and time the sample was drawn. Data should be recorded on the appropriate transmittal form found in RAVE, which must accompany the sample(s).

## 8.3.6 <u>Sample Shipping Instructions</u>

Samples will be shipped on dry-ice to Covance Laboratories at the address below. Samples may be batched, but should be shipped within 1 month of draw.



A notification email should be sent to Mohammad Koupaei with courier name, airway bill number, expected delivery date/time and shipment contact.

## 8.4 Circulating Tumor DNA Study (optional)

#### 8.4.1 Sampling Schedule

An initial sample was previously requested at time of enrollment into the APEC1621SC screening protocol. Additional samples (optional) will be collected into Streck Cell-Free DNA BCT tubes at the following timepoints:

- (1) Cycle 5 Day 1
- (2) At disease progression or end of protocol therapy (for patients receiving  $\geq 5$  cycles of therapy only)

Peripheral blood samples for circulating tumor DNA should be obtained as follows:

- For patients  $\geq 10 \text{ kg collect } 20 \text{ mLs } (10 \text{ mL per tube x 2 tubes})$
- For patients  $\geq 5$  kg but < 10 kg collect 10 mL (one tube)
- For patients < 5 kg research samples will not be collected

In all cases, blood draw volumes should strictly adhere to institutional limitations, taking other blood draws into consideration. However, if a reduction in volume is required, samples should be collected in 10 mL increments (ie. 0, 10, or 20 mL should be collected such that each Streck Cell-Free DNA BCT is completely filled).

Established institutional guidelines should be followed for blood collection via

Version Date: 10/28/2022

CHILDREN'S

ONCOLOGY

**GROUP** 

vascular access devices. Heparin should be avoided in pre-collection flush procedures. If therapeutic heparin dosing contamination is a possibility, venipuncture is recommended as a first choice collection method. If a Streck Cell-Free DNA BCT tube immediately follows a heparin tube in the draw order, we recommend collecting an EDTA tube as a waste tube prior to collection in the Streck Cell-Free DNA BCT.

For patients who do not have indwelling catheters, blood should be collected via venipuncture. To guard against backflow, observe the following precautions:

- Keep patient's arm in the downward position during the collection procedure.
- Hold the tube with the stopper in the uppermost position so that the tube contents do not touch the stopper or the end of the needle during sample collection.
- Release tourniquet once blood starts to flow in the tube, or within 2 minutes of application.
- Fill tube completely.
- Remove tube from adapter and immediately mix by gentle inversion 8 to 10 times. Inadequate or delayed mixing may result in inaccurate test
- Store blood in Streck tube at **room temperature** until shipment

#### 8.4.2 Sample Processing

Samples do not need to be processed at the collection site.

#### 8.4.3 Sample Labeling

Each tube must be labeled with the patient's study registration number, the study I.D (APEC1621D), and the date and time the sample was drawn. Data should be recorded on the appropriate transmittal form found in RAVE, which must accompany the sample(s).

#### 8.4.4 Sample Shipping Instructions

Specimen should be shipped at room temperature to the BPC (address below). Upon arrival separation, extraction, and storage of plasma and cellular DNA will be performed. Samples should be shipped from Monday through Friday for Tuesday through Saturday delivery. If blood is collected in the Streck tube on Friday, over the weekend or on the day before a holiday, the sample can be stored at room temperature until shipped on the next business day.

Ship specimens to the following address:

Biopathology Center Nationwide Children's Hospital Protocol APEC1621D- Peds MATCH\* 700 Children's Drive, WA1340 Columbus, OH 43205

Phone: (614) 722-2865 Fax: (614) 722-2897

Email:BPCBank@nationwidechildrens.org

<sup>\*</sup>Labeling is extremely important for this project. Packages must be labeled "Peds

MATCH" in order to expedite processing at the BPC. Be sure to include the room number. Packages received without the room number may be returned to the sender

Ship samples by FedEx Priority Overnight using a FedEx shipping label obtained through the COG FedEx account. Ship blood for Saturday delivery if shipped on Friday.

# 9.0 **AGENT INFORMATION**

9,1 LY3023414 11/12/2021

NSC# 783668 IND#134661

## 9.1.1 Structure and molecular weight

LY3023414 is an orally available, potent, selective inhibitor of the class I PI3K isoforms, mTOR, and DNA-PK. LY3023414 binds the adenosine triphosphate (ATP) active site of PI3K to competitively inhibit phosphorylation of phosphatidylinositol-4,5-bisphosphate (PIP2) at low nanomolar concentrations. LY3023414 has inhibitory activity against PI3K/mTOR pathway targets in vitro and in vivo. LY3023414 has antiproliferative and cell cycle-arresting effects in cultured cancer cells and antiangiogenesis activity via inhibition of in vitro vascular cord formation.

LY3023414 is a small molecule with an empirical formula of  $C_{23}H_{26}N_4O_3$  and a molecular weight of 406.48. The chemical structure is:

9.1.2 <u>Supplied by:</u> Eli Lilly and Company and distributed by the Pharmaceutical Management Branch, CTEP, DCTD, NCI.

## 9.1.3 Formulation

LY3023414 is supplied for clinical trial use as 50-mg and 100-mg film-coated tablets. The 50-mg tablets are green, modified, capsule-shaped tablets. The 100-mg tablets are dark yellow, modified, capsule-shaped tablets. The tablets are composed of active drug ingredient, microcrystalline cellulose, croscarmellose sodium, silicon dioxide, sodium stearyl fumarate and colorant. Tablets are available in 60-count bottles with desiccant.

9.1.4 <u>Storage</u>: Store intact bottles at controlled room temperature between 15° C to 30° C (59° F to 86° F) according to label.

If a storage temperature excursion is identified, promptly return LY3023414 to controlled room temperature and quarantine the supplies. Provide a detailed report of the excursion (including documentation of temperature monitoring and duration of the excursion) to <a href="mailto:PMBAfterHours@mail.nih.gov">PMBAfterHours@mail.nih.gov</a> for determination of suitability.

## 9.1.5 Stability

Stability studies are ongoing. The manufacturer does not have stability data to support repackaging tablets. Dispense tablets in the original container.

#### 9.1.6 Administration

See Treatment section of the protocol for dosing and administration details. LY3023414 is administered orally.

LY3023414 should be taken without regards to food with a glass of water at approximately the same time each day. Patients should swallow the tablets as a whole and should not chew, dissolve or crush them.

If a patient misses a dose of LY3023414, the dose should be taken as soon as possible as long as it is more than 6 hours before the next scheduled dose. If it is less than 6 hours before the next dose, then the dose should be skipped. If vomiting occurs after taking LY3023414, the patient should skip the dose and take the next dose as scheduled.

## 9.1.7 Potential Drug Interactions

LY3023414 is a weak inhibitor of CYP3A4, based on the increase in midazolam exposure observed after concomitant administration. Therefore, drugs that are either sensitive substrates of CYP3A4 or CYP3A4 substrates with a narrow therapeutic range should be administered with caution in combination with LY3023414.

In vitro data showed that the major enzymes involved in the clearance of LY3023414 were CYP3A (82%), and CYP1A2 (18%). Therefore, it is recommended to avoid moderate to strong inducers and strong inhibitors of CYP3A4. Note: In patients for whom there are no adequate therapeutic alternatives, CYP3A4 inducing anti-epileptic drugs and dexamethasone for CNS tumors or metastases, on a stable dose, are allowed. Strong inducers and inhibitors of CYP1A2 should also be avoided if possible while receiving protocol therapy.

LY3023414 is a substrate for both P-glycoprotein and BCRP; however, current information suggests these transporters appear unlikely to affect oral absorption of agent to any great extent.

#### 9.1.8 Patient Care Considerations

Females and males of reproductive potential should be advised to avoid becoming pregnant or fathering a child during therapy with LY3023414. Both males and females of reproductive potential must agree to use medically approved contraceptive precautions during the study and for at least 3 months following the last dose of the study drug. Women choosing to breastfeed their infants should not take LY3023414.



## 9.1.9 LY3023414 Toxicities

The Comprehensive Adverse Events and Potential Risks list (CAEPR) provides a single list of reported and/or potential adverse events (AE) associated with an agent using a uniform presentation of events by body system. In addition to the comprehensive list, a subset, the Specific Protocol Exceptions to Expedited Reporting (SPEER), appears in a separate column and is identified with bold and italicized text. This subset of AEs (SPEER) is a list of events that are protocol specific exceptions to expedited reporting to NCI (except as noted below). Refer to the 'CTEP, NCI Guidelines: Adverse Event Reporting Requirements' <a href="http://ctep.cancer.gov/protocolDevelopment/electronic applications/docs/aeguidelines.pdf">http://ctep.cancer.gov/protocolDevelopment/electronic applications/docs/aeguidelines.pdf</a> for further clarification. *Frequency is provided based on 165 patients*. Below is the CAEPR for LY3023414.

**NOTE**: Report AEs on the SPEER **ONLY IF** they exceed the grade noted in parentheses next to the AE in the SPEER. If this CAEPR is part of a combination protocol using multiple investigational agents and has an AE listed on different SPEERs, use the lower of the grades to determine if expedited reporting is required.

Version 2.4, January 8, 2021<sup>59</sup>

| Likely (>20%) | Adverse Events with Possible Relationship to LY3023414 (CTCAE 5.0 Term) [n= 165] Likely (>20%) Less Likely (<=20%) Rare but Serious (<3%) | | | |
|---|---|---|---|---|
| BLOOD AND LYMPHATIC SY | | Naie but Serious ( | 3 /0) | |
| | Anemia | | | Anemia (Gr 2) |
| GASTROINTESTINAL DISOR | | | | (01.0) |
| | Abdominal pain | | | |
| | Constipation | | | |
| Diarrhea | | | | Diarrhea (Gr 2) |
| | Gastroesophageal reflux disease | | | |
| | Mucositis oral | | | Mucositis oral (Gr 2) |
| Nausea | | | | Nausea (Gr 2) |
| | Oral dysesthesia | | | Oral dysesthesia (Gr 2) |
| Vomiting | | | | Vomiting (Gr 2) |
| | ADMINISTRATION SITE CON | DITIONS | | |
| Fatigue | | | | Fatigue (Gr 2) |
| | Fever | | | |
| | General disorders and<br>administration site conditions -<br>Other (mucosal inflammation) | | | |
| INFECTIONS AND INFESTAT | TIONS | | | |
| | | Lung infection <sup>2</sup> | | |
| INVESTIGATIONS | | | | |
| | Alanine aminotransferase increased | | | |
| | Aspartate aminotransferase increased | | | |
| | Creatinine increased | | | |
| | | Electrocardiogram QT interval prolonged | corrected | |
| | Platelet count decreased | | | |



| Adverse Events with Possible Relationship to LY3023414 (CTCAE 5.0 Term) [n= 165] | | | Specific Protocol Exceptions<br>to Expedited Reporting<br>(SPEER) |
|---|---|---|---|
| <b>Likely (&gt;20%)</b> | Less Likely (<=20%) | Rare but Serious (<3%) | |
| | Weight loss | | |
| METABOLISM AND NUTF | RITION DISORDERS | | |
| Anorexia | | | Anorexia (Gr 2) |
| | Hyperglycemia | | |
| | Hypokalemia | | |
| | Hyponatremia | | |
| | Hypophosphatemia | | |
| NERVOUS SYSTEM DISO | RDERS | | |
| | Dizziness | | Dizziness (Gr 2) |
| | Dysgeusia | | |
| | Headache | | |
| | Paresthesia | | |
| RESPIRATORY, THORACI | C AND MEDIASTINAL DISORDE | RS | |
| | Dyspnea | | |
| SKIN AND SUBCUTANEO | | | |
| | Dry skin | | |
| | Pruritus | | |
| | Rash maculo-papular | | Rash maculo-papular (Gr 2) |

<sup>&</sup>lt;sup>1</sup> This table will be updated as the toxicity profile of the agent is revised. Updates will be distributed to all Principal Investigators at the time of revision. The current version can be obtained by contacting <u>PIO@CTEP.NCI.NIH.GOV</u>. Your name, the name of the investigator, the protocol and the agent should be included in the e-mail.

Adverse events reported on LY3023414 trials, but for which there is insufficient evidence to suggest that there was a reasonable possibility that LY3023414 caused the adverse event:

**CARDIAC DISORDERS** - Heart failure

GASTROINTESTINAL DISORDERS - Dry mouth; Dyspepsia

GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS - Chills; Edema limbs

**INFECTIONS AND INFESTATIONS - Conjunctivitis** 

INVESTIGATIONS - Blood bilirubin increased; Lymphocyte count decreased; Neutrophil count decreased; White blood cell decreased

**METABOLISM AND NUTRITION DISORDERS** - Dehydration; Hyperkalemia; Hypertriglyceridemia; Hypomagnesemia

**RENAL AND URINARY DISORDERS** - Proteinuria

**RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS** - Cough; Pneumonitis; Respiratory, thoracic and mediastinal disorders - Other (drug-induced lung injury)

SKIN AND SUBCUTANEOUS TISSUE DISORDERS - Alopecia; Rash acneiform

VASCULAR DISORDERS - Hypotension

**Note**: LY3023414 in combination with other agents could cause an exacerbation of any adverse event currently known to be caused by the other agent, or the combination may result in events never previously associated with either agent.

<sup>&</sup>lt;sup>2</sup> Lung infection may be more likely in children that have had lung radiation therapy.



# 9.1.10 Agent Ordering and Agent Accountability

The CTEP assigned protocol number must be used for ordering all CTEP supplied investigational agents. The responsible investigator at each participating institution must be registered with CTEP, DCTD through an annual submission of FDA form 1572 (Statement of Investigator), NCI Biosketch, Agent Shipment Form, and Financial Disclosure Form (FDF). If there are several participating investigators at one institution, CTEP supplied investigational agents for the study should be ordered under the name of one lead participating investigator at that institution.

Note: No starter supplies will be provided. Drug orders of LY3023414 should be placed with CTEP after enrollment and treatment assignment to APEC1621D with consideration for timing of processing and shipping to ensure receipt of drug supply prior to start of protocol therapy. If expedited shipment is required, sites should provide an express courier account through the Online Agent Order Processing (OAOP) application. Provide the patient ID number in the comment box when submitting an order request.

## 9.1.11 Clinical Drug Request

Submit agent requests through the PMB Online Agent Order Processing (OAOP) application. Access to OAOP requires the establishment of a CTEP Identity and Access Management (IAM) account and the maintenance of an "active" account status, a "current" password and active person registration status. For questions about drug orders, transfers, returns, or accountability call or email PMB anytime. Refer to the PMB's website for specific policies and guidelines related to agent management.

## 9.1.12 Agent Inventory Records

The investigator, or a responsible party designated by the investigator, must maintain a careful record of the receipt, dispensing and final disposition of all agents received from the PMB using the appropriate NCI Investigational Agent (Drug) Accountability Record (DARF) available on the CTEP forms page. Store and maintain separate NCI Investigational Agent Accountability Records for each agent, strength, formulation and ordering investigator on this protocol.

# 9.1.13 <u>Useful Links and Contacts</u>

• CTEP Forms, Templates, Documents:

http://ctep.cancer.gov/forms/

• NCI CTEP Registration:

RCRHelpDesk@nih.gov

PMB policies and guidelines:

http://ctep.cancer.gov/branches/pmb/agent management.htm

• PMB Online Agent Order Processing (OAOP) application:

https://ctepcore.nci.nih.gov/OAOP/

• CTEP Identity and Access Management (IAM) account:

https://ctepcore.nci.nih.gov/iam/

| • | PP | | etepeore.ner | <u></u> | - |
|---|-----|---|--------------|---------|---|
| • | PP[ | ) | | | |





Monday through Friday between 8:30 am and 4:30 pm (ET)

# 10.0 CRITERIA FOR REMOVAL FROM PROTOCOL THERAPY AND OFF STUDY CRITERIA

## 10.1 Criteria for Removal from Protocol Therapy

- a) Clinical (including physical examination or serum tumor markers) or radiographic evidence of progressive disease (See Section 12).
- b) Adverse Events requiring removal from protocol therapy (See Section 6).
- c) Refusal of protocol therapy by patient/parent/guardian
- d) Non-compliance that in the opinion of the investigator does not allow for ongoing participation.
- e) Completion of 6 cycles of therapy.
- f) Physician determines it is not in the patient's best interest.
- g) Repeated eligibility laboratory studies (CBC with differential, bilirubin, ALT (SGPT) or serum creatinine) are outside the parameters required for eligibility prior to the start of protocol therapy (See Section 8.1).
- h) Study is terminated by Sponsor.
- i) Pregnancy

Patients who are removed from protocol therapy during cycle 1 should continue to have the required observations in <u>Section 8.1</u> until the originally planned end of the cycle or until all adverse events have resolved per <u>Section 13.4.4</u>, whichever happens LATER. The only exception is with documentation of the patient's withdrawal of consent. Patients who are removed from protocol therapy in subsequent cycles should have the necessary observations to ensure adequate clinical care.

## 10.2 Follow-Up Data Submission and APEC1621SC Off Study Criteria

Patients who are off subprotocol therapy will initially be followed on the therapeutic subprotocol for a 30-day period. During follow-up on the subprotocol, ongoing adverse events, or adverse events that emerge after the patient is removed from protocol therapy, but within 30 days of the last dose of investigational agent, must be followed and reported via RAVE and CTEP-AERS (if applicable). Upon completion of subprotocol follow-up period, the patient will continue to be followed on the APEC1621SC screening protocol. Follow-up data submission will occur until one of the APEC1621SC Off Study Criteria is met (See Section 10 of APEC1621SC for details), consent is withdrawn or the patient dies or is lost to follow-up.

Version Date: 10/28/2022



#### 11.0 STATISTICAL AND ETHICAL CONSIDERATIONS

## 11.1 Sample Size and Study Duration

APEC1621D will require a minimum of 4 evaluable patients and a maximum of 144 patients (up to 98 biomarker-positive patients and up to 46 biomarker-negative patients, allowing for 15% inevaluability). Assuming an enrollment rate of 4-6 biomarker positive patients per year, this subprotocol is expected to be completed within 8-12 years.

As of Amendment #5A, accrual will stop once 20 evaluable patients have been accrued in the study. APEC1621D will require a maximum of 24 patients (allowing for 15% inevaluability). Assuming an enrollment rate of 4-6 biomarker positive patients per year, this subprotocol is expected to be completed within 4-6 years.

# 11.2 **Dosing Considerations**

Pediatric MATCH Sub-arm Dosing in the Absence of Pediatric Phase 1 Data
Please see Section 5.1.1 for a specific discussion of the dosing of LY3023414 to
be used in this study. As there is no prior pediatric phase 1 data for LY3023414,
study investigators have reviewed relevant data with the pharmaceutical partner
to identify a drug specific dosing plan for testing in children with
recurrent/refractory cancer, and trial participants will be closely monitored to
ensure tolerability of the selected dose. Because the adult RP2D of LY3023414 is
the adult MTD, APEC1621D will evaluate an initial cohort of patients at a dose
level approximately 30% below the adult MTD of LY3023414 and then
complete the study using the adult RP2D, assuming that both dose levels are
tolerated. Rules for determining tolerability of these dose levels are described in
Section 11.2.2. Limited pharmacokinetic sampling will be done for patients
enrolled on this arm. In general, the dosing for the Pediatric MATCH
subprotocols will follow the guidelines below:

#### 11.2.2 Determination of Recommended Phase 2 Dose (RP2D)/Tolerable Dose

Because the adult RP2D of LY3023414 is the adult MTD, APEC1621D will evaluate an initial cohort of patients at a dose level approximately 30% below the adult MTD and then complete the study using the adult RP2D, assuming that both dose levels are tolerated. A modified Rolling Six design will be followed. The DLT evaluation period for the purpose of dose escalation will be cycle 1 of therapy. Note that for toxicities which require persistence for a duration of time to be considered a DLT will be included if this time window starts during cycle 1 of therapy (e.g. grade 3 hypercholesterolemia would be considered a DLT if it developed during cycle 1 of therapy and persisted for 35 days). Patients enrolled during the determination of the recommended phase 2 dose who are not evaluable for toxicity during cycle 1 at a given dose level will be replaced.

Enrollment of the initial cohort of six patients will follow the standard rules of the rolling six design to assess safety and tolerability of cycle one of protocol treatment prior to extending accrual to additional patients.

If there are fewer than 2 DLTs in the first 6 toxicity-evaluable subjects enrolled at the starting dose, the dose will be escalated to the dose equivalent to 100% of the adult MTD for subsequent subjects enrolled on the study. If  $\geq$  2 of the first 6 toxicity evaluable subjects enrolled at the higher dose have DLTs, all subsequent



subjects will be enrolled at the original starting dose. Otherwise, remaining subjects will continue to enroll at the dose equivalent to 100% of the adult MTD.

If there are 2 or more DLTs among the first 6 toxicity-evaluable subjects enrolled at the original starting dose, the next cohort will enroll at a reduced dose level. If ≥ 2 of the first 6 toxicity-evaluable subjects enrolled at the reduced dose have DLTs, the study will be closed for toxicity. Otherwise, remaining subjects will continue to enroll at the reduced dose.

#### **Study Design** 11.3

The world's childhood

Each primary cohort and any biomarker negative expansion cohorts defined below will employ single stage A'Hern designs of N=20 and N=10 respectively. The agent will be deemed worthy of further study in the relevant subset of patients (i.e. biomarker positive in any histology, biomarker positive in a particular histology, etc) if the decision rule is met. Operating characteristics are shown below. See Appendix VIII for a list of target tumor histologies.

| Cohort | N | Decision Rule | Alpha | Power |
|----------------------------|----|---------------|-------|-------|
| Primary biomarker positive | 20 | ≥ 3 responses | 10% | 90% |
| Any biomarker negative | | ≥ 2 responses | 9% | 74% |

Histology-specific biomarker positive expansion cohorts will, by definition, be deemed worthy of further study, since they will have at least 3 responses. The table below shows 90% confidence intervals (Wilson method) for a range of observable response rates.

| Cohort Size | Observed Response Rate | 90% Confidence Interval |
|-------------|------------------------|-------------------------|
| 10 | 30% | 13% - 56% |
| 10 | 40% | 19% - 65% |
| 10 | 50% | 27% - 73% |

## 11.3.1 Primary Cohorts:

APEC1621D will evaluate two primary cohorts of 20 mutation-matched ("biomarker positive") evaluable patients of any histology for the primary study aim of determining the objective response rate (CR/PR according to the response criteria in Section 12.3) to LY3023414 (see Appendix VII):

Primary Cohort A: Patients whose tumors have TSC1 or TSC2 loss of function mutations

Primary Cohort B: Patients whose tumors have other PI3K/MTOR pathway activating mutations.

Using an A'Hern design<sup>60</sup> with alpha=10%, a sample of N=20 will provide 90% power to detect an improvement in response rate from 5%, if the treatment is ineffective, to 25% if the targeted therapy is sufficiently effective to warrant further study. If there are at least 3 responses out of 20 in either primary cohort A or B, the biomarker/therapy match will be deemed a success.

As of Amendment #5A, patients from the two primary cohorts will be combined and analyzed together in the primary analysis. The A'Hern design

CHILDREN'S

ONCOLOGY

GROUP

#### with N=20 as described above will be used.

## **Histology-Specific Biomarker Positive Expansion Cohorts:**

If  $\geq 3$  patients in either primary cohort A or B with the same histology show signs of objective response (CR/PR according to the response criteria in Section 12.3), a histology-specific biomarker positive expansion cohort will open after the primary cohort is completed to up to 7 evaluable patients for a total sample size of 10 evaluable biomarker positive patients with that histology. This will allow us to estimate more precisely the activity in biomarker positive patients of that histology.

We will open up to 3 such expansion cohorts for biomarker positive patients for each primary cohort (i.e., if 3 histologies in cohort A and 3 histologies in cohort B have  $\geq 3$  responses, we will open a total of 6 expansion cohorts as described above). Note that this can only happen if the response rate in each primary cohort is at least 45% (9/20) and there cannot be more than 42 additional evaluable patients in total for these expansion cohorts.

As of Amendment #5A, there will be no histology-specific biomarker positive expansion cohort planned for this subprotocol.

#### **Biomarker Negative Expansion Cohorts:** 11.3.3

The following expansion cohorts may open and will preferentially enroll patients to the earliest opened cohort when possible within slot availability/cohort suspension constraints. Patients enrolled in these biomarker negative expansion cohorts will be those whose tumors do NOT have one of the defined PI3K/MTOR pathway activating alterations leading to eligibility for either primary cohort A or B and do NOT have a genomic alteration that results in assignment to any other currently enrolling arm of the pediatric MATCH study.

As of Amendment #5A, there will be no biomarker negative expansion cohort planned for this subprotocol.

## 11.3.3.1 Histology-Agnostic Biomarker Negative Cohort:

If at any time  $\geq 3$  patients in primary cohort A or  $\geq 3$  patients in primary cohort B show signs of objective response, and the responding patients in that cohort include at least 2 different histologies, then a single expansion cohort of 10 biomarker negative patients of any histology will be opened. If in the course of the study  $\geq 3$  responses across primary cohort A and primary cohort B are observed in the same histology, then biomarker negative cohorts will be opened as described in Section 11.3.3.2. Biomarker negative patients for whom a histology-specific cohort is opened after the patient enrolls on the histology-agnostic biomarker negative cohort on APEC1621D will be reallocated to the histologyspecific cohort and not considered in the efficacy analysis for the histology-agnostic biomarker negative cohort (except in the event the criteria in section 11.3.3.3 are met). Biomarker negative patients for whom a histology specific cohort is open or has completed accrual prior to enrollment on APEC1621D will not be eligible to enroll on the histologyagnostic biomarker negative cohort.

This protocol is for research purposes only, see page 1 for usage policy. APEC1621D

Note that this criteria requires 3 responses in at least one of the primary cohorts of 20 patients (rather than both cohorts combined,) ensuring that the response rate is at least 15% in at least one of the primry cohorts before a histology-agnostic biomarker negative cohort would open.

If 2 or more responses are seen in the histology-agnostic biomarker negative cohort, the regimen will be declared active for biomarker negative patients. This will provide a low probability (9%) of carrying forward agents with response rates less than 5% and a moderately high probability (74%) of identifying agents with response rates  $\geq$  25%.

# 11.3.3.2 <u>Histology-Specific Biomarker Negative Cohorts</u>:

If at any time  $\geq 3$  patients in either primary cohort A or B with the same histology show signs of objective response, then an expansion cohort of 10 biomarker negative patients with the same histology will be opened.

Note: The criteria to open a biomarker negative histology-specific criteria applies to the combined set of subjects in primary cohorts A and B. For example, 1 response in primary cohort A and 2 responses in primary cohort B in the same histology would meet the critieria to open a histology specific biomarker negative cohort for that histology.

If 2 or more responses are seen in a histology-specific biomarker negative cohort, the regimen will be declared active for biomarker negative patients of that histology. Using this A'Hern single stage design will assure a low probability (9%) of carrying forward agents with response rates less than 5% and provide a moderately high probability (74%) of identifying agents with response rates  $\geq$  25%. Up to a total of 3 such biomarker negative cohorts can be opened, for a total of 30 biomarker negative patients.

Note: Biomarker negative histology-specific criteria applies to the combined set of subjects in primary cohorts A and B.

#### 11.3.3.3 Histology-Agnostic Biomarker Negative Stopping Rule

If a histology-specific biomarker negative cohort has completed accrual and there are fewer than 2 responses observed, and there have not been any responses observed in the histology-agnostic biomarker-negative expansion cohort (if open), then the histology-agnostic biomarker negative cohort will not open to accrual or will close to accrual if open. In this circumstance, patients from the histology-specific biomarker negative expansion cohort will be included in the efficacy analysis for the histology-agnostic biomarker negative expansion cohort, which will by definition be considered not active with 0-1 responses out of 10-20 subjects.

Note that the histology-agnostic biomarker negative expansion cohort may accrue prior to or in parallel with biomarker negative histology-specific expansion cohorts. Enrollment to the biomarker negative histology-agnostic cohort will continue while waiting to determine if this criteria applies. This criteria will only apply after at least 9 subjects on the



This protocol is for research purposes only, see page 1 for usage policy. APEC1621D

histology-specific biomarker cohort have discontinued treatment such that it is not possible to have  $\geq 2$  responses.

#### 11.4 **Methods of Analysis**

Response criteria are described in <u>Section 12.0</u>. A responder is defined as a patient who achieves a best response of PR or CR on the study. Response rates will be calculated as the percent of evaluable patients who are responders, and confidence intervals will be constructed using the Wilson score interval method.<sup>61</sup> Decision making for A'Hern design cohorts will follow rules described above.

Any responses or lack thereof in patients enrolled during the determination of the Recommended Phase 2 Dose (dose finding phase) will count toward the objective response rate in their respective cohort.

Toxicity tables will be constructed to summarize the observed incidence by type of toxicity and grade. A patient will be counted only once for a given toxicity for the worst grade of that toxicity reported for that patient. Toxicity information recorded will include the type, severity, time of onset, time of resolution, and the probable association with the study regimen.

#### 11.5 **Evaluability for Response**

Any eligible patient who is enrolled and receives at least one dose of protocol therapy on any APEC1621 subprotocol will be considered evaluable for response. Any patient who receives non-protocol anti-cancer therapy during the response evaluation period will be considered a non-responder for the purposes of the statistical rule, unless they show an objective response prior to receiving the non-protocol anti-cancer therapy (in which case they will be considered a responder). Patients who demonstrate a complete or partial response confirmed by central review will be considered to have experienced a response. All other patients will be considered non-responders. Patients who are not evaluable for response evaluation may be replaced for the purposes of the statistical rule. All patients considered to have a response (CR or PR) must have imaging studies reviewed centrally at the COG. Centers will be notified by the COG about requests for scans of patients with stable disease. Preliminary assessment of activity using institutionally provided tumor measurements will be entered into CDUS quarterly. The central review by COG will be provided as the final reviewed assessment of response when such becomes available.

#### 11.6 **Evaluability for Toxicity**

Any patient who experiences a DLT at any time during protocol therapy is considered evaluable for toxicity. Patients without DLT who receive at least 85% of the prescribed dose per protocol guidelines and had the appropriate toxicity monitoring studies performed during cycle 1 are also considered evaluable for toxicity.

#### 11.7 **Progression free survival (PFS)**

Progression free survival will be defined as time from the initiation of protocol treatment to the occurrence of any of the following events: disease progression or disease recurrence or death from any cause. All patients surviving at the time of analyses without events will be censored at their last follow-up date.

PFS along with the confidence intervals will be estimated using the Kaplan-Meier method. Patients with local calls of disease progression (i.e. calls made by the treating institution), will be counted as having had an event, even if the central review does not declare



progression. We will also report PFS based on central radiology review as a secondary analysis, if adequate number of disagreements in progressions exist between the treating institutions and the central radiology review to make such an analysis meaningful.

#### 11.8 Correlative Studies

A descriptive analysis of pharmacokinetic (PK) parameters will be performed to define systemic exposure, drug clearance, and other pharmacokinetic parameters. The PK parameters will be summarized with simple summary statistics, including means, medians, ranges, and standard deviations (if numbers and distribution permit).

A descriptive analysis of the exploratory aims described in <u>Section 1.3</u> will be performed and will be summarized with simple summary statistics. All of these analyses will be descriptive in nature.

# 11.9 Gender and Minority Accrual Estimates

The gender and minority distribution of the study population is expected to be:

| Racial category | Not Hispanic<br>or Latino | | Hispanic or<br>Latino | | |
|---|---|---|---|---|---|
| | Female | Male | Female | Male | Total |
| American Indian/Alaska Native | 0 | 0 | 0 | 0 | 0 |
| Asian | 0 | 0 | 0 | 0 | 0 |
| Native Hawaiian or Other<br>Pacific Islander | 0 | 0 | 0 | 0 | 0 |
| Black or African American | 2 | 3 | 0 | 0 | 5 |
| White | 6 | 10 | 2 | 1 | 19 |
| More than one race | 0 | 0 | 0 | 0 | 0 |
| Total | 8 | 13 | 2 | 1 | 24 |

This distribution was derived from the demographic data for patients enrolled on recent COG Phase 2 trials.



#### 12.0 EVALUATION CRITERIA

# 12.1 Common Terminology Criteria for Adverse Events (CTCAE)

The descriptions and grading scales found in the current version of the NCI Common Terminology Criteria for Adverse Events v5.0 (CTCAE) will be utilized for AE reporting. All appropriate treatment areas should have access to a copy of the current CTCAE v5.0. A copy of the CTCAE v5.0 can be downloaded from the CTEP website (http://ctep.cancer.gov).

## 12.2 **Progression-Free Survival**

Progression-free survival (PFS) is defined as the duration of time from start of subprotocol treatment to time of progression or death, whichever occurs first.

Development of new disease or progression in any established lesions is considered progressive disease, regardless of response in other lesions – e.g., when multiple lesions show opposite responses, the progressive disease takes precedence.

# 12.3 Response Criteria for Patients with Solid Tumors

See the table in <u>section 8.0</u> for the schedule of tumor evaluations. Eligible patients must have measurable disease present at baseline and have had their disease re-evaluated after one dose of protocol therapy. In addition to the scheduled scans, a confirmatory scan should be obtained on the next consecutive cycle following initial documentation of objective response.

As outlined, patients will be assigned to one of the following categories for assessment of response: a) solid tumor (non-CNS) and measurable disease (Section 12.4); b) neuroblastoma with MIBG positive lesions (Section 12.5); c) CNS tumor (Section 12.7); and d) non-Hodgkin lymphoma/hystiocytosis (Section 12.8). Note: Neuroblastoma patients who do not have MIBG positive lesions should be assessed for response as solid tumor patients with measurable disease.

Response and progression will be evaluated in this study using the revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1).<sup>62</sup> Key points are that 5 target lesions are identified and that changes in the *largest* diameter (unidimensional measurement) of the tumor lesions but the *shortest* diameter of malignant lymph nodes are used in the RECIST v 1.1 criteria.

# 12.3.1 Definitions

## 12.3.1.1 Evaluable for objective response:

Eligible patients who receive at least one dose of protocol therapy will be considered evaluable for response. Evaluable patients who demonstrate a complete or partial response confirmed by central review before receiving non-protocol anti-cancer therapy will be considered a responder. All other evaluable patients will be considered non-responders.

## 12.3.1.2 <u>Evaluable Non-Target Disease Response</u>:

Eligible patients who have evaluable but not measurable disease and have received at least one dose of protocol therapy will be considered evaluable for non-target disease. The response assessment is based on



the presence, absence, or unequivocal progression of the lesions.

#### 12.3.2 Disease Parameters

12.3.2.1 <u>Measurable disease</u>: Measurable lesions are defined as those that can be accurately measured in at least one dimension (longest diameter to be recorded) as  $\geq 20$  mm by chest x-ray, as  $\geq 10$  mm with CT scan, or  $\geq 10$  mm with calipers by clinical exam. All tumor measurements must be recorded in millimeters (or decimal fractions of centimeters).

Note: Tumor lesions that are situated in a previously irradiated area might or might not be considered measurable. If the investigator thinks it appropriate to include them, the conditions under which such lesions should be considered must be defined in the protocol.

- 12.3.2.2 <u>Malignant lymph nodes</u>: To be considered pathologically enlarged and measurable, a lymph node must be ≥ 15 mm in short axis when assessed by CT scan (CT scan slice thickness no greater than 5 mm). At baseline and in follow-up, only the short axis will be measured and followed.
- 12.3.2.3 Non-measurable disease: All other lesions (or sites of disease), including small lesions (longest diameter < 10 mm or pathological lymph nodes with  $\geq 10$  to < 15 mm short axis), are considered non-measurable disease. Bone leptomeningeal lesions, disease, ascites, pleural/pericardial effusions. lymphangitis cutis/pulmonitis, inflammatory breast disease, and abdominal masses (not followed by CT or MRI), are considered as non-measurable.

Note: Cystic lesions that meet the criteria for radiographically defined simple cysts should not be considered as malignant lesions (neither measurable nor non-measurable) since they are, by definition, simple cysts. 'Cystic lesions' thought to represent cystic metastases can be considered as measurable lesions, if they meet the definition of measurability described above. However, if non-cystic lesions are present in the same patient, these are preferred for selection as target lesions.

Target lesions: All measurable lesions up to a maximum of 2 lesions per 12.3.2.4 organ and 5 lesions in total, representative of all involved organs, should be identified as target lesions and recorded and measured at baseline. Target lesions should be selected on the basis of their size (lesions with the longest diameter), be representative of all involved organs, but in addition should be those that lend themselves to reproducible repeated measurements. It may be the case that, on occasion, the largest lesion does not lend itself to reproducible measurement in which circumstance the next largest lesion that can be measured reproducibly should be selected. A sum of the diameters (longest for non-nodal lesions, short axis for nodal lesions) for all target lesions will be calculated and reported as the baseline sum diameters. If lymph nodes are to be included in the sum, then only the short axis is added into the sum. The baseline sum diameters will be used as reference to further characterize any objective tumor regression in the measurable dimension of the

disease.

12.3.2.5 <u>Non-target lesions</u>: All other lesions (or sites of disease) including any measurable lesions over and above the 5 target lesions should be identified as non-target lesions and should also be recorded at baseline. Measurements of these lesions are not required, but the presence, absence, or in rare cases unequivocal progression of each should be noted throughout follow-up.

## 12.3.3 Methods for Evaluation of Measurable Disease

All measurements should be taken and recorded in metric notation using a ruler or calipers.

The same method of assessment and the same technique should be used to characterize each identified and reported lesion at baseline and during follow-up. Imaging-based evaluation is preferred to evaluation by clinical examination unless the lesion(s) being followed cannot be imaged but are assessable by clinical exam.

- 12.3.3.1 <u>Clinical lesions</u>: Clinical lesions will only be considered measurable when they are superficial (e.g., skin nodules and palpable lymph nodes) and  $\geq 10$  mm diameter as assessed using calipers (e.g., skin nodules). In the case of skin lesions, documentation by color photography, including a ruler to estimate the size of the lesion, is recommended.
- 12.3.3.2 <u>Chest x-ray</u>: Lesions on chest x-ray are acceptable as measurable lesions when they are clearly defined and surrounded by aerated lung. However, CT is preferable.
- 12.3.3.3 Conventional CT and MRI: This guideline has defined measurability of lesions on CT scan based on the assumption that CT slice thickness is 5 mm or less. If CT scans have slice thickness greater than 5 mm, the minimum size for a measurable lesion should be twice the slice thickness. MRI is also acceptable in certain situations (e.g. for body scans). Ideally, the same type of scanner should be used and the image acquisition protocol should be followed as closely as possible to prior scans.
- 12.3.3.4 PET-CT: At present, the low dose or attenuation correction CT portion of a combined PET-CT is not always of optimal diagnostic CT quality for use with RECIST measurements. However, if the site can document that the CT performed as part of a PET-CT is of identical diagnostic quality to a diagnostic CT (with IV and oral contrast), then the CT portion of the PET-CT can be used for RECIST or International Pediatric non-Hodgkin Lymphoma Response Criteria measurements and can be used interchangeably with conventional CT in accurately measuring cancer lesions over time. Note, however, that the PET portion of the CT introduces additional data which may bias an investigator if it is not routinely or serially performed.
- 12.3.3.5 <u>Tumor markers</u>: Tumor markers alone cannot be used to assess response. If markers are initially above the upper normal limit, they must normalize for a patient to be considered in complete clinical response.



12.3.3.6 <u>Cytology</u>, <u>Histology</u>: These techniques can be used to differentiate between partial responses (PR) and complete responses (CR) in rare cases (e.g., residual lesions in tumor types, such as germ cell tumors, where known residual benign tumors can remain).

Cytology should be obtained if an effusion appears or worsens during treatment when the measurable tumor has met criteria for response or stable disease.

- 12.3.3.7 <u>FDG-PET</u>: While FDG-PET response assessments need additional study, it is sometimes reasonable to incorporate the use of FDG-PET scanning to complement CT scanning in assessment of progression (particularly possible 'new' disease). New lesions on the basis of FDG-PET imaging can be identified according to the following algorithm:
  - a. Negative FDG-PET at baseline, with a positive FDG-PET at followup is a sign of PD based on a new lesion.
  - b. No FDG-PET at baseline and a positive FDG-PET at follow-up: If the positive FDG-PET at follow-up corresponds to a new site of disease confirmed by CT, this is PD. If the positive FDG-PET at follow-up is not confirmed as a new site of disease on CT, additional follow-up CT scans are needed to determine if there is truly progression occurring at that site (if so, the date of PD will be the date of the initial abnormal FDG-PET scan). If the positive FDG-PET at follow-up corresponds to a pre-existing site of disease on CT that is not progressing on the basis of the anatomic images, this is not PD.

Note: A 'positive' FDG-PET scan lesion means one that is FDG avid with an uptake greater than twice that of the surrounding tissue on the attenuation corrected image.

For patients with a positive PET scan at diagnosis, PET can be used to follow response in addition to a CT scan using the International Pediatric non-Hodgkin Lymphoma Response Criteria.<sup>63</sup>

# 12.4 Response Criteria for Patients with Solid Tumor and Measurable Disease

#### 12.4.1 Evaluation of Target Lesions

Complete Response (CR):

Disappearance of all target and non-target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. If immunocytology is available, no disease must be detected by that methodology. Normalization of urinary catecholamines or other tumor markers if elevated at study enrollment (for patients with neuroblastoma).

Partial Response (PR):

At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the



#### baseline sum diameters

Progressive Disease (PD):

At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progressions). Note: in presence of SD or PR in target disease but unequivocal progression in non-target or nonmeasurable disease, the patient has PD if there is an overall level of substantial worsening in nontarget disease such that the overall tumor burden has increased sufficiently to merit discontinuation of therapy

Stable Disease (SD):

Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study

#### 12.4.2 Evaluation of Non-Target Lesions

Complete Response (CR):

Disappearance of all non-target lesions and normalization of tumor marker level. All lymph nodes must be non-pathological in size (<10 mm short axis)

Note: If tumor markers are initially above the upper normal limit, they must normalize for a patient to be considered in complete clinical response.

Non-CR/Non-PD: Persistence of one or more non-target lesion(s)

and/or maintenance of tumor marker level above

the normal limits

Progressive Disease (PD): Appearance of one or more new lesions and/or

> unequivocal progression of existing non-target lesions. Unequivocal progression should not normally trump target lesion status. It must be representative of overall disease status change,

not a single lesion increase.

## 12.4.3 Overall Response Assessment

Table 1: For Patients with Measurable Disease (i.e., Target Disease)

| Target | Non-Target | New | Overall | Best Overall Response when Confirmation is |
|---|---|---|---|---|
| Lesions | Lesions | Lesions | Response | |
| | | | _ | Required* |

Any

| CR | CR | No | CR | ≥ 28 days Confirmation |
|-----|---------------|-----------|----|----------------------------|
| CR | Non- | No | PR | |
| | CR/Non-PD | | | ≥ 28 days Confirmation |
| CR | Not evaluated | No | PR | |
| PR | Non- | No | PR | |
| | CR/Non- | | | |
| | PD/not | | | |
| | evaluated | | | |
| SD | Non- | No | SD | documented at least once ≥ |
| | CR/Non- | | | 28 days from baseline |
| | PD/not | | | |
| | evaluated | | | |
| PD | Any | Yes or No | PD | |
| Any | PD** | Yes or No | PD | no prior SD, PR or CR |

<sup>\*</sup> See RECIST 1.1 manuscript for further details on what is evidence of a new lesion.

Yes

PD

Note: Patients with a global deterioration of health status requiring discontinuation of treatment without objective evidence of disease progression at that time should be reported as "symptomatic deterioration." Every effort should be made to document the objective progression even after discontinuation of treatment.

Table 2: For Patients with Non-Measurable Disease (i.e., Non-Target Disease)

| Non-Target Lesions | New Lesions | Overall Response |
|--------------------|-------------|------------------|
| CR | No | CR |
| Non-CR/non-PD | No | Non-CR/non-PD* |
| Not all evaluated | No | not evaluated |
| Unequivocal PD | Yes or No | PD |
| Any | Yes | PD |

<sup>\* &#</sup>x27;Non-CR/non-PD' is preferred over 'stable disease' for non-target disease since SD is increasingly used as an endpoint for assessment of efficacy in some trials so to assign this category when no lesions can be measured is not advised

Table 3: Overall Response for Patients with Neuroblastoma and Measurable Disease

Any

| CT/MRI | MIBG | Bone Scan | Bone Marrow | Catechol | Overall |
|--------|----------|-----------|-------------|----------|---------|
| PD | Any | Any | Any | Any | PD |
| Any | PD | Any | Any | Any | PD |
| Any | Any | PD | Any | Any | PD |
| Any | Any | Any | PD | Any | PD |
| SD | CR/PR/SD | Non-PD | Non-PD | Any | SD |
| PR | CR/PR | Non-PD | Non-PD | Any | PR |
| CR/PR | PR | Non-PD | Non-PD | Any | PR |
| CR | CR | Non-PD | Non-PD | Elevated | PR |
| CR | CR | CR | CR | Normal | CR |

# 12.4.4 Overall Best Response Assessment

Each patient will be classified according to his "best response" for the purposes of analysis of treatment effect. Best response is determined as outlined in <u>Section 12.9</u> from a sequence of overall response assessments.

<sup>\*\*</sup> In exceptional circumstances, unequivocal progression in non-target lesions may be accepted as disease progression.



## 12.5 Response Criteria for Neuroblastoma Patients with MIBG Positive Lesions

## 12.5.1 MIBG Positive Lesions

Patients who have a positive MIBG scan at the start of therapy will be evaluable for MIBG response. The use of <sup>123</sup>I for MIBG imaging is recommended for all scans. If the patient has only one MIBG positive lesion and that lesion was radiated, a biopsy must be done at least 28 days after radiation was completed and must show yiable neuroblastoma.

12.5.2 <u>The following criteria will be used to report MIBG response by the treating institution:</u>

Complete response: Complete resolution of all MIBG positive lesions

Partial Response: Resolution of at least one MIBG positive lesion, with

persistence of other MIBG positive lesions

Stable disease: No change in MIBG scan in number of positive lesions

Progressive disease: Development of new MIBG positive lesions

12.5.3 The response of MIBG lesions will be assessed on central review using the Curie scale14 as outlined below. Central review responses will be used to assess efficacy for study endpoint. See Section 8.2 for details on transferring images to the Imaging Research Center.

NOTE: This scoring should also be done by the treating institution for end of course response assessments.

The body is divided into 9 anatomic sectors for osteomedullary lesions, with a 10<sup>th</sup> general sector allocated for any extra-osseous lesion visible on MIBG scan. In each region, the lesions are scored as follows. The **absolute extension score** is graded as:

0 = no site per segment,

1 = 1 site per segment,

2 = more than one site per segment,

3 = massive involvement (>50% of the segment).

The **absolute score** is obtained by adding the score of all the segments. See diagram of sectors below:





The **relative score** is calculated by dividing the absolute score at each time point by the corresponding pre-treatment absolute score. The relative score of each patient is calculated at each response assessment compared to baseline and classified as below:

- 1. **Complete response:** all areas of uptake on MIBG scan completely resolved. If morphological evidence of tumor cells in bone marrow biopsy or aspiration is present at enrollment, no tumor cells can be detected by routine morphology on two subsequent bilateral bone marrow aspirates and biopsies done at least 21 days apart to be considered a Complete Response.
- 2. **Partial response**: Relative score  $\leq 0.2$  (lesions almost disappeared) to  $\leq 0.5$ (lesions strongly reduced).
- 3. **Stable disease**: Relative score > 0.5 (lesions weakly but significantly reduced) to 1.0 (lesions not reduced).
- 4. **Progressive disease**: New lesions on MIBG scan.

## 12.5.4 Overall Response Assessment

# Table 4: Overall Response Evaluation for Neuroblastoma Patients and MIBG Positive Disease

If patients are enrolled without disease measurable by CT/MRI, any new or newly identified lesion by CT/MRI that occurs during therapy would be considered progressive disease.

| MIBG | CT/MRI | Bone Scan | <b>Bone Marrow</b> | Catechol | Overall |
|------|---------------|-----------|--------------------|----------|---------|
| PD | Any | Any | Any | Any | PD |
| Any | New Lesion | Any | Any | Any | PD |
| Any | Any | PD | Any | Any | PD |
| Any | Any | Any | PD | Any | PD |
| SD | No New Lesion | Non-PD | Non-PD | Any | SD |
| PR | No New Lesion | Non-PD | Non-PD | Any | PR |
| CR | No New Lesion | Non-PD | Non-PD | Elevated | PR |
| CR | No New Lesion | CR | CR | Normal | CR |



# 12.5.5 Overall Best Response Assessment

Each patient will be classified according to his "best response" for the purposes of analysis of treatment effect. Best response is determined from the sequence of the overall response assessments as described in Section 12.9.

#### 12.6 Response Criteria for Neuroblastoma Patients with Bone Marrow Involvement

#### 12.6.1 Bone Marrow Involvement

**Note:** patients with bone marrow as the ONLY site of disease are not eligible for this study. Response criteria in this section are intended to be used when assessing marrow involvement as a component of overall response.

Histologic analysis at the local institution of marrow tumor cell involvement is **required** for patients with a history of marrow involvement. Marrow aspirate and biopsy should be evaluated at baseline and every 2 cycles thereafter. Note: If progressive disease is documented by RECIST criteria using tumor measurements or by MIBG scan, then a repeat BM is not needed to confirm PD.

Complete Response: No tumor cells detectable by routine morphology on 2

consecutive bilateral bone marrow aspirates and biopsies performed at least 21 days apart. Normalization of urinary catecholamines or other tumor markers if elevated at

study enrollment.

Progressive Disease: In patients who enroll with neuroblastoma in bone

marrow by morphology have progressive disease if there is a doubling in the amount of tumor in the marrow AND a minimum of 25% tumor in bone marrow by morphology. (For example, a patient entering with 5% tumor in marrow by morphology must increase to  $\geq 25\%$  tumor to have progressive disease; a patient entering with

30% tumor must increase to > 60%).

In patients who enroll without evidence of neuroblastoma in bone marrow will be defined as progressive disease if tumor is detected in 2 consecutive bone marrow biopsies

or aspirations done at least 21 days apart.

<u>Stable Disease</u>: Persistence of tumor in bone marrow that does not meet

the criteria for either complete response or progressive

disease.

## 12.6.2 Overall Best Response Assessment

Each patient will be classified according to his "best response" for the purposes of analysis of treatment effect. Best response is determined from the sequence of the overall response assessments as described in <u>Section 12.9</u>.

# 12.7 Response Criteria for Patients with CNS Tumors

## 12.7.1 Measurable Disease

THIS PROTOCOL IS FOR RESEARCH PURPOSES ONLY. SEE PAGE 1 FOR USAGE POLICY. APEC1621D

Any lesion that is at minimum 10 mm in one dimension on standard MRI or CT, for CNS tumors.

## 12.7.2 Evaluable Disease

The world's childhood

Evaluable disease is defined as at least one lesion, with no lesion that can be accurately measured in at least one dimension. Such lesions may be evaluable by nuclear medicine techniques, immunocytochemistry techniques, tumor markers, CSF cytology, or other reliable measures.

## 12.7.3 Selection of Target and Non-Target Lesions

For most CNS tumors, only one lesion/mass is present and therefore is considered a "target" for measurement/follow up to assess for tumor progression/response. If multiple measurable lesions are present, up to 5 should be selected as "target" lesions. Target lesions should be selected on the basis of size and suitability for accurate repeated measurements. All other lesions will be followed as non-target lesions. The lower size limit of the target lesion(s) should be at least twice the thickness of the slices showing the tumor to decrease the partial volume effect (e.g., 8 mm lesion for a 4 mm slice).

Any change in size of non-target lesions should be noted, though does not need to be measured.

# 12.7.4 Response Criteria for Target Lesions

Response criteria are assessed based on the product of the longest diameter and its longest perpendicular diameter. Development of new disease or progression in any established lesions is considered progressive disease, regardless of response in other lesions — e.g., when multiple lesions show opposite responses, the progressive disease takes precedence. Response Criteria for target lesions:

- <u>Complete Response (CR):</u> Disappearance of all target lesions. Off all steroids with stable or improving neurologic examination.
- Partial response (PR): ≥ 50% decrease in the sum of the products of the two perpendicular diameters of all target lesions (up to 5), taking as reference the initial baseline measurements; on a stable or decreasing dose of steroids with a stable or improving neurologic examination.
- <u>Stable Disease (SD):</u> Neither sufficient decrease in the sum of the products of the two perpendicular diameters of all target lesions to qualify for PR, nor sufficient increase in a single target lesion to qualify for PD; on a stable or decreasing dose of steroids with a stable or improving neurologic examination.
- Progressive Disease (PD): 25% or more increase in the sum of the products of the perpendicular diameters of the target lesions, taking as reference the smallest sum of the products observed since the start of treatment, or the appearance of one or more new lesions.

Increasing doses of corticosteroids required to maintain stable neurological status should be strongly considered as a sign of clinical progression unless in the context of recent wean or transient neurologic change due e.g. to radiation


effects.

The world's childhood

# 12.7.5 Response Criteria for Non-Target Lesions:

- <u>Complete Response (CR):</u> Disappearance of all non-target lesions.
- <u>Incomplete Response/Stable Disease (IR/SD):</u> The persistence of one or more non-target lesions.
- **Progressive Disease (PD):** The appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions.

## 12.7.6 Response criteria for tumor markers (if available):

Tumor markers will be classified simply as being at normal levels or at abnormally high levels.

# 12.7.7 Overall Response Assessment

The overall response assessment takes into account response in both target and non-target lesions, the appearance of new lesions and normalization of markers (where applicable), according to the criteria described in the table below. The overall response assessment is shown in the last column, and depends on the assessments of target, non-target, marker and new lesions in the preceding columns.

| Target Lesions | Non-target Lesions | Markers | New Lesions | Overall<br>Response |
|---|---|---|---|---|
| CR | CR | Normal | No | CR |
| CR | IR/SD | Normal | No | PR |
| CR | CR, IR/SD | Abnormal | No | PR |
| PR | CR, IR/SD | Any | No | PR |
| SD | CR, IR/SD | Any | No | SD |
| PD | Any | Any | Yes or No | PD |
| Any | PD | Any | Yes or No | PD |
| Any | Any | Any | Yes | PD |

Each patient will be classified according to his "best response" for the purposes of analysis of treatment effect. Best response is determined as outlined in <u>Section 12.9</u> from a sequence of overall response assessments.

# 12.8 Response Criteria for Patients with non-Hodgkin Lymphoma/Histiocytosis

Response and progression will be evaluated in this study using the new international criteria proposed by the revised Response Evaluation Criteria in Pediatric non-Hodgkin Lymphoma Criteria<sup>63</sup>, with modification from the Lugano classification.<sup>64</sup>

#### 12.8.1 Disease Parameters

12.8.1.1 <u>Measurable disease</u>: A measurable node must have an LDi (longest diameter) greater than 1.5 cm. A measurable extranodal lesion should



This protocol is for research purposes only, see page 1 for usage policy. APEC1621D

have an LDi greater than 1.0 cm. All tumor measurements must be recorded in millimeters (or decimal fractions of centimeters).

- 12.8.1.2Non-measured disease: All other lesions (including nodal, extranodal, and assessable disease) should be followed as nonmeasured disease (e.g., cutaneous, GI, bone, spleen, liver, kidneys, pleural or pericardial effusions, ascites).
- 12.8.1.3 Target lesions: For patients staged with CT, up to six of the largest target nodes, nodal masses, or other lymphomatous lesions that are measurable in two diameters (longest diameter [LDi] and shortest diameter) should be identified from different body regions representative of the patient's overall disease burden and include mediastinal and retroperitoneal disease, if involved.

#### 12.8.2 Evaluation of Measurable Disease

# Complete Response (CR)

Disappearance of all disease. CT or MRI should be free of residual mass or evidence of new disease. FDG-PET should be negative.

#### Complete Response Unconfirmed (CRu)

Residual mass is negative by FDG-PET; no new lesions by imaging examination; no new and/or progressive disease elsewhere

#### Partial Response (PR)

50% decrease in SPD (the sum of the products of the largest diameter and the perpendicular diameter for a tumor mass) on CT or MRI; FDG-PET may be positive (Deauville score or 4 or 5 with reduced lesional uptake compared with baseline); no new and/or PD; morphologic evidence of disease may be present in BM if present at diagnosis; however, there should be 50% reduction in percentage of lymphoma cells.

## No Response (Stable Disease)

Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.

## Progressive disease

For those with > 25% increase in SPD on CT or MRI, Deauville score 4 or 5 on FDG-PET with increase in lesional uptake from baseline, or development of new morphologic evidence of disease in BM

12.8.3 Evaluation of Non-measured Lesions (CT-based response, PET/CT based response not applicable)<sup>64</sup>

Complete Response (CR): Absent non-measured lesions.

Partial response (PR): Absent/normal, regressed, lesions, but no increase.

Stable Disease (SD): No increase consistent with progression



<u>Progressive Disease (PD)</u>: New or clear progression of preexisting

non-measured lesions.

# 12.8.4 Evaluation of organ enlargement<sup>64</sup>

<u>Complete Response (CR)</u>: Regress to normal

Partial response (PR): Spleen must have regressed by >50% in length

beyond normal

<u>Stable Disease (SD):</u> No increase consistent with progression

<u>Progressive Disease (PD)</u>: In the setting of splenomegaly, the splenic length

must increase by 50% of the extent of its prior increase beyond baseline. If no prior splenomegaly,

must increase by at least 2 cm from baseline.

New or recurrent splenomegaly

## 12.9 **Best Response**

Two objective status determinations of disease status, obtained on two consecutive determinations, separated by at least a 3 week time period, are required to determine the patient's overall best response. Two objective status determinations of CR before progression are required for best response of CR. Two determinations of PR or better before progression, but not qualifying for a CR, are required for a best response of PR. Two determinations of stable/no response or better before progression, but not qualifying as CR or PR, are required for a best response of stable/no response; if the first objective status is unknown, only one such determination is required. Patients with an objective status of progression on or before the second evaluations (the first evaluation is the first radiographic evaluation after treatment has been administered) will have a best response of progressive disease. Best response is unknown if the patient does not qualify for a best response of progressive disease and if all objective statuses after the first determination and before progression are unknown.

# 12.9.1 Evaluation of Best Overall Response

The best overall response is the best response recorded from the start of the treatment until disease progression/recurrence (taking as reference for progressive disease the smallest measurements recorded since the treatment started). The patient's best response assignment will depend on the achievement of both measurement and confirmation criteria.

Table 5. Sequences of overall response assessments with corresponding best response.

| 1st Assessment | 2 <sup>nd</sup> Assessment | Best Response |
|----------------|----------------------------|-------------------------|
| Progression | | Progressive disease |
| Stable, PR, CR | Progression | Progressive disease |
| Stable | Stable | Stable |
| Stable | PR, CR | Stable |
| Stable | Not done | Not RECIST classifiable |

This protocol is for research purposes only. See page 1 for usage policy. APEC1621D

| PR | PR | PR |
|--------|----------|-------------------------|
| PR | CR | PR |
| PR, CR | Not done | Not RECIST classifiable |
| CR | CR | CR |

## 12.9.2 **Duration of Response**

<u>Duration of overall response</u>: The duration of overall response is measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started).

The duration of overall CR is measured from the time measurement criteria are first met for CR until the first date that progressive disease is objectively documented.

<u>Duration of stable disease</u>: Stable disease is measured from the start of the treatment until the criteria for progression are met, taking as reference the smallest measurements recorded since the treatment started, including the baseline measurements.



# 13.0 ADVERSE EVENT REPORTING REQUIREMENTS

Adverse event data collection and reporting which are required as part of every clinical trial, are done to ensure the safety of patients enrolled in the studies as well as those who will enroll in future studies using similar agents. Adverse events are reported in a routine manner at scheduled times during a trial. (Please follow directions for routine reporting provided in the Case Report Forms for this protocol). Additionally, certain adverse events must be reported in an expedited manner to allow for optimal monitoring of patient safety and care. The following sections provide information about expedited reporting.

Reporting requirements may include the following considerations: 1) whether the patient has received an investigational agent; 2) whether the adverse event is considered serious; 3) the grade (severity); and 4) whether or not hospitalization or prolongation of hospitalization was associated with the event.

An <u>investigational agent</u> is a protocol drug administered under an Investigational New Drug Application (IND). In some instances, the investigational agent may be available commercially, but is actually being tested for indications not included in the approved package label.

# 13.1 Expedited Reporting Requirements – Serious Adverse Events (SAEs)

Any AE that is serious qualifies for expedited reporting. An AE is defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. A Serious Adverse Event (SAE) is any adverse drug event (experience) occurring at any dose that results in ANY of the following outcomes:

- 1) Death.
- 2) A life-threatening adverse drug experience.
- 3) An adverse event resulting in inpatient hospitalization or prolongation of existing hospitalization (for ≥ 24 hours). This does not include hospitalizations that are part of routine medical practice.
- 4) A persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions.
- 5) A congenital anomaly/birth defect.
- 6) Important Medical Events (IME) that may not result in death, be life threatening, or require hospitalization may be considered a serious adverse drug experience when, based upon medical judgment, they may jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the outcomes listed in this definition.

## 13.1.1 Reporting Requirements - Investigator Responsibility

Clinical investigators in the treating institutions and ultimately the Study Chair have the primary responsibility for AE identification, documentation, grading, and assignment of attribution to the investigational agent/intervention. It is the responsibility of the treating physician to supply the medical documentation needed to support the expedited AE reports in a timely manner.

Any medical documentation supporting an expedited report (eg, H & P, admission and/or notes, consultations, ECG results, etc.) MUST be faxed within 48-72 hours to the NCI. NOTE: English is required for supporting documentation submitted to the numbers listed below in order for the NCI to



## meet the regulatory reporting timelines.

Fax supporting documentation for AEs related to investigational agents supplied under a CTEP IND to: PPD

Also: Fax or email supporting documentation to COG for **all** IND studies (Fax# (310) 640-9193; email: <u>COGAERS@childrensoncologygroup.org</u>; Attention: COG AERS Coordinator).

- ALWAYS include the ticket number on all faxed documents.
- Use the NCI protocol number and the protocol-specific patient ID provided during trial registration on all reports.

# 13.1.2 CTEP-AERS Expedited Reporting Methods

Expedited AE reporting for this study must only use CTEP-AERS (Adverse Event Expedited Reporting System), accessed via the CTEP home page <a href="https://eapps-ctep.nci.nih.gov/ctepaers">https://eapps-ctep.nci.nih.gov/ctepaers</a>.

Send supporting documentation to the NCI by fax (fax# 301-640-9193) and by email to the APEC1621D COG Study Assigned Research Coordinator and <a href="COGAERS@childrensoncologygroup.org">COGAERS@childrensoncologygroup.org</a>; Attention: COG AERS Coordinator. ALWAYS include the ticket number on all faxed and emailed documents.

# 13.2 Steps to Determine If an Adverse Event Is To Be Reported In an Expedited Manner

Step 1: Identify the type of adverse event using the current version of the NCI CTCAE V 5.0. The descriptions and grading scales found in the current version of the CTCAE V 5.0 will be used for AE reporting. All appropriate treatment areas should have access to a copy of the CTCAE v5.0. A copy of the CTCAE v5.0 can be downloaded from the CTEP website (<a href="http://ctep.cancer.gov">http://ctep.cancer.gov</a>).

Step 2: Grade the adverse event using the NCI CTCAE v5.0.

Step 3: Review Table A in this section to determine if:

- the adverse event is considered serious;
- there are any protocol-specific requirements for expedited reporting of specific adverse events that require special monitoring; and/or
- there are any protocol-specific exceptions to the reporting requirements.
- Any medical event equivalent to CTCAE v5.0 grade 3, 4, or 5 that precipitates hospitalization (or prolongation of existing hospitalization) must be reported regardless of attribution and designation as expected or unexpected with the exception of any events identified as protocol-specific expedited adverse event reporting exclusions.
- Any event that results in persistent or significant disabilities/incapacities, congenital anomalies, or birth defects must be reported via CTEP-AERS if the event occurs following treatment with an agent under a CTEP IND.
- Use the NCI protocol number and the protocol-specific patient ID provided during trial registration on all reports.
- As referenced in the CTEP Adverse Events Reporting Requirements, an AE that resolves and then recurs during a subsequent cycle does not require CTEP-AERS



- reporting unless (1) the Grade increases; or (2) hospitalization is associated with the recurring AE.
- Some adverse events require notification **within 24 hours** (refer to Table A) to NCI via the web at <a href="http://ctep.cancer.gov">http://ctep.cancer.gov</a> (telephone CTEP at: 301-897-7497 within 24 hours of becoming aware of the event if the CTEP-AERS 24-Hour Notification web-based application is unavailable). Once internet connectivity is restored, a 24-hour notification phoned in must be entered electronically into CTEP-AERS by the original submitter at the site.
- When the adverse event requires expedited reporting, submit the report within 5 or 7 calendar days of learning of the event (refer to <u>Table A</u>).

Table A: Phase 1 and Early Phase 2 Studies: Expedited Reporting Requirements for Adverse Events that Occur on Studies under an IND/IDE within 30 Days of the Last Administration of the Investigational Agent/Intervention 1,2

#### FDA REPORTING REQUIREMENTS FOR SERIOUS ADVERSE EVENTS (21 CFR Part 312)

**NOTE:** Investigators <u>MUST</u> immediately report to the sponsor <u>ANY</u> Serious Adverse Events, whether or not they are considered related to the investigational agent(s)/intervention (21 CFR 312.64)

An adverse event is considered serious if it results in **ANY** of the following outcomes:

- 1) Death
- 2) A life-threatening adverse event
- An adverse event that results in inpatient hospitalization or prolongation of existing hospitalization for ≥ 24 hours
- 4) A persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions
- 5) A congenital anomaly/birth defect.
- 6) Important Medical Events (IME) that may not result in death, be life threatening, or require hospitalization may be considered serious when, based upon medical judgment, they may jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the outcomes listed in this definition. (FDA, 21 CFR 312.32; ICH E2A and ICH E6).

<u>ALL SERIOUS</u> adverse events that meet the above criteria MUST be immediately reported via CTEP-AERS within the timeframes detailed in the table below.

| Hospitalization | Grade 1 and Grade 2 Timeframes | Grade 3-5<br>Timeframes |
|---|---|---|
| Resulting in<br>Hospitalization<br>≥ 24 hrs | 7 Calendar Days | 24-Hour 5 Calendar |
| Not resulting in<br>Hospitalization<br>≥ 24 hrs | Not required | Days |

**NOTE:** Protocol specific exceptions to expedited reporting of serious adverse events are found in the Specific Protocol Exceptions to Expedited Reporting (SPEER) portion of the CAEPR.

#### Expedited AE reporting timelines are defined as:

- "24-Hour; 5 Calendar Days" The AE must initially be reported via CTEP-AERS within 24 hours of learning of the AE, followed by a complete expedited report within 5 calendar days of the initial 24-hour report.
- "7 Calendar Days" A complete expedited report on the AE must be submitted within 7 calendar days of learning of the AE.

<sup>1</sup>Serious adverse events that occur more than 30 days after the last administration of investigational agent/intervention and have an attribution of possible, probable, or definite require reporting as follows:

Expedited 24-hour notification followed by complete report within 5 calendar days for:

All Grade 3, 4, and Grade 5 AEs

# Expedited 7 calendar day reports for:

• Grade 2 AEs resulting in hospitalization or prolongation of hospitalization



<sup>2</sup> For studies using PET or SPECT IND agents, the AE reporting period is limited to 10 radioactive half-lives, rounded UP to the nearest whole day, after the agent/intervention was last administered. Footnote "1" above applies after this reporting period.

Effective Date: May 5, 2011

## 13.3 Exceptions to CTEP-AERS Expedited Reporting Requirements:

- Myelosuppression, (Grade 1 through Grade 4 adverse events as defined in the table below), does not require expedited reporting, unless it is associated with hospitalization.

| Category | Adverse Events |
|----------------------------|----------------------------|
| INVESTIGATIONS | Platelet count decreased |
| INVESTIGATIONS | White blood cell decreased |
| INVESTIGATIONS | Neutrophil count decreased |
| INVESTIGATIONS | Lymphocyte count decreased |
| BLOOD/LYMPHATICS DISORDERS | Anemia |

- Grade 1 and 2 adverse events listed in the table below do **not** require expedited reporting via CTEP-AERS, unless it is associated with hospitalization.

| Category | Adverse Events |
|------------------------------------|------------------------------------|
| GASTROINTESTINAL DISORDERS | Constipation |
| GASTROINTESTINAL DISORDERS | Oral dysesthesia |
| INVESTIGATIONS | Alanine aminotransferase increased |
| INVESTIGATIONS | Creatinine increased |
| INVESTIGATIONS | Weight Loss |
| METABOLISM AND NUTRITION DISORDERS | Hyperglycemia |
| NERVOUS SYSTEM DISORDERS | Headache |
| NERVOUS SYSTEM DISORDERS | Paresthesia |
| RESPIRATORY, THORACIC AND | Dryammaa |
| MEDIASTINAL DISORDERS | Dyspnea |
| SKIN AND SUBCUTANEOUS TISSUE | Dry skin |
| DISORDERS | Dry skill |
| SKIN AND SUBCUTANEOUS TISSUE | Pruritus |
| DISORDERS | |

- See also the Specific Protocol Exceptions to Expedited Reporting (SPEER) in <u>Section 9.1.8</u> of the protocol.

#### 13.4 Definition of Onset and Resolution of Adverse Events

**Note:** These guidelines below are for reporting adverse events on the COG case report forms and do not alter the guidelines for CTEP-AERS reporting.

- 13.4.1 If an adverse event occurs more than once in a course (cycle) of therapy only the most severe grade of the event should be reported.
- 13.4.2 If an adverse event progresses through several grades during one course of therapy, only the most severe grade should be reported.
- 13.4.3 The duration of the AE is defined as the duration of the highest (most severe) grade of the Adverse Effects.
The world's childhood



- 13.4.4 The resolution date of the AE is defined as the date at which the AE returns to baseline or less than or equal to Grade 1, whichever level is higher (note that the resolution date may therefore be different from the date at which the grade of the AE decreased from its highest grade). If the AE does not return to baseline the resolution date should be recorded as "ongoing."
- 13.4.5 An adverse event that persists from one course to another should only be reported once unless the grade becomes more severe in a subsequent course. An adverse event which resolves and then recurs during a different course, must be reported each course it recurs.

## 13.5 Other Recipients of Adverse Event Reports

- 13.5.1 Events that do not meet the criteria for CTEP-AERS reporting (Section 13.2) should be reported at the end of each cycle using the forms provided in the CRF packet (See Section 14.1).
- 13.5.2 Adverse events determined to be reportable must also be reported according to the local policy and procedures to the Institutional Review Board responsible for oversight of the patient.

## 13.6 Specific Examples for Expedited Reporting

## 13.6.1 Reportable Categories of Death

- Death attributable to a CTCAE v5.0 term.
- Death Neonatal: A disorder characterized by "Newborn deaths occurring during the first 28 days after birth."
- Sudden Death NOS: A sudden (defined as instant or within one hour of the onset of symptoms) or an unobserved cessation of life that cannot be attributed to a CTCAE v5.0 term associated with Grade 5.
- Death NOS: A cessation of life that cannot be attributed to a CTCAE term associated with Grade 5.
- Death due to progressive disease should be reported as *Grade 5 "Disease progression"* under the system organ class (SOC) of "*General disorders and administration site conditions*." Evidence that the death was a manifestation of underlying disease (*e.g.*, radiological changes suggesting tumor growth or progression: clinical deterioration associated with a disease process) should be submitted.
- Any death occurring within 30 days of the last dose, regardless of attribution to the investigational agent/intervention requires expedited reporting within 24 hours.
- Any death that occurs more than 30 days after the last dose of treatment with an investigational agent which can be attributed (possibly, probably, or definitely) to the agent and is not clearly due to progressive disease must be reported via CTEP-AERS per the timelines outlined in the table above.

This protocol is for research purposes only. See page 1 for usage policy. APEC1621D

## 13.6.2 Reporting Secondary Malignancy

# Secondary Malignancy:

A secondary malignancy is a cancer caused by treatment for a previous malignancy (e.g., treatment with investigational agent/intervention, radiation or chemotherapy). A secondary malignancy is not considered a metastasis of the initial neoplasm.

CTEP requires all secondary malignancies that occur following treatment with an agent under an NCI IND/IDE be reported via CTEP-AERS. Three options are available to describe the event:

- 1) Leukemia secondary to oncology chemotherapy (e.g., acute myelocytic leukemia [AML])
- 2) Myelodysplastic syndrome (MDS)
- 3) Treatment-related secondary malignancy.

Any malignancy possibly related to cancer treatment (including AML/MDS) should also be reported via the routine reporting mechanisms outlined in each protocol.

# Second Malignancy:

A *second malignancy* is one unrelated to the treatment of a prior malignancy (and is **NOT** a metastasis from the initial malignancy). Second malignancies require **ONLY** routine reporting via CDUS unless otherwise specified.

## 13.6.3 Reporting Pregnancy, Pregnancy Loss, and Death Neonatal

When submitting CTEP-AERS reports for "Pregnancy", "Pregnancy loss", or "Neonatal loss", the Pregnancy Information Form, available at: <a href="http://ctep.cancer.gov/protocolDevelopment/electronic applications/docs/PregnancyReportForm.pdf">http://ctep.cancer.gov/protocolDevelopment/electronic applications/docs/PregnancyReportForm.pdf</a>, needs to be completed and faxed along with any additional medical information to (301) 230-0159. The potential risk of exposure of the fetus to the investigational agent should be documented in the "Description of Event" section of the CTEP-AERS report.

<u>Pregnancy</u>: Patients who become pregnant on study risk intrauterine exposure of the fetus to agents that may be teratogenic. For this reason, pregnancy needs to be reported in an expedited manner via CTEP-AERS as **Grade 3** "*Pregnancy*, puerperium and perinatal conditions - Other (pregnancy)" under the *Pregnancy*, puerperium and perinatal conditions SOC.

Pregnancy needs to be followed **until the outcome of the pregnancy is known** at intervals deemed appropriate by her physicians. The "Pregnancy Information Form" should be used for all necessary follow-ups. This form is available at <a href="http://ctep.cancer.gov/protocolDevelopment/electronic applications/docs/PregnancyReportForm.pdf">http://ctep.cancer.gov/protocolDevelopment/electronic applications/docs/PregnancyReportForm.pdf</a>. If the baby is born with a birth defect or anomaly, then a second CTEP-AERS report is required.

Any pregnancy loss needs to be reported expeditiously, as **Grade 4** "*Pregnancy*, puerperium and perinatal conditions - Other (pregnancy loss)". Do NOT report a pregnancy loss as a Grade 5 event since CTEP-AERS recognizes any Grade 5



event as a patient death.

<u>Death Neonatal</u>: Neonatal death, defined in CTCAE v5.0 as "Newborn deaths occurring during the first 28 days after birth" that is felt by the investigator to be at least possibly due to the investigational agent/intervention, should be reported expeditiously, as **Grade 4** "Death Neonatal" under the system organ class (SOC) of "General disorders and administration site conditions." When the death is the result of a patient pregnancy or pregnancy in partners of men on study. Do NOT report a neonatal death resulting from a patient pregnancy or pregnancy in partners of men on study as a Grade 5 event since CTEP-AERS recognizes any Grade 5 event as a patient death.

# 14.0 RECORDS, REPORTING, AND DATA AND SAFETY MONITORING PLAN

#### 14.1 Categories of Research Records

Research records for this study can be divided into three categories

- 1. Non-computerized Information: Roadmaps, Pathology Reports, Surgical Reports. These forms are uploaded into RAVE.
- 2. Reference Labs, Biopathology Reviews, and Imaging Center data: These data accompany submissions to these centers, which forward their data electronically to the COG Statistics & Data Center.
- 3. Computerized Information Electronically Submitted: All other data will be entered in RAVE with the aid of schedules and worksheets (essentially paper copies of the OPEN and RAVE screens) provided in the case report form (CRF) packet.

See separate CRF Packet, which includes submission schedule.

#### 14.2 **CDUS**

This study will be monitored by the Clinical Data Update System (CDUS) version 3.0. Cumulative protocol- and patient-specific CDUS data will be submitted electronically to CTEP on a quarterly basis by FTP burst of data. Reports are due January 31, April 30, July 31 and October 31. Instructions for submitting data using the CDUS can be found on the CTEP Web site (http://ctep.cancer.gov/reporting/cdus.html).

Note: This study has been assigned to CDUS-Complete reporting, all adverse events (both routine and expedited) that have occurred on the study and meet the mandatory CDUS reporting guidelines must be reported via the monitoring method identified above.

## 14.3 CRADA/CTA/CSA

The agent(s) supplied by CTEP, DCTD, NCI used in this protocol is/are provided to the NCI under a Collaborative Agreement (CRADA, CTA, CSA) between the Pharmaceutical Company(ies) (hereinafter referred to as "Collaborator(s)") and the NCI Division of Cancer Treatment and Diagnosis. Therefore, the following obligations/guidelines, in addition to the provisions in the "Intellectual Property Option to Collaborator" (http://ctep.cancer.gov/industryCollaborations2/intellectual property.htm) contained

The world's childhood



within the terms of award, apply to the use of the Agent(s) in this study:

- 1. Agent(s) may not be used for any purpose outside the scope of this protocol, nor can Agent(s) be transferred or licensed to any party not participating in the clinical study. Collaborator(s) data for Agent(s) are confidential and proprietary to Collaborator(s) and shall be maintained as such by the investigators. The protocol documents for studies utilizing investigational Agents contain confidential information and should not be shared or distributed without the permission of the NCI. If a copy of this protocol is requested by a patient or patient's family member participating on the study, the individual should sign a confidentiality agreement. A suitable model agreement can be downloaded from: http://ctep.cancer.gov.
- 2. For a clinical protocol where there is an investigational Agent used in combination with (an)other investigational Agent(s), each the subject of different collaborative agreements, the access to and use of data by each Collaborator shall be as follows (data pertaining to such combination use shall hereinafter be referred to as "Multi-Party Data"):
  - a. NCI will provide all Collaborators with prior written notice regarding the existence and nature of any agreements governing their collaboration with NIH, the design of the proposed combination protocol, and the existence of any obligations that would tend to restrict NCI's participation in the proposed combination protocol.
  - b. Each Collaborator shall agree to permit use of the Multi-Party Data from the clinical trial by any other Collaborator solely to the extent necessary to allow said other Collaborator to develop, obtain regulatory approval or commercialize its own investigational Agent.
  - c. Any Collaborator having the right to use the Multi-Party Data from these trials must agree in writing prior to the commencement of the trials that it will use the Multi-Party Data solely for development, regulatory approval, and commercialization of its own investigational Agent.
- 3. Clinical Trial Data and Results and Raw Data developed under a Collaborative Agreement will be made available exclusively to Collaborator(s), the NCI, and the FDA, as appropriate and unless additional disclosure is required by law or court order described IP Option Collaborator as the (http://ctep.cancer.gov/industryCollaborations2/intellectual property.htm). Additionally, all Clinical Data and Results and Raw Data will be collected, used and disclosed consistent with all applicable federal statutes and regulations for the protection of human subjects, including, if applicable, the Standards for Privacy of Individually Identifiable Health Information set forth in 45 C.F.R. Part 164.
- 4. When a Collaborator wishes to initiate a data request, the request should first be sent to the NCI, who will then notify the appropriate investigators (Group Chair for Cooperative Group studies, or PI for other studies) of Collaborator's wish to contact them.
- 5. Any data provided to Collaborator(s) for Phase 3 studies must be in accordance with the guidelines and policies of the responsible Data Monitoring Committee (DMC), if there is a DMC for this clinical trial.



6. Any manuscripts reporting the results of this clinical trial must be provided to CTEP for immediate delivery to Collaborator(s) for advisory review and comment prior to submission for publication. Collaborator(s) will have 30 days from the date of receipt for review. Collaborator shall have the right to request that publication be delayed for up to an additional 30 days in order to ensure that Collaborator's confidential and proprietary data, in addition to Collaborator(s)'s intellectual property rights, are protected. Copies of abstracts must be provided to CTEP for forwarding to Collaborator(s) for courtesy review as soon as possible and preferably at least three (3) days prior to submission, but in any case, prior to presentation at the meeting or publication in the proceedings. Press releases and other media presentations must also be forwarded to CTEP prior to release. Copies of any manuscript, abstract and/or press release/ media presentation should be sent to: Email: ncicteppubs@mail.nih.gov

The Regulatory Affairs Branch will then distribute them to Collaborator(s). No publication, manuscript or other form of public disclosure shall contain any of Collaborator's confidential/proprietary information.

## 14.4 Data and Safety Monitoring Plan

Data and safety is ensured by several integrated components including the COG Data and Safety Monitoring Committee.

#### 14.4.1 Data and Safety Monitoring Committee

This study will be monitored in accordance with the Children's Oncology Group policy for data and safety monitoring of Phase 1 and 2 studies. In brief, the role of the COG Data and Safety Monitoring Committee is to protect the interests of patients and the scientific integrity for all Phase 1 and 2 studies. The DSMC consists of a chair; a statistician external to COG; one external member; one consumer representative; the lead statistician of the developmental therapy scientific committee; and a member from the NCI. The DSMC meets at least every 6 months to review current study results, as well as data available to the DSMC from other related studies. Approximately 6 weeks before each meeting of the Phase 1 and 2 DSMC, study chairs will be responsible for working with the study statistician to prepare study reports for review by the DSMC. The DSMC will provide recommendations to the COG Developmental Therapeutics Chair and the Group Chair for each study reviewed to change the study or to continue the study unchanged. Data and Safety Committee reports for institutional review boards can be prepared using the public data monitoring report as posted on the COG Web site.

#### 14.4.2 Monitoring by the Study Chair and MATCH Leadership

The study chair will monitor the study regularly and enter evaluations of patients' eligibility, evaluability, and dose limiting toxicities into the study database. In addition, study data and the study chair's evaluations will be reviewed by the MATCH Chair, Vice Chair and Statistician on a weekly conference call.



#### **REFERENCES**

- 1. Agaram NP, Chen CL, Zhang L, LaQuaglia MP, Wexler L, Antonescu CR. Recurrent MYOD1 mutations in pediatric and adult sclerosing and spindle cell rhabdomyosarcomas: evidence for a common pathogenesis. *Genes Chromosomes Cancer*. 2014;53(9):779-787.
- 2. Grill J, Puget S, Andreiuolo F, Philippe C, MacConaill L, Kieran MW. Critical oncogenic mutations in newly diagnosed pediatric diffuse intrinsic pontine glioma. *Pediatr Blood Cancer*. 2012;58(4):489-491.
- 3. Perry JA, Kiezun A, Tonzi P, et al. Complementary genomic approaches highlight the PI3K/mTOR pathway as a common vulnerability in osteosarcoma. *Proceedings of the National Academy of Sciences of the United States of America*. 2014;111(51):E5564-5573.
- 4. Shern JF, Chen L, Chmielecki J, et al. Comprehensive genomic analysis of rhabdomyosarcoma reveals a landscape of alterations affecting a common genetic axis in fusion-positive and fusion-negative tumors. *Cancer discovery*. 2014;4(2):216-231.
- 5. Parsons DW, Roy A, Yang Y, et al. Diagnostic Yield of Clinical Tumor and Germline Whole-Exome Sequencing for Children With Solid Tumors. *JAMA oncology*. 2016.
- 6. Harris MH, DuBois SG, Glade Bender JL, et al. Multicenter Feasibility Study of Tumor Molecular Profiling to Inform Therapeutic Decisions in Advanced Pediatric Solid Tumors: The Individualized Cancer Therapy (iCat) Study. *JAMA oncology*. 2016.
- 7. Hoogeveen-Westerveld M, Wentink M, van den Heuvel D, et al. Functional assessment of variants in the TSC1 and TSC2 genes identified in individuals with Tuberous Sclerosis Complex. *Human mutation*. 2011;32(4):424-435.
- 8. Weigelt B, Downward J. Genomic Determinants of PI3K Pathway Inhibitor Response in Cancer. *Front Oncol.* 2012;2:109.
- 9. Brachmann SM, Hofmann I, Schnell C, et al. Specific apoptosis induction by the dual PI3K/mTor inhibitor NVP-BEZ235 in HER2 amplified and PIK3CA mutant breast cancer cells. *Proceedings of the National Academy of Sciences of the United States of America*. 2009;106(52):22299-22304.
- 10. Di Nicolantonio F, Arena S, Tabernero J, et al. Deregulation of the PI3K and KRAS signaling pathways in human cancer cells determines their response to everolimus. *The Journal of clinical investigation*. 2010;120(8):2858-2866.
- 11. Lehmann BD, Bauer JA, Chen X, et al. Identification of human triple-negative breast cancer subtypes and preclinical models for selection of targeted therapies. *The Journal of clinical investigation*. 2011;121(7):2750-2767.
- 12. O'Brien C, Wallin JJ, Sampath D, et al. Predictive biomarkers of sensitivity to the phosphatidylinositol 3' kinase inhibitor GDC-0941 in breast cancer preclinical models. *Clinical cancer research : an official journal of the American Association for Cancer Research.* 2010;16(14):3670-3683.
- 13. Sanchez CG, Ma CX, Crowder RJ, et al. Preclinical modeling of combined phosphatidylinositol-3-kinase inhibition with endocrine therapy for estrogen receptor-positive breast cancer. *Breast Cancer Res.* 2011;13(2):R21.
- 14. Serra V, Markman B, Scaltriti M, et al. NVP-BEZ235, a dual PI3K/mTOR inhibitor, prevents PI3K signaling and inhibits the growth of cancer cells with activating PI3K mutations. *Cancer Res.* 2008;68(19):8022-8030.
- 15. She QB, Chandarlapaty S, Ye Q, et al. Breast tumor cells with PI3K mutation or HER2 amplification are selectively addicted to Akt signaling. *PloS one.* 2008;3(8):e3065.
- 16. Weigelt B, Warne PH, Downward J. PIK3CA mutation, but not PTEN loss of function, determines the sensitivity of breast cancer cells to mTOR inhibitory drugs. *Oncogene*. 2011;30(29):3222-3233.
- 17. Tanaka H, Yoshida M, Tanimura H, et al. The selective class I PI3K inhibitor CH5132799 targets human cancers harboring oncogenic PIK3CA mutations. *Clin Cancer Res.* 2011;17(10):3272-3281.
- 18. Yu K, Toral-Barza L, Shi C, Zhang WG, Zask A. Response and determinants of cancer cell susceptibility to PI3K inhibitors: combined targeting of PI3K and Mek1 as an effective anticancer



- strategy. Cancer Biol Ther. 2008;7(2):307-315.
- 19. Engelman JA, Luo J, Cantley LC. The evolution of phosphatidylinositol 3-kinases as regulators of growth and metabolism. *Nat Rev Genet*. 2006;7(8):606-619.
- 20. Jia S, Liu Z, Zhang S, et al. Essential roles of PI(3)K-p110beta in cell growth, metabolism and tumorigenesis. *Nature*. 2008;454(7205):776-779.
- 21. Wee S, Wiederschain D, Maira SM, et al. PTEN-deficient cancers depend on PIK3CB. *Proc Natl Acad Sci U S A*. 2008;105(35):13057-13062.
- 22. Edgar KA, Wallin JJ, Berry M, et al. Isoform-specific phosphoinositide 3-kinase inhibitors exert distinct effects in solid tumors. *Cancer Res.* 2010;70(3):1164-1172.
- 23. Franz DN, Belousova E, Sparagana S, et al. Efficacy and safety of everolimus for subependymal giant cell astrocytomas associated with tuberous sclerosis complex (EXIST-1): a multicentre, randomised, placebo-controlled phase 3 trial. *Lancet*. 2013;381(9861):125-132.
- 24. Kingswood JC, Jozwiak S, Belousova ED, et al. The effect of everolimus on renal angiomyolipoma in patients with tuberous sclerosis complex being treated for subependymal giant cell astrocytoma: subgroup results from the randomized, placebo-controlled, Phase 3 trial EXIST-1. *Nephrol Dial Transplant*. 2014;29(6):1203-1210.
- 25. Kwiatkowski DJ, Choueiri TK, Fay AP, et al. Mutations in TSC1, TSC2, and MTOR Are Associated with Response to Rapalogs in Patients with Metastatic Renal Cell Carcinoma. *Clinical cancer research: an official journal of the American Association for Cancer Research.* 2016;22(10):2445-2452.
- 26. Iyer G, Hanrahan AJ, Milowsky MI, et al. Genome sequencing identifies a basis for everolimus sensitivity. *Science (New York, NY)*. 2012;338(6104):221.
- 27. Voss MH, Hakimi AA, Pham CG, et al. Tumor genetic analyses of patients with metastatic renal cell carcinoma and extended benefit from mTOR inhibitor therapy. *Clinical cancer research : an official journal of the American Association for Cancer Research.* 2014;20(7):1955-1964.
- 28. Janku F, Tsimberidou AM, Garrido-Laguna I, et al. PIK3CA mutations in patients with advanced cancers treated with PI3K/AKT/mTOR axis inhibitors. *Mol Cancer Ther*. 2011;10(3):558-565.
- 29. Garrido-Laguna I, Hong DS, Janku F, et al. KRASness and PIK3CAness in patients with advanced colorectal cancer: outcome after treatment with early-phase trials with targeted pathway inhibitors. *PloS one.* 2012;7(5):e38033.
- 30. Janku F, Wheler JJ, Naing A, et al. PIK3CA mutation H1047R is associated with response to PI3K/AKT/mTOR signaling pathway inhibitors in early-phase clinical trials. *Cancer Res.* 2013;73(1):276-284.
- 31. Moroney JW, Schlumbrecht MP, Helgason T, et al. A phase I trial of liposomal doxorubicin, bevacizumab, and temsirolimus in patients with advanced gynecologic and breast malignancies. *Clinical cancer research : an official journal of the American Association for Cancer Research.* 2011;17(21):6840-6846.
- 32. Hortobagyi GN, Chen D, Piccart M, et al. Correlative Analysis of Genetic Alterations and Everolimus Benefit in Hormone Receptor-Positive, Human Epidermal Growth Factor Receptor 2-Negative Advanced Breast Cancer: Results From BOLERO-2. *Journal of clinical oncology : official journal of the American Society of Clinical Oncology.* 2016;34(5):419-426.
- 33. Janku F, Wheler JJ, Westin SN, et al. PI3K/AKT/mTOR inhibitors in patients with breast and gynecologic malignancies harboring PIK3CA mutations. *Journal of clinical oncology : official journal of the American Society of Clinical Oncology*. 2012;30(8):777-782.
- Wagle N, Grabiner BC, Van Allen EM, et al. Activating mTOR mutations in a patient with an extraordinary response on a phase I trial of everolimus and pazopanib. *Cancer discovery*. 2014;4(5):546-553.
- Engelman JA, Chen L, Tan X, et al. Effective use of PI3K and MEK inhibitors to treat mutant Kras G12D and PIK3CA H1047R murine lung cancers. *Nature medicine*. 2008;14(12):1351-1356.
- 36. Ihle NT, Lemos R, Jr., Wipf P, et al. Mutations in the phosphatidylinositol-3-kinase pathway predict for antitumor activity of the inhibitor PX-866 whereas oncogenic Ras is a dominant



- predictor for resistance. Cancer Res. 2009;69(1):143-150.
- 37. Meuillet EJ, Zuohe S, Lemos R, et al. Molecular pharmacology and antitumor activity of PHT-427, a novel Akt/phosphatidylinositide-dependent protein kinase 1 pleckstrin homology domain inhibitor. *Mol Cancer Ther.* 2010;9(3):706-717.
- 38. Garnett MJ, Edelman EJ, Heidorn SJ, et al. Systematic identification of genomic markers of drug sensitivity in cancer cells. *Nature*. 2012;483(7391):570-575.
- 39. Janku F, Lee JJ, Tsimberidou AM, et al. PIK3CA Mutations Frequently Coexist with RAS and BRAF Mutations in Patients with Advanced Cancers. *PloS one*. 2011;6(7).
- 40. Houghton PJ, Morton CL, Kolb EA, et al. Initial testing (stage 1) of the mTOR inhibitor rapamycin by the pediatric preclinical testing program. *Pediatr Blood Cancer*. 2008;50(4):799-805.
- 41. Reynolds CP, Kang MH, Carol H, et al. Initial testing (stage 1) of the phosphatidylinositol 3' kinase inhibitor, SAR245408 (XL147) by the pediatric preclinical testing program. *Pediatr Blood Cancer*. 2013;60(5):791-798.
- 42. Kang MH, Reynolds CP, Maris JM, et al. Initial testing (stage 1) of the investigational mTOR kinase inhibitor MLN0128 by the pediatric preclinical testing program. *Pediatr Blood Cancer*. 2014;61(8):1486-1489.
- 43. Houghton PJ, Gorlick R, Kolb EA, et al. Initial testing (stage 1) of the mTOR kinase inhibitor AZD8055 by the pediatric preclinical testing program. *Pediatr Blood Cancer*. 2012;58(2):191-199.
- 44. Mascarenhas LM, W.H; Lyden, E; Rodeberg, D.A; Indelicato, D. J.; Linardic, C. M.; Anderson, R.; Hawkins, D.S. Randomized phase II trial of bevacizumab and temsirolimus in combination with vinorelbine (V) and cylcophosphamide (C) for first relapse/disease progression of rhabdomyosarcoma (RMS): A report from the Children's Oncology Group. American Society of Oncology Annual Meeting; 2014.
- 45. Noh WC, Mondesire WH, Peng J, et al. Determinants of rapamycin sensitivity in breast cancer cells. *Clinical cancer research : an official journal of the American Association for Cancer Research*. 2004;10(3):1013-1023.
- 46. Meric-Bernstam F, Akcakanat A, Chen H, et al. PIK3CA/PTEN mutations and Akt activation as markers of sensitivity to allosteric mTOR inhibitors. *Clinical cancer research : an official journal of the American Association for Cancer Research.* 2012;18(6):1777-1789.
- 47. Iwenofu OH, Lackman RD, Staddon AP, Goodwin DG, Haupt HM, Brooks JS. Phospho-S6 ribosomal protein: a potential new predictive sarcoma marker for targeted mTOR therapy. *Modern pathology: an official journal of the United States and Canadian Academy of Pathology, Inc.* 2008;21(3):231-237.
- 48. Behbakht K, Sill MW, Darcy KM, et al. Phase II trial of the mTOR inhibitor, temsirolimus and evaluation of circulating tumor cells and tumor biomarkers in persistent and recurrent epithelial ovarian and primary peritoneal malignancies: a Gynecologic Oncology Group study. *Gynecol Oncol.* 2011;123(1):19-26.
- 49. Galanis E, Buckner JC, Maurer MJ, et al. Phase II trial of temsirolimus (CCI-779) in recurrent glioblastoma multiforme: a North Central Cancer Treatment Group Study. *Journal of clinical oncology: official journal of the American Society of Clinical Oncology.* 2005;23(23):5294-5304.
- 50. Tarhini A, Kotsakis A, Gooding W, et al. Phase II study of everolimus (RAD001) in previously treated small cell lung cancer. *Clinical cancer research : an official journal of the American Association for Cancer Research.* 2010;16(23):5900-5907.
- 51. Cho D, Signoretti S, Dabora S, et al. Potential histologic and molecular predictors of response to temsirolimus in patients with advanced renal cell carcinoma. *Clin Genitourin Cancer*. 2007;5(6):379-385.
- 52. Chawla SP, Staddon AP, Baker LH, et al. Phase II study of the mammalian target of rapamycin inhibitor ridaforolimus in patients with advanced bone and soft tissue sarcomas. *Journal of clinical oncology: official journal of the American Society of Clinical Oncology.* 2012;30(1):78-84.
- 53. Soria JC, Shepherd FA, Douillard JY, et al. Efficacy of everolimus (RAD001) in patients with advanced NSCLC previously treated with chemotherapy alone or with chemotherapy and EGFR



- inhibitors. Ann Oncol. 2009;20(10):1674-1681.
- 54. Ellard SL, Clemons M, Gelmon KA, et al. Randomized phase II study comparing two schedules of everolimus in patients with recurrent/metastatic breast cancer: NCIC Clinical Trials Group IND.163. *Journal of clinical oncology: official journal of the American Society of Clinical Oncology.* 2009;27(27):4536-4541.
- 55. Lilly. LY3023414 Investigator's Brochure. 2015.
- 56. Smith GC, Ong WK, Rewcastle GW, Kendall JD, Han W, Shepherd PR. Effects of acutely inhibiting PI3K isoforms and mTOR on regulation of glucose metabolism in vivo. *The Biochemical journal*. 2012;442(1):161-169.
- 57. Blumenthal G, Orbach R, Zineh I, Cortazar P, Justice R, Pazdur R. Early targeted drug development: Pilot FDA review of PI3K inhibitor phase I studies using a knowledge management database. *J Clin Oncol (Meeting Abstracts)*. 2011;29(suppl):Abstract 3060.
- 58. Schwartz GJ, Gauthier B. A simple estimate of glomerular filtration rate in adolescent boys. *J Pediatr.* 1985;106(3):522-526.
- 59. This table will be updated as the toxicity profile of the agent is revised. Updates will be distributed to all Principal Investigators at the time of revision. The current version can be obtained by contacting PIO@CTEP.NCI.NIH.GOV. Your name, the name of the investigator, the protocol and the agent should be included in the e-mail. In.
- 60. A'Hern RP. Sample size tables for exact single-stage phase II designs. *Stat Med.* 2001;20(6):859-866.
- 61. Agresti A, Coull BA. Approximate Is Better than "Exact" for Interval Estimation of Binomial Proportions. *The American Statistician*. 1998;52(2):119-126.
- 62. Eisenhauer EA, Therasse P, Bogaerts J, et al. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). *Eur J Cancer*. 2009;45(2):228-247.
- 63. Sandlund JT, Guillerman RP, Perkins SL, et al. International Pediatric Non-Hodgkin Lymphoma Response Criteria. *Journal of clinical oncology : official journal of the American Society of Clinical Oncology*. 2015;33(18):2106-2111.
- 64. Cheson BD, Fisher RI, Barrington SF, et al. Recommendations for initial evaluation, staging, and response assessment of Hodgkin and non-Hodgkin lymphoma: the Lugano classification. *Journal of clinical oncology: official journal of the American Society of Clinical Oncology.* 2014;32(27):3059-3068.

The world's childhood



# APPENDIX I: PERFORMANCE STATUS SCALES/SCORES

| Karnofsky | | Lansk | y |
|---|---|---|---|
| Score | Description | Score | Description |
| 100 | Normal, no complaints, no evidence of disease | 100 | Fully active, normal. |
| 90 | Able to carry on normal activity, minor signs or symptoms of disease. | 90 | Minor restrictions in physically strenuous activity. |
| 80 | Normal activity with effort; some signs or symptoms of disease. | 80 | Active, but tires more quickly |
| 70 | Cares for self, unable to carry on normal activity or do active work. | 70 | Both greater restriction of and less time spent in play activity. |
| 60 | Required occasional assistance, but is able to care for most of his/her needs. | 60 | Up and around, but minimal active play; keeps busy with quieter activities. |
| 50 | Requires considerable assistance and frequent medical care. | 50 | Gets dressed, but lies around much of the day; no active play, able to participate in all quiet play and activities. |
| 40 | Disabled, requires special care and assistance. | 40 | Mostly in bed; participates in quiet activities. |
| 30 | Severely disabled, hospitalization indicated. Death not imminent. | 30 | In bed; needs assistance even for quiet play. |
| 20 | Very sick, hospitalization indicated. Death not imminent. | 20 | Often sleeping; play entirely limited to very passive activities. |
| 10 | Moribund, fatal processes progressing rapidly. | 10 | No play; does not get out of bed. |



# APPENDIX II: CYP3A4 SUBSTRATES, INDUCERS AND INHIBITORS

This is not an inclusive list. Because the lists of these agents are constantly changing, it is important to regularly consult frequently updated medical references.

| CYP3A4 substrates | Strong | Moderate | Strong | Moderate |
|---|---|---|---|---|
| | Inhibitors <sup>1</sup> | Inhibitors | Inducers | Inducers |
| abemaciclib | atazanavir | aprepitant | apalutamide | bosentan |
| acalabrutinib <sup>5</sup> | boceprevir | conivaptan | barbiturates | cenobamate |
| alfentanil <sup>4,5</sup> | clarithromycin | crizotinib | carbamazepin | dabrafenib |
| alprazolam <sup>5</sup> | ceritinib | diltiazem | e | efavirenz |
| amiodarone <sup>4</sup> | cobicistat | dronedarone | enzalutamide<br>fosphenytoin | eslicarbazepine<br>etravirine |
| amlodapine | danoprevir/ritonav | duvelisib | lumacaftor/ | lorlatinib |
| aprepitant/fosaprepitant | ir | erythromycin | ivacaftor | modafinil |
| atorvastatin <sup>5</sup> | darunavir | fedratinib | mitotane | nafcillin |
| avanafil <sup>5</sup> | delavirdine | fluconazole | phenobarbital | pexidartinib |
| axitinib | elivitegravir/ritona | fosamprenavir | phenytoin | rifabutin |
| bortezomib | vir | fosnetupitant | primidone | rifapentin |
| bosutinib <sup>5</sup> | grapefruit <sup>3</sup> | grapefruit <sup>3</sup> | rifampin<br>St. John's wort | |
| brexpiprazole | grapefruit juice <sup>3</sup> | grapefruit juice <sup>3</sup> | St. John's wort | |
| brigatinib | idelalisib | imatinib | | |
| budesonide <sup>5</sup> | indinavir/ritonavir | isavuconazole | | |
| buspirone <sup>5</sup> | itraconazole | lefamulin | | |
| calcium channel blockers | ketoconazole | letermovir | | |
| cisapride | lopinavir/ritonavir<br>ombitasvi +/- | mifepristone | | |
| citalopram/escitalopram | ombitasvi +/-<br>dasabuvir | netupitant<br>nilotinib | | |
| cobimetinib <sup>5</sup> | nefazodone | ribociclib | | |
| colchicine <sup>5</sup> | nelfinavir | verapamil | | |
| conivaptan <sup>5</sup> | paritaprevir/ritona | Verapaiiii | | |
| copanlisib | vir | | | |
| crizotinib | posaconazole | | | |
| cyclosporine <sup>4</sup> | ritonavir | | | |
| dabrafenib | saquinavir | | | |
| dapsone | telaprevir | | | |
| darifenacin <sup>5</sup> | telithromycin | | | |
| darunavir <sup>5</sup> | tipranavir/ritonavir | | | |
| dasatinib <sup>5</sup> | tucatinib | | | |
| dexamethasone <sup>2</sup> | voriconazole | | | |
| diazepam | | | | |
| dihydroergotamine | | | | |
| docetaxel | | | | |
| doxorubicin | | | | |
| dronedarone <sup>5</sup> | | | | |
| ebastine <sup>5</sup> | | | | |
| eletriptan <sup>5</sup> | | | | |
| eliglustat <sup>5</sup> | | | | |
| eplerenone <sup>5</sup> | | | | |
| ergotamine <sup>4</sup> | | | | |
| erlotinib | | | | |
| estrogens | | | | |
| etoposide | | | | |

| CHILDREN'S |
|------------|
| ONCOLOGY |
| GROUP |

| 1* 5 | T | |
|----------------------------|---|------|
| everolimus <sup>5</sup> | | |
| felodipine <sup>5</sup> | | |
| fentany1 <sup>4</sup> | | |
| gefitinib | | |
| haloperidol | | |
| ibrutinib <sup>5</sup> | | |
| idelalisib | | |
| imatinib | | |
| indinavir <sup>5</sup> | | |
| irinotecan | | |
| isavuconazole <sup>5</sup> | | |
| itraconazole | | |
| ivacaftor | | |
| ketoconazole | | |
| lansoprazole | | |
| lapatinib | | |
| lomitapide <sup>5</sup> | | |
| lorlatinib | | |
| losartan | | |
| lovastatin <sup>5</sup> | | |
| lurasidone <sup>5</sup> | | |
| macrolide antibiotics | | |
| maraviroc <sup>5</sup> | | |
| medroxyprogesterone | | |
| methadone | | |
| midazolam <sup>5</sup> | | |
| midostaurin <sup>5</sup> | | |
| modafinil | | |
| naloxegol <sup>5</sup> | | |
| nefazodone | | |
| nilotinib | | |
| olaparib | | |
| ondansetron | | |
| osimertinib | | |
| paclitaxel | | |
| palbociclib | | |
| pazopanib | | |
| pimozide <sup>5</sup> | | |
| quetiapine <sup>5</sup> | | |
| quinidine <sup>4</sup> | | |
| regorafenib | | |
| rilpivirine <sup>5</sup> | | |
| rivaroxaban <sup>5</sup> | | |
| romidepsin | | |
| saquinavir <sup>5</sup> | | |
| sildenafil <sup>5</sup> | | |
| simvastatin <sup>5</sup> | | |
| sirolimus <sup>4,5</sup> | | |
| sonidegib | | |
| sunitinib | | |
| tacrolimus <sup>4,5</sup> | | <br> |
| | | <br> |



THIS PROTOCOL IS FOR RESEARCH PURPOSES ONLY. SEE PAGE 1 FOR USAGE POLICY. APEC 1621D

| tamoxifen |
|-------------------------|
| tadalafil <sup>5</sup> |
| telaprevir |
| temsirolimus |
| teniposide |
| tetracycline |
| ticagrelor <sup>5</sup> |
| tipranavir <sup>5</sup> |
| tolvaptan <sup>5</sup> |
| triazolam <sup>5</sup> |
| trimethoprim |
| vardenafil <sup>5</sup> |
| vemurafenib |
| venetoclax <sup>5</sup> |
| vinca alkaloids |
| zolpidem |

<sup>&</sup>lt;sup>1</sup> Certain fruits, fruit juices and herbal supplements (star fruit, Seville oranges, pomegranate, gingko, goldenseal) may inhibit CYP 3A4 isozyme, however, the degree of that inhibition is unknown.

<sup>&</sup>lt;sup>2</sup>Refer to Section 7.5 regarding use of corticosteroids. Dexamethasone is considered a weak CYP3A4 inducer.

<sup>&</sup>lt;sup>3</sup>The effect of grapefruit juice (strong vs moderate CYP3A4 inhibition) varies widely among brands and is concentration-, dose-, and preparation-dependent.

<sup>&</sup>lt;sup>4</sup>Narrow therapeutic range substrates

<sup>&</sup>lt;sup>5</sup>Sensitive substrates



#### APPENDIX III-A: MEDICATION DIARY FOR LY3023414

| COG Patient ID: | Acc# | Institution : |
|-------------------------------|--------------------|---------------|
| Please do not write patient n | ames on this form. | |

Complete each day with the time and dose given for LY3023414. If a dose is not due or is accidentally skipped leave that day blank. *Make note of other drugs and supplements taken under the Comments section below*. LY3023414 tablets should not be cut, dissolved or crushed but should be swallowed whole. If the tablet is crushed and the drug gets on skin, wash the exposed area with as much water as necessary. Inform your study doctor or nurse if that occurs. LY3023414 should be taken without regard to meals, with a glass of water. You should take LY3023414, at about the same time each day. If you vomit after taking the medication, the dose should not be repeated. This should be noted in the comments section. If you forget a dose and remember it within 6 hours of the time the dose was due, you should take the dose at that time. If it is less than 6 hours before the next dose, then the forgotten dose should be skipped. Either way, the next dose should be taken at the usual time. Add the dates to the calendar below and return the completed diary to the study clinic at each visit (weekly during Cycle 1, and then after each treatment cycle).

| EXAMPLE | | | Number of LY | 3023414 <i>tablets</i> | Comments |
|---|---|---|---|---|---|
| | Date | Time | 50 mg | 100 mg | |
| Day 1 | 1/15/14 | 8:30 AM | 2 | 1 | He felt nauseated an hour after taking<br>the drug but did not vomit. |

| | Cycle #: Start Date: / / / End Date: _ / / Dose Level:mg/m²/dose | | | | |
|---|---|---|---|---|---|
| | | | | 4 tablets prescribed to take | Comments (Describe any missed or extra doses, vomiting and/or bothersome effects.) |
| WEEK 1 | D-4- | Time | 50 mg | 100 mg | |
| WEEKI | Date | Time | AM# | AM# | |
| | | | PM# | PM# | |
| | | | | 23414 tablets taken | |
| | | | 50 mg | 100 mg | |
| D 1 | | AM | | | |
| Day 1 | 1 P | PM | | | |
| | | AM | | | |
| Day 2 | | PM | | | |
| | | AM | | | |
| Day 3 | | PM | | | |
| D 4 | | AM | | | |
| Day 4 | | PM | | | |
| Day 5 | | AM | | | |
| Day 3 | | PM | | | |
| Day 6 | | AM | | | |
| Day 0 | | PM | | | |
| Day 7 | | AM | | | |
| Day / | | PM | | | |



| | Cycle #: | Start Date: _<br>End Date: | <u>/ </u> | Dose Level: | _mg/m²/dose |
|---|---|---|---|---|---|
| WEEK 3 | Date | # of LY3023414 tablets prescribed to take | | Comments<br>(Describe any missed or extra doses, vomiting<br>and/or bothersome effects.) | |
| WEEK 3 | Date | Time | 50 mg | 100 mg | |
| | | | AM# | AM# | |
| | | AM | PM# | PM# | |
| Day 8 | | PM | | | |
| | | AM | | | |
| Day 9 | | PM | | | |
| Day 10 | - | AM | | | |
| | | PM | | | |
| Day 11 | | AM | | | |
| | | PM | | | |
| Day 12 | - | AM | | | |
| | | PM | | | |
| Day 13 | | AM | | | |
| | | PM | | | |
| Day 14 | | AM | | | |
| · | | PM | | | |
| | | | # of LY302341 | 4 tablets prescribed to take | Comments (Describe any missed or extra doses, vomiting and/or bothersome effects.) |
| | | | 50 mg | take<br>100 mg | (Describe any missed or extra doses, vomiting |
| WEEK 3 | Date | Time | 50 mg<br>AM# | 100 mg AM# | (Describe any missed or extra doses, vomiting |
| WEEK 3 | Date | Time | 50 mg<br>AM#<br>PM# | take<br>100 mg | (Describe any missed or extra doses, vomiting |
| WEEK 3 | Date | Time | 50 mg<br>AM#<br>PM# | 100 mg AM# PM# | (Describe any missed or extra doses, vomiting |
| | Date | Time | 50 mg AM# PM# # of LY302 | 100 mg AM# PM# 3414 tablets taken | (Describe any missed or extra doses, vomiting |
| WEEK 3 Day 15 | Date | AM | 50 mg AM# PM# # of LY302 | 100 mg AM# PM# 3414 tablets taken | (Describe any missed or extra doses, vomiting |
| Day 15 | Date | | 50 mg AM# PM# # of LY302 | 100 mg AM# PM# 3414 tablets taken | (Describe any missed or extra doses, vomiting |
| | Date | AM PM | 50 mg AM# PM# # of LY302 | 100 mg AM# PM# 3414 tablets taken | (Describe any missed or extra doses, vomiting |
| Day 15 | Date | AM PM AM PM | 50 mg AM# PM# # of LY302 | 100 mg AM# PM# 3414 tablets taken | (Describe any missed or extra doses, vomiting |
| Day 15 | Date | AM PM AM PM AM | 50 mg AM# PM# # of LY302 | 100 mg AM# PM# 3414 tablets taken | (Describe any missed or extra doses, vomiting |
| Day 15 Day 16 Day 17 | Date | AM PM AM PM AM PM | 50 mg AM# PM# # of LY302 | 100 mg AM# PM# 3414 tablets taken | (Describe any missed or extra doses, vomiting |
| Day 15 | Date | AM PM AM PM AM PM AM AM | 50 mg AM# PM# # of LY302 | 100 mg AM# PM# 3414 tablets taken | (Describe any missed or extra doses, vomiting |
| Day 15 Day 16 Day 17 Day 18 | Date | AM PM AM PM AM PM AM PM AM PM | 50 mg AM# PM# # of LY302 | 100 mg AM# PM# 3414 tablets taken | (Describe any missed or extra doses, vomiting |
| Day 15 Day 16 Day 17 | Date | AM PM AM PM AM PM AM PM AM AM AM | 50 mg AM# PM# # of LY302 | 100 mg AM# PM# 3414 tablets taken | (Describe any missed or extra doses, vomiting |
| Day 15 Day 16 Day 17 Day 18 Day 19 | Date | AM PM AM PM AM PM AM PM AM PM AM PM | 50 mg AM# PM# # of LY302 | 100 mg AM# PM# 3414 tablets taken | (Describe any missed or extra doses, vomiting |
| Day 15 Day 16 Day 17 Day 18 | Date | AM PM AM PM AM PM AM PM AM PM AM PM AM AM | 50 mg AM# PM# # of LY302 | 100 mg AM# PM# 3414 tablets taken | (Describe any missed or extra doses, vomiting |
| Day 15 Day 16 Day 17 Day 18 Day 19 Day 20 | Date | AM PM | 50 mg AM# PM# # of LY302 | 100 mg AM# PM# 3414 tablets taken | (Describe any missed or extra doses, vomiting |
| Day 15 Day 16 Day 17 Day 18 Day 19 | Date | AM PM AM PM AM PM AM PM AM PM AM PM AM AM | 50 mg AM# PM# # of LY302 | 100 mg AM# PM# 3414 tablets taken | (Describe any missed or extra doses, vomiting |

CHILDREN'S ONCOLOGY GROUP



This protocol is for research purposes only. See page 1 for usage policy. APEC1621D

| | Cycle # | : Start Da<br>End Dat | te: <br>te: | / <u> </u> | Dose Level: _ | mg/m²/dose |
|---|---|---|---|---|---|---|
| | | | | # of LY3023414 tablets<br>prescribed to take | | Comments (Describe any missed or extra doses, vomiting and/or bothersome effects.) |
| WEEK 4 | Date Time | Time | | 50 mg<br>AM#<br>PM# | 100 mg<br>AM#<br>PM# | |
| | | | | | 414 tablets taken | |
| | | | | 50 mg | 100 mg | |
| Day 22 | | | AM<br>PM | | | |
| Day 23 | | | AM | | | |
| • | | I | PM | | | |
| Day 24 | | | AM<br>PM | | | |
| <b>Day 25</b> | | | AM<br>PM | | | |
| | | | 4M | | | |
| <b>Day 26</b> | | | PM | | | |
| | | . A | AM | | | |
| <b>Day 27</b> | | I | PM | | | |
| Day 28 | | A | <b>AM</b> | | | |
| Day 26 | | I | PM | | | |
| | | will be used as a<br>this form below | | irce document | , the site personne | el who administered the study drug must |
| Signa | ature:(s | ite personnel wh | no ac | lministered the | e study drug) | Date: |



#### APPENDIX III-B: PATIENT DRUG INTERACTIONS HANDOUT AND WALLET CARD

Information for Patients, Their Caregivers and Non-Study Healthcare Team on Possible Interactions with Other Drugs and Herbal Supplements

Patient Diagnosis: Trial #:

Name:

<u>Study Doctor</u> <u>Study</u> LY3023414

Doctor: Phone #: Drug(s):

Please show this paper to all your healthcare providers (doctors, physician assistants, nurse practitioners, pharmacists), and tell them you are taking part in a clinical trial sponsored by the National Cancer Institute.

## These are the things that your healthcare providers need to know:

LY3023414 interacts with certain enzymes in your liver or other tissues like the gut, certain transport proteins that help move drugs in and out of cells and the heart's electrical activity.

#### **Explanation**

| СҮР | The enzymes in question are CYP 1A2 and 3A4. LY3023414 is broken down by CYP 1A2 and 3A4 and may be affected by other drugs that inhibit or induce these enzymes. |
|---|---|
| isoenzymes | LY3203414 weakly inhibits CYP 3A4, 2C9, 1A2 and may affect other drugs that are |
| | broken down by these enzymes. |
| | The transporter proteins in question are P-gp, BCRP, OATP1B1, OATP1B3, OCT1 |
| | and OCT2. LY3203414 is a substrate for P-gp, BCRP and OCT1 transport proteins and |
| Protein | other drugs that are potent inhibitors or inducers of these proteins may alter how |
| transporters | LY3203414 moves in and out of cells. LY3203414 may inhibit the ability of other |
| ti ansporters | drugs that require P-gp, BCRP, OATP1B1, OATP1B3, OCT1 or OCT2 to move in and |
| | out of cells. Avoid sensitive substrates of OATP1B1, OATP1B3, OCT1 or OCT2 |
| | transport proteins especially those with narrow therapeutic index. |
| Heart's | The heart's electrical activity may be affected by LY3023414. The study doctor may |
| electrical | be concerned about QTc prolongation and any other medicine that is associated with |
| activities | greater risk for having QTc prolongation. |

## These are the things that you need to know:

The study drug LY3023414, may interact with other drugs which can cause side effects. For this reason, it is very important to tell your doctors about all your medicines, including: (a) medicines you are taking before this clinical trial, (b) medicines you start or stop taking during this study, (c) medicines you buy without a prescription (over-the-counter remedy), (d) herbals or supplements (e.g. St. John's Wort). It is helpful to bring your medication bottles or an updated medication list with you.

Before you enroll onto the clinical trial, your study doctor will work with your regular health care providers to review any medicines and herbal supplements that are considered "strong inducers/inhibitors of CYP 1A2, 3A4, P-gp, BCRP or OCT1, are sensitive substrates of CYP 3A, 2C9 and 1A2, P-gp, BCRP, OATP1B1, OATP1B3, OCT1 or OCT2 or cause QTc prolongation."

- Please be very careful! Over-the-counter drugs (including herbal supplements) may contain ingredients that could interact with your study drug. Speak to your doctors or pharmacist to determine if there could be any side effects.
  - o Avoid ingesting grapefruit, grapefruit juice and Seville oranges while taking LY3023414.





This protocol is for research purposes only. See page 1 for usage policy. APEC1621D

- Make sure your doctor knows to avoid certain prescription medications.
- Your regular health care provider should check a frequently updated medical reference or call your study doctor before prescribing any new medicine or discontinuing any medicine.

Version JAN/2019

(Next page: Patient Drug Interaction Wallet Card)



# PATIENT DRUG INTERACTION WALLET CARD

| NIH NATIONAL CANCER INSTIT | NIH NATIONAL CANCER INSTIT | NIH NATIONAL CANCER INSTIT | NIH NATIONAL CANCER INSTI |
|---|---|---|---|
| EMERGENCY<br>NFORMATION | | DRUG INTE | ERACTIONS |
| Show this card to all of your healthcare providers. Keep it with you in case you go to the emergency room. | Tell your doctors before you start or stop any medicines. Check with your doctor or pharmacist if you need to use an over-the-counter medicine or herbal supplement! | Carry this card with you at all times LY3023414 interacts with interacts with certain enzymes in your or other tissues like the gut, certain transport proteins that help n drugs in and out of cells and the heart's electrical activity and mube used very carefully with other medicines. | |
| Patient Name: | Use caution and avoid the following drugs if possible: | Your healthcare providers should be | be aware of any medicines that are |
| Diagnosis: | Tonowing at ags it possible. | "strong inducers/inhibitors of CYF are sensitive substrates of CYP 3A | |
| Study Doctor: | Grapefruit, grapefruit juice, St.<br>John's Wort | OATP1B1, OATP1B3, OCT1 or C | |
| Study Doctor Phone #: | | | |
| NCI Trial #: | | Before prescribing new medic | cines, your health care provider |
| Study Drug(S): | | should check a <b>frequently-updat</b><br><b>drugs to avoid</b> or con | ed medical reference for a list of tact your study doctor. |
| | | | Version JAN/2019 |
| For more information: 1-800-4-<br>CANCER | For more information: 1-800-4-<br>CANCER | For more information: 1-800-4-<br>CANCER | For more information: 1-800-4-<br>CANCER |
| cancer gov clinicaltrials gov | cancer gov clinicaltrials gov | cancer gov clinicaltrials gov | cancer gov clinicaltrials gov |

Fold at dotted lines:





## APPENDIX IV: LY3023414 DOSING NOMOGRAM

Drug doses should be adjusted based on the BSA calculated from height and weight measured within 7 days prior to the beginning of each cycle.

# \*\*Please note the PM Dose on Cycle 1 Day 1 will be omitted for PK collection in patients participating on the dose-escalation portion of the study\*\*

LY3043414 Dose Assignment: 55 mg/m²/dose BID (Dose Level -1)

| BSA (m <sup>2</sup> ) | <b>Total Daily Dose</b> | AM Dose | PM Dose | <b>Dose Reduction For</b> | AM Dose | PM Dose |
|---|---|---|---|---|---|---|
| | (mg/day) | (mg) | (mg) | Toxicity (mg/day) | (mg) | (mg) |
| 0.75-1.09 | 100 | 50 | 50 | 50 | | 50 |
| 1.10-1.54 | 150 | 50 | 100 | 100 | 50 | 50 |
| ≥ 1.55 | 200 | 100 | 100 | 150 | 50 | 100 |

# LY3043414 Dose Assignment: 80 mg/m²/dose BID (Dose Level 1)

| BSA (m <sup>2</sup> ) | <b>Total Daily Dose</b> | AM Dose | PM Dose | <b>Dose Reduction For</b> | AM Dose | PM Dose |
|---|---|---|---|---|---|---|
| | (mg/day) | (mg) | (mg) | Toxicity (mg/day) | (mg) | (mg) |
| 0.52-0.74 | 100 | 50 | 50 | 50 | | 50 |
| 0.75-1.09 | 150 | 50 | 100 | 100 | 50 | 50 |
| 1.10-1.54 | 200 | 100 | 100 | 150 | 50 | 100 |
| ≥ 1.55 | 300 | 150 | 150 | 200 | 100 | 100 |

# LY3043414 Dose Assignment: 115 mg/m²/dose BID (Dose Level 2)

| BSA (m <sup>2</sup> ) | <b>Total Daily Dose</b> | AM Dose | PM Dose | <b>Dose Reduction For</b> | AM Dose | PM Dose |
|---|---|---|---|---|---|---|
| | (mg/day) | (mg) | (mg) | Toxicity (mg/day) | (mg) | (mg) |
| 0.37-0.51 | 100 | 50 | 50 | 50 | - | 50 |
| 0.52-0.74 | 150 | 50 | 100 | 100 | 50 | 50 |
| 0.75-1.09 | 200 | 100 | 100 | 150 | 50 | 100 |
| 1.10-1.54 | 300 | 150 | 150 | 200 | 100 | 100 |
| ≥ 1.55 | 400 | 200 | 200 | 300 | 150 | 150 |



# APPENDIX V: CORRELATIVE STUDIES GUIDE

| Completive | | Blood Volume | | |
|---|---|---|---|---|
| Correlative<br>Study | Section | Volume per Sample | Total<br>Cycle<br>1 | Tube Type |
| Pharmacokinetics | <u>8.3</u> | 2 mL | 18<br>mL* | K <sub>2</sub> EDTA lavender top |
| Total Blood Volume in<br>Cycle 1 | | | 18<br>mL | |

<sup>\*</sup> Collected from patients enrolled during the determination of the recommended phase 2 dose/ tolerable dose. All other patients will have two sample timepoints collected for a total of 4 mL during Cycle 1.

| Correlative | | Blood Volume | Blood Volume | |
|---|---|---|---|---|
| Study | Section | Volume per Sample | Total<br>Cycle 5<br>Day 1 | Tube Type |
| Circulating tumor<br>DNA (optional) | <u>8.4</u> | <ul> <li>For patients ≥ 10 kg collect 20 mLs (10 mL per tube x 2 tubes)</li> <li>For patients &gt; 2 kg but &lt; 10 kg collect 10 mL (one tube)</li> <li>For patients &lt; 2 kg research samples will not be collected</li> </ul> | 10mL | Streck Cell-Free DNA BCT tubes |
| Total Blood Volume in<br>Cycle 5 Day 1 | | | 10 mL | |

| Convolativo | | Blood Volur | ne | Tube Type |
|---|---|---|---|---|
| Correlative<br>Study | Section | Volume per Sample | Total 'Time of progression' or 'End of protocol therapy' | |
| Circulating<br>tumor DNA<br>(optional) | <u>8.4</u> | <ul> <li>For patients ≥ 10 kg collect 20 mLs (10 mL per tube x 2 tubes)</li> <li>For patients &gt; 2 kg but &lt; 10 kg collect 10 mL (one tube)</li> <li>For patients &lt; 2 kg research samples will not be collected</li> </ul> | 10mL* | Streck Cell-Free<br>DNA BCT tubes |
| Total Blood Volume in 'Time of progression or End of protocol therapy' | | | 10mL | |

<sup>\*</sup> Only collected from patients from whom the sample at Cycle 5 Day 1 is collected.



# APPENDIX VI: APEC1621D THERAPY DELIVERY MAP

| Therapy Delivery Map – Cycle 1 This Therapy Delivery Map (TDM) relates to Cycle 1. Each cycle lasts 28 days. | Patient COG ID number |
|---|---|
| | Accession number |

Criteria to start each cycle are listed in <u>Section 5.2</u>. Extensive treatment details are in <u>Section 5.1</u>.

| DRUG | ROUTE | DOSAGE | DAYS | IMPORTANT NOTES |
|---|---|---|---|---|
| LY3023414 | PO | Dose Level 2: 115 mg/m <sup>2</sup> /dose BID | 1-28 | LY3023414 should be taken without regards to |
| IND# | | (Recommended Phase 2 Dose) | | food with a glass of water at approximately the |
| 134661 | | | | same time each day. Patients should swallow the |
| | | Refer to dosing nomogram in | | tablets as a whole and should not chew or crush |
| | | Appendix IV. | | them. If a patient misses a dose of LY3023414, the |
| | | | | dose should be taken as soon as possible as long as |
| | | | | it is more than 6 hours before the next scheduled |
| | | | | dose. If it is less than 6 hours before the next dose, |
| | | | | then the dose should be skipped. If vomiting |
| | | | | occurs after taking LY3023414, the patient should |
| | | | | skip the dose and take the next dose as scheduled |

| Enter Cycle #: | D | ose Lev | vel:Ht | em Wt | kg BSA | m² |
|---|---|---|---|---|---|---|
| Date Due | Date Given | Day | LY3023414 | | Studies | |
| | | | mg AM | | | |
| | | | Enter calculated dose a | | | |
| | | | | dose administered below | | |
| | | 1 | mg AM | mg PM | a-1, n, o | |
| | | 2 | | mg PM | n | |
| | | 3 | mg AM | | f | |
| | | 4 | mg AM | | | |
| | | 5 | mg AM | | | |
| | | 6 | mg AM | mg PM | | |
| | | 7 | mg AM | mg PM | 1 21 1 | |
| | | 8 | mg AM | mg PM | a, b, f, h, i, m | |
| | | 9 | mg AM | mg PM | | |
| | | 10 | mg AM | mg PM | | |
| | | 11 | mg AM | mg PM | | |
| | | 12 | mg AM | mg PM | f | |
| | | 13 | mg AM | mg PM | | |
| | | 14 | mg AM | mg PM | 1 01 : | |
| | | 15 | mg AM | mg PM | a, b, f, h, i, m, n | |
| | | 16 | mg AM | mg PM | | |
| | | 17 | mg AM | mg PM | C | |
| | | 18 | mg AM | mg PM | f | |
| | | 19 | mg AM | mg PM | | |
| | | 20 | mg AM | mg PM | | |
| | | 21 | mg AM | mg PM | 1 (1 : | |
| | | 22 | mg AM | mg PM | a, b, f, h, i, m | |
| | | 23 | mg AM | mg PM | | |
| | | 24 | mg AM | mg PM | f | |
| | | | mg AM | mg PM | I | |
| | | 26<br>27 | mg AM | mg PM | | |
| | | 1 | mg AM | mg PM | a a f h i m | |
| | | 28/1 | mg AM _ | mg PM | a-c, f, h-j, m | |



See Section 6.0 for Dose Modifications for Toxicities and the COG Member website for Supportive Care Guidelines.

Required Observations in Cycle 1

All baseline studies must be performed prior to starting protocol therapy unless otherwise indicated below.

- a. History/Physical Exam (including VS)
- b. Neurological Exam
- c. Ht/Wt/BSA
- d. Performance Status
- e. Pregnancy Test. Women of childbearing potential require a negative pregnancy test prior to starting treatment; sexually active patients must use an acceptable method of birth control. Abstinence is an acceptable method of birth control.
- f. CBC/differential/platelets- If patients have Grade 4 neutropenia then CBCs should be checked at least every other day until recovery to Grade 3 or until meeting the criteria for dose limiting toxicity.
- g. Urinalysis
- h. Electrolytes including Ca++, PO4, Mg++
- i. Creatinine, ALT, bilirubin; Glucose
- j. Albumin; Total cholesterol, triglycerides
- k. Tumor Disease Evaluation
- 1. Bone Marrow Aspirate and/or biopsy- At baseline, only required for patients suspected of having bone marrow metastasis on the basis of history, symptoms, laboratory evaluation or other clinical data.
- m. Patient Diary- (see <u>Appendix III</u>) should be reviewed after completion of each treatment cycle and uploaded into RAVE. The patient diary should be collected weekly.
- n. Pharmacokinetics- see <u>Section 8.3</u> for details of PK studies.
- o. EKG

This listing only includes evaluations necessary to answer the primary and secondary aims. OBTAIN OTHER STUDIES AS REQUIRED FOR GOOD CLINICAL CARE.

| Comments |
|-------------------------------------------------|
| (Include any held doses, or dose modifications) |



# **All Subsequent Cycles**

Therapy Delivery Map – All Subsequent Cycles

This Therapy Delivery Map (TDM) relates to all subsequent cycles. Each cycle lasts 28 days. Treatment may continue in the absence of disease progression or unacceptable toxicity. Use a copy of this page once for each cycle (please note cycle number below).

Patient COG ID number

Accession number

Criteria to start each cycle are listed in <u>Section 5.2</u>. Extensive treatment details are in <u>Section 5.1</u>.

| DRUG | ROUTE | DOSAGE | DAYS | IMPORTANT NOTES |
|---|---|---|---|---|
| LY3023414 | PO | Dose Level 2: 115 mg/m <sup>2</sup> /dose BID | 1-28 | LY3023414 should be taken without regards to |
| IND # 134661 | | (Recommended Phase 2 Dose) | | food with a glass of water at approximately the |
| | | | | same time each day. Patients should swallow the |
| | | Refer to dosing nomogram in | | tablets as a whole and should not chew or crush |
| | | Appendix IV. | | them. If a patient misses a dose of LY3023414, |
| | | | | the dose should be taken as soon as possible as |
| | | | | long as it is more than 6 hours before the next |
| | | | | scheduled dose. If it is less than 6 hours before |
| | | | | the next dose, then the dose should be skipped. If |
| | | | | vomiting occurs after taking LY3023414, the |
| | | | | patient should skip the dose and take the next |
| | | | | dose as scheduled. |

| Enter Cycle # | : D | ose Le | vel:Ht | cm Wt_ | kg | BSA | m |
|---|---|---|---|---|---|---|---|
| Date Due | Date Given | Day | LY3023414 | | Studies | | |
| | | · | mg AM | mg PM | | | |
| | | | Enter calculated dose al | | | | |
| | | | dosing nomogram and a | ctual dose | | | |
| | | | administered below | | | | |
| | | 1 | mg AM | mg PM | a-f, | | |
| | | 2 | mg AM | mg PM | | | |
| | | 3 | mg AM | mg PM | | | |
| | | 4 | mg AM | mg PM | | | |
| | | 5 | mg AM | mg PM | | | |
| | | 6 | mg AM | mg PM | | | |
| | | 7 | mg AM | mg PM | | | |
| | | 8 | mg AM | mg PM | c | | |
| | | 9 | mg AM | mg PM | | | |
| | | 10 | mg AM | mg PM | | | |
| | | 11 | mg AM | mg PM | | | |
| | | 12 | mg AM | mg PM | | | |
| | | 13 | mg AM | mg PM | | | |
| | | 14 | mg AM | mg PM | | | |
| | | 15 | mg AM | mg PM | c | | |
| | | 16 | mg AM | mg PM | | | |
| | | 17 | mg AM | mg PM | | | |
| | | 18 | mg AM | mg PM | | | |
| | | 19 | mg AM | mg PM | | | |
| | | 20 | mg AM | mg PM | | | |
| | | 21 | mg AM | mg PM | | | |
| | | 22 | mg AM | mg PM | c | | |
| | | 23 | mg AM | mg PM | | | |
| | | 24 | mg AM | mg PM | | | |
| | | 25 | mg AM | mg PM | | | |
| | | 26 | mg AM | mg PM | | | |
| | | 27 | mg AM | mg PM | | | |
| | | 28/1 | mg AM | mg PM | a-f. i | | |

Version Date: 10/28/2022



# Required Observations in All Subsequent Cycles

- a. History/Physical Exam (including VS and neurological exam)
- b. Ht/Wt/BSA
- c. CBC/differential/platelets If patients develop Grade 4 neutropenia then CBCs should be checked every 3 to 4 days until recovery to Grade 3
- d. Electrolytes including Ca++, PO4, Mg++
- e. Creatinine, ALT, bilirubin; Glucose
- f. Albumin; Total cholesterol, triglycerides
- g. Tumor Disease Evaluation Every other cycle. Tumor Disease Evaluation should be obtained on the next consecutive cycle after initial documentation of either a PR or CR. Subsequent scans may restart 2 cycles after the confirmatory scan. If the institutional investigator determines that the patient has progressed based on clinical or laboratory evidence, he/she may opt not to confirm this finding radiographically
- h. Bone Marrow Aspirate and/or biopsy- Every other cycle. Should only be performed on patients with known bone marrow involvement at baseline.
- i. Patient Diary- (see <u>Appendix III</u>) should be reviewed after completion of each treatment cycle and uploaded into RAVE. The patient diary should be collected weekly.
- j. Circulating Tumor DNA (ctDNA-optional)- With consent, two samples will be collected on this protocol (Cycle 5 Day 1; and for patients receiving ≥ 5 cycles, at progression or end of protocol therapy) see Section 8.4 for details of the ctDNA studies.

This listing only includes evaluations necessary to answer the primary and secondary aims. OBTAIN OTHER STUDIES AS REQUIRED FOR GOOD CLINICAL CARE.

| Comments |
|-------------------------------------------------|
| (Include any held doses, or dose modifications) |

Version Date: 10/28/2022



# APPENDIX VII-A: EXAMPLES OF ACTIONABLE MUTATIONS OF INTEREST FOR APEC1621D COHORT A (TSC)

| NON-HOTSPOT | RULES | | |
|-------------|-------------|--------------|-----|
| Gene Name | Description | Variant Type | LOE |
| TSC1 | Include | Deleterious | 3 |
| TSC2 | Include | Deleterious | 3 |
| NF1 | Exclude | Deleterious | |
| NF2 | Exclude | Deleterious | |

| EXCLUSION | VARIANTS | | |
|-----------|------------|---------|--------|
| Hotspots | | | |
| | | Variant | |
| Gene Name | Variant ID | Туре | aMOI |
| NRAS | COSM586 | SNV | p.Q61H |
| NRAS | COSM585 | SNV | p.Q61H |
| NRAS | COSM583 | SNV | p.Q61L |
| NRAS | COSM582 | SNV | p.Q61P |
| NRAS | COSM584 | SNV | p.Q61R |
| NRAS | COSM30646 | MNV | p.Q61L |
| NRAS | COSM33693 | MNV | p.Q61R |
| NRAS | COSM580 | SNV | p.Q61K |
| NRAS | COSM581 | SNV | p.Q61E |
| NRAS | COSM53223 | MNV | p.Q61K |
| NRAS | COSM12725 | MNV | p.Q61L |
| NRAS | COSM579 | MNV | p.Q61R |
| NRAS | COSM12730 | MNV | p.Q61K |
| NRAS | COSM574 | SNV | p.G13V |
| NRAS | COSM573 | SNV | p.G13D |
| NRAS | COSM575 | SNV | p.G13A |
| NRAS | COSM572 | MNV | p.G13V |
| NRAS | COSM569 | SNV | p.G13R |
| NRAS | COSM570 | SNV | p.G13C |
| NRAS | COSM571 | SNV | p.G13S |
| NRAS | COSM564 | SNV | p.G12D |
| NRAS | COSM565 | SNV | p.G12A |
| NRAS | COSM566 | SNV | p.G12V |
| NRAS | COSM561 | SNV | p.G12R |
| NRAS | COSM563 | SNV | p.G12S |



| NRAS | COSM562 | SNV | p.G12C |
|------|-------------|-----|----------|
| HRAS | COSM503 | SNV | p.Q61H |
| HRAS | COSM502 | SNV | p.Q61H |
| HRAS | COSM499 | SNV | p.Q61R |
| HRAS | COSM500 | SNV | p.Q61P |
| HRAS | COSM498 | SNV | p.Q61L |
| HRAS | COSM33695 | MNV | p.Q61R |
| HRAS | COSM501 | MNV | p.Q61R |
| HRAS | COSM497 | SNV | p.Q61E |
| HRAS | COSM496 | SNV | p.Q61K |
| HRAS | COSM52978 | MNV | p.Q61L |
| HRAS | COSM490 | SNV | p.G13D |
| HRAS | COSM489 | SNV | p.G13V |
| HRAS | COSM488 | SNV | p.G13C |
| HRAS | COSM487 | SNV | p.G13S |
| HRAS | COSM486 | SNV | p.G13R |
| HRAS | COSM483 | SNV | p.G12V |
| HRAS | COSM484 | SNV | p.G12D |
| HRAS | COSM485 | SNV | p.G12A |
| HRAS | COSM482 | SNV | p.G12R |
| HRAS | COSM481 | SNV | p.G12C |
| HRAS | COSM480 | SNV | p.G12S |
| KRAS | COSM19900 | MNV | p.A146V |
| KRAS | COSM19404 | SNV | p. A146T |
| KRAS | COSM19940 | MNV | p.K117N |
| KRAS | COSM28519 | MNV | p.K117N |
| KRAS | COSM554 | SNV | p.Q61H |
| KRAS | COSM555 | SNV | p.Q61H |
| KRAS | COSM553 | SNV | p.Q61L |
| KRAS | COSM552 | SNV | p.Q61R |
| KRAS | COSM551 | SNV | p.Q61P |
| KRAS | COSM1168052 | MNV | p.Q61R |
| KRAS | COSM550 | SNV | p.Q61E |
| KRAS | COSM549 | SNV | p.Q61K |
| KRAS | COSM87298 | MNV | p.Q61K |
| KRAS | COSM539 | SNV | p.G15D |
| KRAS | COSM538 | SNV | p.G15S |
| KRAS | COSM87280 | SNV | p.G13E |
| KRAS | COSM30567 | SNV | p.G13E |
| KRAS | COSM533 | SNV | p.G13A |



| KRAS | COSM534 | SNV | p.G13V |
|------|-------------|-----|---------|
| KRAS | COSM532 | SNV | p.G13D |
| KRAS | COSM531 | MNV | p.G13D |
| KRAS | COSM530 | MNV | p.G13V |
| KRAS | COSM12721 | MNV | p.G13V |
| KRAS | COSM528 | SNV | p.G13S |
| KRAS | COSM527 | SNV | p.G13C |
| KRAS | COSM529 | SNV | p.G13R |
| KRAS | COSM13643 | SNV | p.G12N |
| KRAS | COSM512 | SNV | p.G12F |
| KRAS | COSM514 | SNV | p.G12L |
| KRAS | COSM87281 | MNV | p.G13C |
| KRAS | COSM520 | SNV | p.G12V |
| KRAS | COSM521 | SNV | p.G12D |
| KRAS | COSM522 | SNV | p.G12A |
| KRAS | COSM14209 | MNV | p.G12D |
| KRAS | COSM515 | MNV | p.G12V |
| KRAS | COSM518 | SNV | p.G12R |
| KRAS | COSM517 | SNV | p.G12S |
| KRAS | COSM516 | SNV | p.G12C |
| KRAS | COSM513 | MNV | p.G12C |
| KRAS | COSM5413585 | MNV | p.G12A |
| KRAS | COSM1716372 | MNV | p.G12L |
| KRAS | COSM249888 | MNV | p.G12R |
| KRAS | COSM4387522 | MNV | p.G12V |
| KRAS | COSM4745557 | MNV | p.G13R |
| ARAF | COSM5044705 | SNV | p.S214C |
| ARAF | COSM1742787 | SNV | p.S214A |
| ARAF | COSM612884 | SNV | p.S214F |
| BRAF | COSM1132 | SNV | p.K601N |
| BRAF | COSM6265 | SNV | p.K601N |
| BRAF | COSM308550 | MNV | p.V600D |
| BRAF | COSM477 | MNV | p.V600D |
| BRAF | COSM475 | MNV | p.V600E |
| BRAF | COSM1127 | MNV | p.V600R |
| BRAF | COSM1583011 | MNV | p.V600R |
| BRAF | COSM473 | MNV | p.V600K |
| BRAF | COSM474 | MNV | p.V600R |
| BRAF | COSM6137 | SNV | p.V600G |
| BRAF | COSM18443 | SNV | p.V600A |



| BRAF | COSM249889 | MNV | p.V600Q |
|------|--------------|-----|-----------------|
| BRAF | COSM476 | SNV | p.V600E |
| BRAF | COSM1130 | SNV | p.V600M |
| BRAF | COSM219798 | SNV | p.V600L |
| BRAF | COSM33808 | SNV | p.V600L |
| BRAF | COSM1133 | DEL | p.V600_K601>E |
| BRAF | PM_COSM30730 | INS | p.T599_V600insT |
| BRAF | PM_COSM26625 | INS | p.A598_T599insV |
| BRAF | COSM457 | SNV | p.G469R |
| BRAF | COSM455 | SNV | p.G469R |
| BRAF | COSM1112 | SNV | p.G466R |
| BRAF | COSM478 | SNV | p.K601E |
| BRAF | COSM472 | SNV | p.T599I |
| BRAF | COSM21549 | SNV | p.A598V |
| BRAF | COSM1126 | MNV | p.L597S |
| BRAF | COSM1125 | SNV | p.L597Q |
| BRAF | COSM471 | SNV | p.L597R |
| BRAF | COSM470 | SNV | p.L597V |
| BRAF | COSM469 | SNV | p.G596R |
| BRAF | COSM53198 | SNV | p.F595L |
| BRAF | COSM468 | SNV | p.F595L |
| BRAF | COSM21612 | SNV | p.F595L |
| BRAF | COSM466 | SNV | p.D594V |
| BRAF | COSM467 | SNV | p.D594G |
| BRAF | COSM211600 | MNV | p.D594N |
| BRAF | COSM1583010 | SNV | p.D594A |
| BRAF | COSM27639 | SNV | p.D594N |
| BRAF | COSM463 | SNV | p.E586K |
| BRAF | COSM462 | SNV | p.N581S |
| BRAF | COSM1133046 | SNV | p.Y472C |
| BRAF | COSM459 | SNV | p.G469V |
| BRAF | COSM460 | SNV | p.G469A |
| BRAF | COSM461 | SNV | p.G469E |
| BRAF | COSM451 | SNV | p.G466V |
| BRAF | COSM453 | SNV | p.G466E |
| BRAF | COSM452 | SNV | p.G466A |
| BRAF | COSM253328 | SNV | p.G466R |
| BRAF | COSM449 | SNV | p.G464E |
| BRAF | COSM450 | SNV | p.G464V |
| BRAF | COSM1448615 | SNV | p.G464R |



| 1 | | | |
|--------|----------------|-----|------------------------|
| BRAF | COSM1111 | SNV | p.G464R |
| BRAF | COSM448 | SNV | p.I463S |
| BRAF | COSM447 | SNV | p.R462I |
| MAP2K1 | PM_E1 | DEL | p.F53_Q58delFLTQKQaddL |
| MAP2K1 | PM_E2 | DEL | p.Q56_V60delQKQKV |
| MAP2K1 | COSM1235481 | SNV | p.Q56P |
| MAP2K1 | COSM4756761 | SNV | p.K57T |
| MAP2K1 | COSM1235478 | SNV | p.K57N |
| MAP2K1 | COSM5520914 | SNV | p.K57N |
| MAP2K1 | PM_COSM4166150 | DEL | p.K57_G61del |
| MAP2K1 | PM_COSM5031101 | DEL | p.Q58_E62delQKVGE |
| MAP2K1 | PM_COSM5031100 | DEL | p.Q58_E62delQKVGE |
| MAP2K1 | PM_COSM1235479 | SNV | p.D67N |
| MAP2K1 | COSM1678546 | SNV | p.D67N |
| MAP2K1 | PM_COSM404998 | DEL | p.E102_l103delEl |
| MAP2K1 | PM_COSM4166152 | DEL | p.E102_I103del |
| MAP2K1 | PM_COSM4166153 | DEL | p.E102_I103del |
| MAP2K1 | PM_COSM5730253 | DEL | p.I103_K104delIK |
| MAP2K1 | PM_COSM5702512 | DEL | p.I103_K104del |
| MAP2K1 | PM_E3 | SNV | p.E120Q |
| MAP2K1 | COSM555601 | SNV | p.C121S |
| MAP2K1 | COSM1315829 | SNV | p.C121S |
| MAP2K1 | PM_E4 | SNV | p.S123T |
| MAP2K1 | COSM1374186 | SNV | p.G128D |
| MAP2K1 | COSM232755 | SNV | p.E203K |
| GNA11 | COSM52969 | SNV | p.Q209L |
| GNA11 | COSM52970 | SNV | p.Q209P |
| GNAQ | COSM28757 | SNV | p.Q209L |
| GNAQ | COSM28758 | SNV | p.Q209P |
| GNAQ | COSM28760 | SNV | p.Q209R |
| GNAQ | COSM52975 | SNV | p.R183Q |

# **Fusions**

| | | Variant | |
|-----------|----------------------------|---------|------------------|
| Gene Name | Variant ID | Type | aMOI |
| BRAF | AGAP3-BRAF.A10B11 | Fusion | BRAF Gene Fusion |
| BRAF | AGAP3-BRAF.A9B9 | Fusion | BRAF Gene Fusion |
| BRAF | AGK-BRAF.A2B8 | Fusion | BRAF Gene Fusion |
| BRAF | AGTRAP-BRAF.A5B8.COSF828.1 | Fusion | BRAF Gene Fusion |
| BRAF | AKAP9-BRAF.A21B10 | Fusion | BRAF Gene Fusion |



| BRAF | AKAP9-BRAF.A22B9 | Fusion | <b>BRAF Gene Fusion</b> |
|------|------------------------------|--------|-------------------------|
| BRAF | AKAP9-BRAF.A28B9 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | AKAP9-BRAF.A7B11 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | AKAP9-BRAF.A8B9.COSF1013.1 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | AP3B1-BRAF.A22B9 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | ARMC10-BRAF.A4B11 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | ATG7-BRAF.A18B9 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | BAIAP2L1-BRAF.B12B9 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | BBS9-BRAF.B19B4 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | BCL2L11-BRAF.B3B10 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | BRAF-AP3B1.B8A23 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | BRAF-BRAF.B1B11 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | BRAF-BRAF.B1B9 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | BRAF-BRAF.B3B11 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | BRAF-BRAF.B3B9 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | BRAF-CIITA.B9C6 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | BRAF-MACF1.B8M15 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | BRAF-MRPS33.B1M2 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | BRAF-SLC26A4.B3S7 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | BRAF-SUGCT.B1S13 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | BTF3L4-BRAF.B3B11 | Fusion | <b>BRAF</b> Gene Fusion |
| BRAF | C7orf73-BRAF.C2B9 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | CCDC6-BRAF.C1B9 | Fusion | <b>BRAF</b> Gene Fusion |
| BRAF | CCDC91-BRAF.C11B9 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | CCNY-BRAF.C1B10 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | CDC27-BRAF.C16B9.1 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | CEP89-BRAF.C16B9 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | CLCN6-BRAF.C2B11.COSF1440 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | CLIP2-BRAF.C6B11 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | CUL1-BRAF.C7B9 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | CUX1-BRAF.C10B9 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | DYNC1I2-BRAF.D7B10 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | EML4-BRAF.E6B10 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | EPS15-BRAF.E22B10 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | ERC1-BRAF.E12B10 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | ERC1-BRAF.E17B8 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | FAM114A2-BRAF.F9B11 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | FAM131B-BRAF.F1B10.COSF1191 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | FAM131B-BRAF.F2B9.COSF1189.1 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | FAM131B-BRAF.F3B9.COSF1193 | Fusion | <b>BRAF Gene Fusion</b> |



| BRAF | FCHSD1-BRAF.F13B9.COSF403 | Fusion | <b>BRAF Gene Fusion</b> |
|------|---------------------------------|--------|-------------------------|
| BRAF | FXR1-BRAF.F13B10 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | GATM-BRAF.G2B11 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | GHR-BRAF.G1B10 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | GNAI1-BRAF.G1B10.COSF1442 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | GTF2I-BRAF.G4B10 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | HERPUD1-BRAF.H4B7 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | KCTD7-BRAF.K3B8 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | KCTD7-BRAF.K4B8 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | KDM7A-BRAF.K11B11 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | KIAA1549-BRAF.K12B11 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | KIAA1549-BRAF.K12B9.COSF1474 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | KIAA1549-BRAF.K13B9 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | KIAA1549-BRAF.K14B11.COSF1226 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | KIAA1549-BRAF.K14B9.COSF483 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | KIAA1549-BRAF.K15B10.COSF1283.1 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | KIAA1549-BRAF.K15B11.COSF485.1 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | KIAA1549-BRAF.K15B9.COSF481.1 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | KIAA1549-BRAF.K16B10 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | KIAA1549-BRAF.K17B10.COSF509 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | KIAA1549-BRAF.K18B9.COSF511 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | KIAA1549-BRAF.K9B9 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | KLHL7-BRAF.K5B9 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | LSM12-BRAF.L3B9 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | LSM14A-BRAF.L9B9 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | MACF1-BRAF.M60B9 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | MAD1L1-BRAF.M16B9 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | MAD1L1-BRAF.M17B10 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | MKRN1-BRAF.M4B11.COSF1444 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | MKRN1-BRAF.M4B9 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | MYRIP-BRAF.M16B9 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | MZT1-BRAF.M2B11 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | NUB1-BRAF.N3B9 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | NUDCD3-BRAF.N4B9 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | NUP214-BRAF.N21B10 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | PAPSS1-BRAF.P5B9.1 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | PLIN3-BRAF.P1B9 | Fusion | BRAF Gene Fusion |
| BRAF | RAD18-BRAF.R7B10 | Fusion | BRAF Gene Fusion |
| BRAF | RBMS3-BRAF.R11B11 | Fusion | BRAF Gene Fusion |
| BRAF | RNF11-BRAF.R1B11 | Fusion | BRAF Gene Fusion |



| i contract of the contract of | | | |
|---|---|---|---|
| BRAF | RNF130-BRAF.R3B9.COSF1483 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | RP2-BRAF.R3B10 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | SLC12A7-BRAF.S17B11 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | SLC45A3-BRAF.S1B8.COSF871 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | SND1-BRAF.S10B11 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | SND1-BRAF.S10B9 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | SND1-BRAF.S11B11 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | SND1-BRAF.S14B11 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | SND1-BRAF.S14B9 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | SND1-BRAF.S16B9.1 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | SND1-BRAF.S18B10 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | SND1-BRAF.S9B2 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | SND1-BRAF.S9B9 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | SOX6-BRAF.S5B9 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | SOX6-BRAF.S6B9 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | STRN3-BRAF.S3B10 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | TANK-BRAF.T4B9 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | TAX1BP1-BRAF.T8B11.1 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | TMEM178B-BRAF.T2B9 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | TMPRSS2-BRAF.T3B11 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | TRIM24-BRAF.T10B9 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | TRIM24-BRAF.T11B2 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | TRIM24-BRAF.T3B10 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | TRIM24-BRAF.T3B11 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | TRIM24-BRAF.T5B8 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | TRIM24-BRAF.T9B9.1 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | TRIM4-BRAF.T6B10 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | UBN2-BRAF.U3B11 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | ZC3HAV1-BRAF.Z3B10 | Fusion | BRAF Gene Fusion |
| BRAF | ZC3HAV1-BRAF.Z7B11 | Fusion | BRAF Gene Fusion |
| BRAF | ZKSCAN5-BRAF.Z2B9 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | ZSCAN30-BRAF.Z3B10 | Fusion | BRAF Gene Fusion |

| INCLUSION | VARIANTS | | | |
|-----------|----------------|---------|-------------|-----|
| Hotspots | | | | |
| | | Variant | | |
| Gene Name | Variant ID | Type | aMOI | LOE |
| TSC1 | PM_MCH12 | SNV | p. Q527* | 3 |
| TSC1 | PM_COSM1636659 | DEL | p.E636fs*51 | 3 |



| TSC1 | PM_MCH11 | SNV | p. Q781* | 3 | ı |
|------|----------------|-------|-------------------|---|---|
| TSC1 | PM_D22 | SNV | F158S | 3 | ı |
| TSC1 | PM_D23 | SNV | F216S | 3 | ı |
| TSC1 | PM_D24 | SNV | G132D | 3 | ı |
| TSC1 | PM_D25 | SNV | G305R | 3 | ı |
| TSC1 | PM_D26 | SNV | G305W | 3 | ı |
| TSC1 | PM_D27 | SNV | 176N | 3 | ì |
| TSC1 | PM_D28 | SNV | K121R | 3 | ı |
| TSC1 | PM_D29 | SNV | L117P | 3 | ı |
| TSC1 | PM_D30 | SNV | L180P | 3 | ı |
| TSC1 | PM_D31 | SNV | L191H | 3 | ı |
| TSC1 | PM_D32 | SNV | L191R | 3 | ı |
| TSC1 | PM_D33 | SNV | L50P | 2 | ı |
| TSC1 | COSM5013848 | SNV | L61P | 3 | ı |
| TSC1 | PM_D34 | SNV | L61R | 3 | ı |
| TSC1 | COSM277850 | SNV | L72P | 3 | ı |
| TSC1 | PM_D35 | SNV | L93R | 3 | ı |
| TSC1 | PM_D36 | SNV | M224R | 3 | ı |
| TSC1 | PM_D1 | DEL | p.128delV | 3 | ı |
| TSC1 | PM_D2 | INDEL | p.N198F199delinsI | 3 | ı |
| TSC1 | COSM1314592 | SNV | R190P | 3 | ı |
| TSC1 | PM_D37 | SNV | R204P | 3 | ı |
| TSC1 | PM_D38 | SNV | R246K | 3 | ı |
| TSC1 | PM_D39 | SNV | R246T | 3 | ı |
| TSC1 | PM_D3 | DEL | S201del | 3 | ı |
| TSC1 | PM_D40 | SNV | V133F | 3 | ı |
| TSC2 | PM_COSM4440414 | SNV | p. Q1178* | 3 | ì |
| TSC2 | PM_D41 | SNV | A1141T | 3 | ı |
| TSC2 | PM_D42 | SNV | A328P | 3 | ı |
| TSC2 | PM_D43 | SNV | A607E | 3 | ı |
| TSC2 | PM_D44 | SNV | A614D | 3 | ı |
| TSC2 | PM_D45 | SNV | A889P | 3 | ı |
| TSC2 | PM_D46 | SNV | A889V | 3 | ı |
| TSC2 | PM_D47 | SNV | C244R | 3 | ı |
| TSC2 | PM_D48 | SNV | C696Y | 3 | ì |
| TSC2 | PM_D49 | SNV | C804R | 3 | ì |
| TSC2 | PM_D50 | SNV | D1028N | 3 | ì |
| TSC2 | PM_D51 | SNV | D1535A/D1512A | 3 | ı |
| TSC2 | PM_D4 | DEL | E1552del/E1529del | 3 | ì |
| TSC2 | PM_D52 | SNV | E337K | 3 | |



| i | | | | |
|------|--------|-------|-----------------------|----|
| TSC2 | PM_D53 | SNV | E412V | 3 |
| TSC2 | PM_D54 | SNV | E75G | 3 |
| TSC2 | PM_D55 | SNV | F615S | 3 |
| TSC2 | PM_D56 | SNV | F897S | 3 |
| TSC2 | PM_D57 | SNV | G1204E | 3 |
| TSC2 | PM_D58 | SNV | G1567D/D1544D | 3 |
| TSC2 | PM_D59 | SNV | G1567V/G1544V | 3 |
| TSC2 | PM_D60 | SNV | G1579S/G1556S | 3 |
| TSC2 | PM_D61 | SNV | G1596V/G1573V | 3 |
| TSC2 | PM_D62 | SNV | G1642D/G1619D | 3 |
| TSC2 | PM_D5 | SNV | G305V | 3 |
| TSC2 | PM_D63 | SNV | H1620R/H1597R | 3 |
| TSC2 | PM_D64 | SNV | H1640Y/H1617Y | 3 |
| TSC2 | PM_D65 | SNV | H597Y | 3 |
| TSC2 | PM_D66 | SNV | L1061P | 3 |
| TSC2 | PM_D67 | SNV | L146R | 3 |
| TSC2 | PM_D68 | SNV | L1534H/L1511H | 3 |
| TSC2 | PM_D69 | SNV | L1548P/L1525P | 3 |
| TSC2 | PM_D70 | SNV | L1578P/L1555P | 3 |
| TSC2 | PM_D71 | SNV | L1584R/L1561R | 3 |
| TSC2 | PM_D6 | INDEL | L1750Afs25/L1727Afs25 | 3 |
| TSC2 | PM_D72 | SNV | L219P | 3 |
| TSC2 | PM_D73 | SNV | L340P | 3 |
| TSC2 | PM_D74 | SNV | L410R | 3 |
| TSC2 | PM_D75 | SNV | L448P | 3 |
| TSC2 | PM_D76 | SNV | L466P | 3 |
| TSC2 | PM_D77 | SNV | L493P | 3 |
| TSC2 | PM_D7 | SNV | L612P | 2 |
| TSC2 | PM_D78 | SNV | L693P | 3 |
| TSC2 | PM_D8 | SNV | L713R | 2 |
| TSC2 | PM_D79 | SNV | L737P | 2 |
| TSC2 | PM_D80 | SNV | L792R | 3 |
| TSC2 | PM_D81 | SNV | L826P | 3 |
| TSC2 | PM_D82 | SNV | L830R | 3 |
| TSC2 | PM_D83 | SNV | L844R | 3 |
| TSC2 | PM_D84 | SNV | L850P | 2 |
| TSC2 | PM_D9 | SNV | L916R | 3 |
| TSC2 | PM_D85 | SNV | M1I - no start codon | 3 |
| TSC2 | PM_D86 | SNV | M788R | 3 |
| TSC2 | PM_D87 | SNV | N1643H/N1620H | 3 |
| • | | | | Į. |



| TSC2 | PM_D88 | SNV | N1643I/N1620I | 3 |
|------|---------|-----|---------------------|---|
| TSC2 | PM_D89 | SNV | N1643K/N1620K | 3 |
| TSC2 | PM_D90 | SNV | N1643S/N1620S | 3 |
| TSC2 | PM_D10 | INS | p.105insALL | 3 |
| TSC2 | PM_D12 | DEL | p.1746del6/1723del6 | 3 |
| TSC2 | PM_D13 | DEL | p.275delN | 3 |
| TSC2 | PM_D14 | DEL | p.412del8 | 3 |
| TSC2 | PM_D16 | INS | p.597insH | 3 |
| TSC2 | PM_D17 | INS | p.609insS | 3 |
| TSC2 | PM_D18 | DEL | p.820dell | 3 |
| TSC2 | PM_D91 | SNV | P1202H | 3 |
| TSC2 | PM_D92 | SNV | P1497R/P1474R | 3 |
| TSC2 | PM_D93 | SNV | P1497S/P1474S | 3 |
| TSC2 | PM_D94 | SNV | P1497T/P1474T | 3 |
| TSC2 | PM_D95 | SNV | P1675L/P1652L | 2 |
| TSC2 | PM_D96 | SNV | P1709L/P1686L | 3 |
| TSC2 | PM_D97 | SNV | P419S | 3 |
| TSC2 | PM_D98 | SNV | Q1503P/Q1480P | 3 |
| TSC2 | PM_D99 | SNV | Q1554H/Q1531H | 3 |
| TSC2 | PM_D100 | SNV | Q1686P/Q1663P | 3 |
| TSC2 | PM_D101 | SNV | Q373P | 3 |
| TSC2 | PM_D102 | SNV | R1032P | 3 |
| TSC2 | PM_D103 | SNV | R1200W | 3 |
| TSC2 | PM_D104 | SNV | R1713H/R1690H | 3 |
| TSC2 | PM_D105 | SNV | R1743Q/R1720Q | 2 |
| TSC2 | PM_D106 | SNV | R1743W/R1720W | 2 |
| TSC2 | PM_D107 | SNV | R261P | 3 |
| TSC2 | PM_D108 | SNV | R462C | 3 |
| TSC2 | PM_D109 | SNV | R462H | 3 |
| TSC2 | PM_D19 | SNV | R462P | 3 |
| TSC2 | PM_D110 | SNV | R57H | 3 |
| TSC2 | PM_D111 | SNV | R611Q | 2 |
| TSC2 | PM_D112 | SNV | R611W | 2 |
| TSC2 | PM_D113 | SNV | R622W | 3 |
| TSC2 | PM_D114 | SNV | R628G | 3 |
| TSC2 | PM_D115 | SNV | R905G | 3 |
| TSC2 | PM_D116 | SNV | R905Q | 3 |
| TSC2 | PM_D117 | SNV | R905W | 2 |
| TSC2 | PM_D118 | SNV | R98W | 3 |
| TSC2 | PM_D119 | SNV | S1036P | 3 |


| 3 | S1653F/S1630F | SNV | PM_D120 | TSC2 |
|---|---|---|---|---|
| 3 | S1653P/S1630P | SNV | PM_D121 | TSC2 |
| 3 | T1068I | SNV | PM_D20 | TSC2 |
| 3 | T1203K | SNV | PM_D122 | TSC2 |
| 3 | T1623I/T1600I | SNV | PM_D123 | TSC2 |
| 3 | V1199G | SNV | PM_D124 | TSC2 |
| 3 | V1500G/V1477G | SNV | PM_D125 | TSC2 |
| 3 | V1646G/V1623G | SNV | PM_D126 | TSC2 |
| 3 | V1673D/V1650D | SNV | PM_D127 | TSC2 |
| 3 | V1673F/V1650F | SNV | PM_D128 | TSC2 |
| 3 | V241del | DEL | PM_D21 | TSC2 |
| 3 | V299G | SNV | PM_D129 | TSC2 |
| 3 | V334A | SNV | PM_D130 | TSC2 |
| 3 | V334G | SNV | PM_D131 | TSC2 |
| 3 | V560M | SNV | PM_D132 | TSC2 |
| 3 | V705E | SNV | PM_D133 | TSC2 |
| 3 | V705M | SNV | PM_D134 | TSC2 |
| 3 | V769E | SNV | PM_D135 | TSC2 |
| 3 | W1610G/W1587G | SNV | PM_D136 | TSC2 |
| 3 | Y1571N/Y1548N | SNV | PM_D137 | TSC2 |
| 3 | Y598C | SNV | PM_D138 | TSC2 |
| 3 | Y598H | SNV | PM_D139 | TSC2 |
| | 3<br>3 | S1653P/S1630P T1068I T1068I T1203K 3 T1623I/T1600I V1199G 3 V1500G/V1477G V1646G/V1623G V1673D/V1650D 3 V1673F/V1650F 3 V241del 3 V299G 3 V334A 3 V334G 3 V560M 3 V705E 3 V705M 3 V769E 3 W1610G/W1587G 3 Y1571N/Y1548N 3 Y598C 3 | SNV S1653P/S1630P 3 SNV T1068I 3 SNV T1203K 3 SNV T1623I/T1600I 3 SNV V1199G 3 SNV V1500G/V1477G 3 SNV V1646G/V1623G 3 SNV V1673D/V1650D 3 SNV V1673F/V1650F 3 DEL V241del 3 SNV V299G 3 SNV V334A 3 SNV V334G 3 SNV V705E 3 SNV V705M 3 SNV V769E 3 SNV V1571N/Y1548N 3 SNV Y1571N/Y1548N 3 SNV Y598C 3 | PM_D121 SNV S1653P/S1630P 3 PM_D20 SNV T1068I 3 PM_D122 SNV T1203K 3 PM_D123 SNV T1623I/T1600I 3 PM_D124 SNV V1199G 3 PM_D125 SNV V1500G/V1477G 3 PM_D126 SNV V1646G/V1623G 3 PM_D127 SNV V1673D/V1650D 3 PM_D128 SNV V1673F/V1650F 3 PM_D128 SNV V1673F/V1650F 3 PM_D129 SNV V299G 3 PM_D130 SNV V334A 3 PM_D130 SNV V334A 3 PM_D131 SNV V334G 3 PM_D132 SNV V560M 3 PM_D133 SNV V705E 3 PM_D134 SNV V705E 3 PM_D135 SNV V705M 3 PM_D135 SNV V769E 3 PM_D136 SNV W1610G/W1587G 3 PM_D137 SNV Y598C 3 |



# APPENDIX VII-B: EXAMPLES OF ACTIONABLE MUTATIONS OF INTEREST FOR APEC1621D COHORT B (PI3K)

| NON-HOTSPOT | RULES | | | |
|---|---|---|---|---|
| Gene Name | Description | Variant Type | LOE | Region: |
| PTEN | Include | Deleterious | 3 | |
| | | | | iSH2 domain aa 414- |
| PIK3R1 | Include | Deleterious | 3 | 622 |
| TSC1 | Exclude | Deleterious | (Included in cohort A) | |
| TSC2 | Exclude | Deleterious | (Included in cohort A) | |
| NF1 | Exclude | Deleterious | | |
| NF2 | Exclude | Deleterious | | |
| | | | | nSH2 domain aa 331- |
| PIK3R1 | Exclude | Deleterious | | 413 |

| EXCLUSION | VARIANTS | | |
|-----------|------------|---------|--------|
| Hotspots | | | |
| | | Variant | |
| Gene Name | Variant ID | Type | aMOI |
| NRAS | COSM586 | SNV | p.Q61H |
| NRAS | COSM585 | SNV | p.Q61H |
| NRAS | COSM583 | SNV | p.Q61L |
| NRAS | COSM582 | SNV | p.Q61P |
| NRAS | COSM584 | SNV | p.Q61R |
| NRAS | COSM30646 | MNV | p.Q61L |
| NRAS | COSM33693 | MNV | p.Q61R |
| NRAS | COSM580 | SNV | p.Q61K |
| NRAS | COSM581 | SNV | p.Q61E |
| NRAS | COSM53223 | MNV | p.Q61K |
| NRAS | COSM12725 | MNV | p.Q61L |
| NRAS | COSM579 | MNV | p.Q61R |
| NRAS | COSM12730 | MNV | p.Q61K |
| NRAS | COSM574 | SNV | p.G13V |
| NRAS | COSM573 | SNV | p.G13D |
| NRAS | COSM575 | SNV | p.G13A |
| NRAS | COSM572 | MNV | p.G13V |
| NRAS | COSM569 | SNV | p.G13R |
| NRAS | COSM570 | SNV | p.G13C |
| NRAS | COSM571 | SNV | p.G13S |
| NRAS | COSM564 | SNV | p.G12D |



| NRAS | COSM565 | SNV | p.G12A |
|------|-------------|-----|----------|
| NRAS | COSM566 | SNV | p.G12V |
| NRAS | COSM561 | SNV | p.G12R |
| NRAS | COSM563 | SNV | p.G12S |
| NRAS | COSM562 | SNV | p.G12C |
| HRAS | COSM503 | SNV | p.Q61H |
| HRAS | COSM502 | SNV | p.Q61H |
| HRAS | COSM499 | SNV | p.Q61R |
| HRAS | COSM500 | SNV | p.Q61P |
| HRAS | COSM498 | SNV | p.Q61L |
| HRAS | COSM33695 | MNV | p.Q61R |
| HRAS | COSM501 | MNV | p.Q61R |
| HRAS | COSM497 | SNV | p.Q61E |
| HRAS | COSM496 | SNV | p.Q61K |
| HRAS | COSM52978 | MNV | p.Q61L |
| HRAS | COSM490 | SNV | p.G13D |
| HRAS | COSM489 | SNV | p.G13V |
| HRAS | COSM488 | SNV | p.G13C |
| HRAS | COSM487 | SNV | p.G13S |
| HRAS | COSM486 | SNV | p.G13R |
| HRAS | COSM483 | SNV | p.G12V |
| HRAS | COSM484 | SNV | p.G12D |
| HRAS | COSM485 | SNV | p.G12A |
| HRAS | COSM482 | SNV | p.G12R |
| HRAS | COSM481 | SNV | p.G12C |
| HRAS | COSM480 | SNV | p.G12S |
| KRAS | COSM19900 | MNV | p.A146V |
| KRAS | COSM19404 | SNV | p. A146T |
| KRAS | COSM19940 | MNV | p.K117N |
| KRAS | COSM28519 | MNV | p.K117N |
| KRAS | COSM554 | SNV | p.Q61H |
| KRAS | COSM555 | SNV | p.Q61H |
| KRAS | COSM553 | SNV | p.Q61L |
| KRAS | COSM552 | SNV | p.Q61R |
| KRAS | COSM551 | SNV | p.Q61P |
| KRAS | COSM1168052 | MNV | p.Q61R |
| KRAS | COSM550 | SNV | p.Q61E |
| KRAS | COSM549 | SNV | p.Q61K |
| KRAS | COSM87298 | MNV | p.Q61K |
| KRAS | COSM539 | SNV | p.G15D |



| KRAS | COSM538 | SNV | p.G15S |
|------|-------------|-----|---------|
| KRAS | COSM87280 | SNV | p.G13E |
| KRAS | COSM30567 | SNV | p.G13E |
| KRAS | COSM533 | SNV | p.G13A |
| KRAS | COSM534 | SNV | p.G13V |
| KRAS | COSM532 | SNV | p.G13D |
| KRAS | COSM531 | MNV | p.G13D |
| KRAS | COSM530 | MNV | p.G13V |
| KRAS | COSM12721 | MNV | p.G13V |
| KRAS | COSM528 | SNV | p.G13S |
| KRAS | COSM527 | SNV | p.G13C |
| KRAS | COSM529 | SNV | p.G13R |
| KRAS | COSM13643 | SNV | p.G12N |
| KRAS | COSM512 | SNV | p.G12F |
| KRAS | COSM514 | SNV | p.G12L |
| KRAS | COSM87281 | MNV | p.G13C |
| KRAS | COSM520 | SNV | p.G12V |
| KRAS | COSM521 | SNV | p.G12D |
| KRAS | COSM522 | SNV | p.G12A |
| KRAS | COSM14209 | MNV | p.G12D |
| KRAS | COSM515 | MNV | p.G12V |
| KRAS | COSM518 | SNV | p.G12R |
| KRAS | COSM517 | SNV | p.G12S |
| KRAS | COSM516 | SNV | p.G12C |
| KRAS | COSM513 | MNV | p.G12C |
| KRAS | COSM5413585 | MNV | p.G12A |
| KRAS | COSM1716372 | MNV | p.G12L |
| KRAS | COSM249888 | MNV | p.G12R |
| KRAS | COSM4387522 | MNV | p.G12V |
| KRAS | COSM4745557 | MNV | p.G13R |
| ARAF | COSM5044705 | SNV | p.S214C |
| ARAF | COSM1742787 | SNV | p.S214A |
| ARAF | COSM612884 | SNV | p.S214F |
| BRAF | COSM1132 | SNV | p.K601N |
| BRAF | COSM6265 | SNV | p.K601N |
| BRAF | COSM308550 | MNV | p.V600D |
| BRAF | COSM477 | MNV | p.V600D |
| BRAF | COSM475 | MNV | p.V600E |
| BRAF | COSM1127 | MNV | p.V600R |
| BRAF | COSM1583011 | MNV | p.V600R |



| BRAF | COSM473 | MNV | p.V600K |
|------|--------------|-----|-----------------|
| BRAF | COSM474 | MNV | p.V600R |
| BRAF | COSM6137 | SNV | p.V600G |
| BRAF | COSM18443 | SNV | p.V600A |
| BRAF | COSM249889 | MNV | p.V600Q |
| BRAF | COSM476 | SNV | p.V600E |
| BRAF | COSM1130 | SNV | p.V600M |
| BRAF | COSM219798 | SNV | p.V600L |
| BRAF | COSM33808 | SNV | p.V600L |
| BRAF | COSM1133 | DEL | p.V600_K601>E |
| BRAF | PM_COSM30730 | INS | p.T599_V600insT |
| BRAF | PM_COSM26625 | INS | p.A598_T599insV |
| BRAF | COSM457 | SNV | p.G469R |
| BRAF | COSM455 | SNV | p.G469R |
| BRAF | COSM1112 | SNV | p.G466R |
| BRAF | COSM478 | SNV | p.K601E |
| BRAF | COSM472 | SNV | p.T599I |
| BRAF | COSM21549 | SNV | p.A598V |
| BRAF | COSM1126 | MNV | p.L597S |
| BRAF | COSM1125 | SNV | p.L597Q |
| BRAF | COSM471 | SNV | p.L597R |
| BRAF | COSM470 | SNV | p.L597V |
| BRAF | COSM469 | SNV | p.G596R |
| BRAF | COSM53198 | SNV | p.F595L |
| BRAF | COSM468 | SNV | p.F595L |
| BRAF | COSM21612 | SNV | p.F595L |
| BRAF | COSM466 | SNV | p.D594V |
| BRAF | COSM467 | SNV | p.D594G |
| BRAF | COSM211600 | MNV | p.D594N |
| BRAF | COSM1583010 | SNV | p.D594A |
| BRAF | COSM27639 | SNV | p.D594N |
| BRAF | COSM463 | SNV | p.E586K |
| BRAF | COSM462 | SNV | p.N581S |
| BRAF | COSM1133046 | SNV | p.Y472C |
| BRAF | COSM459 | SNV | p.G469V |
| BRAF | COSM460 | SNV | p.G469A |
| BRAF | COSM461 | SNV | p.G469E |
| BRAF | COSM451 | SNV | p.G466V |
| BRAF | COSM453 | SNV | p.G466E |
| BRAF | COSM452 | SNV | p.G466A |



| BRAF CUSMI25322 SNV p.G464E BRAF COSM450 SNV p.G464V BRAF COSM450 SNV p.G464V BRAF COSM1111 SNV p.G464R BRAF COSM448 SNV p.1663S BRAF COSM447 SNV p.R462I MAP2K1 PM_E1 DEL p.F53_OS8delFLTQKQaddL MAP2K1 PM_E2 DEL p.Q56_V60delQkQkV MAP2K1 COSM4756761 SNV p.K57T MAP2K1 COSM4756761 SNV p.K57N MAP2K1 COSM5235478 SNV p.K57N MAP2K1 COSM5520914 SNV p.K57N MAP2K1 PM_COSM166150 DEL p.K57_G61del MAP2K1 PM_COSM5031101 DEL p.C58_E62delQkVGE MAP2K1 PM_COSM5031100 DEL p.C58_E62delQkVGE MAP2K1 PM_COSM604998 DEL p.E102_1103del MAP2K1 PM_COSM466152 DEL p.E102_1103del | DDAE | COCN 4252220 | CNIV | ~ C4CCD |
|---|---|---|---|---|
| BRAF COSM450 SNV p.G464V BRAF COSM1448615 SNV p.G464R BRAF COSM1111 SNV p.G464R BRAF COSM448 SNV p.H63S BRAF COSM447 SNV p.R62I MAP2K1 PM_E1 DEL p.F53_Q58delFLTQKQaddL MAP2K1 PM_E2 DEL p.056_V60delQKQKV MAP2K1 COSM1235481 SNV p.K57T MAP2K1 COSM4756761 SNV p.K57T MAP2K1 COSM4756761 SNV p.K57N MAP2K1 COSM5320914 SNV p.K57N MAP2K1 PM_COSM4166150 DEL p.K57_G61del MAP2K1 PM_COSM5031101 DEL p.C58_E62delQKVGE MAP2K1 PM_COSM5031100 DEL p.C58_E62delQKVGE MAP2K1 PM_COSM4166152 SNV p.D67N MAP2K1 PM_COSM4166152 DEL p.E102_1103del MAP2K1 PM_COSM4166153 DEL p.E102_1103del | BRAF | COSM253328 | SNV | p.G466R |
| BRAF COSM1418615 SNV p.G464R BRAF COSM1111 SNV p.G464R BRAF COSM448 SNV p.1463S BRAF COSM447 SNV p.R462I MAPZK1 PM_E1 DEL p.F53_DS8delFLTQKQaddL MAPZK1 PM_E2 DEL p.Q56_V60delQkQkV MAPZK1 COSM1235481 SNV p.K57T MAPZK1 COSM1235478 SNV p.K57N MAPZK1 COSM1235478 SNV p.K57N MAPZK1 COSM5520914 SNV p.K57N MAPZK1 PM_COSM4166150 DEL p.K57_G61del MAPZK1 PM_COSM5031101 DEL p.C58_E62delQkVGE MAPZK1 PM_COSM5031100 DEL p.C58_E62delQkVGE MAPZK1 PM_COSM503125479 SNV p.D67N MAPZK1 PM_COSM4166152 DEL p.E102_I103delEl MAPZK1 PM_COSM4166153 DEL p.E102_I103del MAPZK1 PM_COSM5702512 DEL p.I103_K | | | | |
| BRAF COSM1111 SNV p.G464R BRAF COSM448 SNV p.1463S BRAF COSM447 SNV p.753_Q58delFLTQKQaddL MAP2K1 PM_E1 DEL p.Q56_V60delQkQkV MAP2K1 COSM1235481 SNV p.Q56P MAP2K1 COSM235481 SNV p.K57T MAP2K1 COSM4756761 SNV p.K57T MAP2K1 COSM52914 SNV p.K57N MAP2K1 COSM529914 SNV p.K57N MAP2K1 PM_COSM4166150 DEL p.K57_G61del MAP2K1 PM_COSM5031101 DEL p.Q58_E62delQkVGE MAP2K1 PM_COSM5031100 DEL p.Q58_E62delQkVGE MAP2K1 PM_COSM1235479 SNV p.D67N MAP2K1 PM_COSM404998 DEL p.E102_I103del MAP2K1 PM_COSM4166152 DEL p.E102_I103del MAP2K1 PM_COSM5702512 DEL p.I103_K104del MAP2K1 PM_COSM5702512 DEL | | | | |
| BRAF COSM448 SNV p.14635 BRAF COSM447 SNV p.R4621 MAP2K1 PM_E1 DEL p.753_QS8delFLTQKQaddL MAP2K1 PM_E2 DEL p.Q56_V60delQKQKV MAP2K1 COSM1235481 SNV p.Q56_F MAP2K1 COSM4756761 SNV p.K57T MAP2K1 COSM5235478 SNV p.K57N MAP2K1 COSM5520914 SNV p.K57N MAP2K1 PM_COSM4166150 DEL p.K57_G61del MAP2K1 PM_COSM5031101 DEL p.Q58_E62delQKVGE MAP2K1 PM_COSM5031100 DEL p.Q58_E62delQKVGE MAP2K1 PM_COSM5031100 DEL p.Q58_E62delQKVGE MAP2K1 PM_COSM1235479 SNV p.D67N MAP2K1 PM_COSM1678546 SNV p.D67N MAP2K1 PM_COSM4166152 DEL p.E102_I103del MAP2K1 PM_COSM570253 DEL p.E102_I103del MAP2K1 PM_E3 SNV <td< td=""><td></td><td></td><td></td><td>·</td></td<> | | | | · |
| BRAF COSM447 SNV p.R462I MAP2K1 PM_E1 DEL p.F53_Q58delFLTQKQaddL MAP2K1 PM_E2 DEL p.Q56_V60delQkQkV MAP2K1 COSM1235481 SNV p.Q56_P MAP2K1 COSM4756761 SNV p.K57T MAP2K1 COSM523478 SNV p.K57N MAP2K1 COSM5520914 SNV p.K57N MAP2K1 PM_COSM531101 DEL p.K57_G61del MAP2K1 PM_COSM5031101 DEL p.Q58_E62delQkVGE MAP2K1 PM_COSM5031100 DEL p.Q58_E62delQkVGE MAP2K1 PM_COSM5031100 DEL p.Q58_E62delQkVGE MAP2K1 PM_COSM5031300 DEL p.Q58_E62delQkVGE MAP2K1 PM_COSM1235479 SNV p.D67N MAP2K1 PM_COSM1235479 SNV p.D67N MAP2K1 PM_COSM404998 DEL p.E102_1103del MAP2K1 PM_COSM5730253 DEL p.E102_1103del MAP2K1 PM_COSM5702512 | | | | · |
| MAP2K1 PM_E1 DEL p.F53_Q58delFLTQKQaddL MAP2K1 PM_E2 DEL p.Q56_V60delQkQkV MAP2K1 COSM1235481 SNV p.Q56P MAP2K1 COSM4756761 SNV p.K57T MAP2K1 COSM523478 SNV p.K57N MAP2K1 COSM5520914 SNV p.K57N MAP2K1 PM_COSM4166150 DEL p.K57_G61del MAP2K1 PM_COSM5031101 DEL p.Q58_E62delQkVGE MAP2K1 PM_COSM5031100 DEL p.Q58_E62delQkVGE MAP2K1 PM_COSM1235479 SNV p.D67N MAP2K1 PM_COSM1678546 SNV p.D67N MAP2K1 PM_COSM404998 DEL p.E102_I103delEl MAP2K1 PM_COSM4166152 DEL p.E102_I103del MAP2K1 PM_COSM5730253 DEL p.I103_K104dellK MAP2K1 PM_COSM5750253 DEL p.I103_K104dellK MAP2K1 PM_E3 SNV p.C1215 MAP2K1 PM_E3 SNV | | | | · |
| MAP2K1 PM_E2 DEL p.Q56_V60delQKQkV MAP2K1 COSM1235481 SNV p.Q56P MAP2K1 COSM4756761 SNV p.K57T MAP2K1 COSM1235478 SNV p.K57N MAP2K1 COSM520914 SNV p.K57N MAP2K1 PM_COSM5031101 DEL p.K57_G61del MAP2K1 PM_COSM5031100 DEL p.C58_E62delQKVGE MAP2K1 PM_COSM1235479 SNV p.D67N MAP2K1 PM_COSM1678546 SNV p.D67N MAP2K1 PM_COSM404998 DEL p.E102_l103del MAP2K1 PM_COSM4166152 DEL p.E102_l103del MAP2K1 PM_COSM4166153 DEL p.E102_l103del MAP2K1 PM_COSM5730253 DEL p.1103_K104dell MAP2K1 PM_COSM5702512 DEL p.E120Q MAP2K1 PM_E3 SNV p.C1215 MAP2K1 COSM1315829 SNV p.C1215 MAP2K1 COSM13174186 SNV <td< td=""><td></td><td>COSM447</td><td></td><td>•</td></td<> | | COSM447 | | • |
| MAP2K1 COSM1335481 SNV p.Q56P MAP2K1 COSM4756761 SNV p.K57T MAP2K1 COSM1235478 SNV p.K57N MAP2K1 COSM520914 SNV p.K57N MAP2K1 PM_COSM4166150 DEL p.K57_661del MAP2K1 PM_COSM5031100 DEL p.Q58_E62delQkVGE MAP2K1 PM_COSM5031100 DEL p.Q58_E62delQkVGE MAP2K1 PM_COSM1235479 SNV p.D67N MAP2K1 PM_COSM1678546 SNV p.D67N MAP2K1 PM_COSM404998 DEL p.E102_I103del MAP2K1 PM_COSM4166152 DEL p.E102_I103del MAP2K1 PM_COSM4166153 DEL p.E102_I103del MAP2K1 PM_COSM5730253 DEL p.I103_K104dellK MAP2K1 PM_COSM5702512 DEL p.I103_K104del MAP2K1 PM_E3 SNV p.C1215 MAP2K1 COSM53755 SNV p.C1215 MAP2K1 PM_E4 SNV | | <del>-</del> | | · = |
| MAP2K1 COSM4756761 SNV p.K57T MAP2K1 COSM1235478 SNV p.K57N MAP2K1 COSM5520914 SNV p.K57N MAP2K1 PM_COSM5031101 DEL p.K57_G61del MAP2K1 PM_COSM5031101 DEL p.Q58_E62delQKVGE MAP2K1 PM_COSM5031100 DEL p.Q58_E62delQKVGE MAP2K1 PM_COSM1235479 SNV p.D67N MAP2K1 PM_COSM1235479 SNV p.D67N MAP2K1 PM_COSM404998 DEL p.E102_1103del MAP2K1 PM_COSM4166152 DEL p.E102_1103del MAP2K1 PM_COSM5730253 DEL p.I103_K104dellK MAP2K1 PM_COSM5702512 DEL p.I103_K104del MAP2K1 PM_E3 SNV p.C121S MAP2K1 PM_E3 SNV p.C121S MAP2K1 COSM555601 SNV p.C121S MAP2K1 COSM1315829 SNV p.C121S MAP2K1 COSM1374186 SNV <t< td=""><td>MAP2K1</td><td>PM_E2</td><td>DEL</td><td>p.Q56_V60delQKQKV</td></t<> | MAP2K1 | PM_E2 | DEL | p.Q56_V60delQKQKV |
| MAP2K1 COSM1235478 SNV p.K57N MAP2K1 COSM5520914 SNV p.K57N MAP2K1 PM_COSM4166150 DEL p.K57_G61del MAP2K1 PM_COSM5031101 DEL p.C58_E62delQkVGE MAP2K1 PM_COSM5031100 DEL p.Q58_E62delQkVGE MAP2K1 PM_COSM1235479 SNV p.D67N MAP2K1 PM_COSM1235479 SNV p.D67N MAP2K1 PM_COSM1235479 SNV p.D67N MAP2K1 PM_COSM404998 DEL p.E102_1103delEI MAP2K1 PM_COSM4166152 DEL p.E102_1103del MAP2K1 PM_COSM5730253 DEL p.I103_K104delIK MAP2K1 PM_COSM5702512 DEL p.I103_K104del MAP2K1 PM_E3 SNV p.C121S MAP2K1 PM_E3 SNV p.C121S MAP2K1 COSM555601 SNV p.C121S MAP2K1 COSM1315829 SNV p.C121S MAP2K1 COSM2375186 SNV | MAP2K1 | COSM1235481 | SNV | p.Q56P |
| MAP2K1 COSM5520914 SNV p.K57N MAP2K1 PM_COSM4166150 DEL p.K57_G61del MAP2K1 PM_COSM5031101 DEL p.Q58_E62delQkVGE MAP2K1 PM_COSM5031100 DEL p.Q58_E62delQkVGE MAP2K1 PM_COSM1235479 SNV p.D67N MAP2K1 PM_COSM1235479 SNV p.D67N MAP2K1 PM_COSM404998 DEL p.E102_l103delEl MAP2K1 PM_COSM404998 DEL p.E102_l103delEl MAP2K1 PM_COSM4166152 DEL p.E102_l103del MAP2K1 PM_COSM4166153 DEL p.E102_l103del MAP2K1 PM_COSM5730253 DEL p.I103_k104dell MAP2K1 PM_COSM5702512 DEL p.I103_k104dell MAP2K1 PM_E3 SNV p.E120Q MAP2K1 PM_E3 SNV p.C1215 MAP2K1 COSM5555601 SNV p.C1215 MAP2K1 PM_E4 SNV p.G128D MAP2K1 COSM1374186 <td< td=""><td>MAP2K1</td><td>COSM4756761</td><td>SNV</td><td>p.K57T</td></td<> | MAP2K1 | COSM4756761 | SNV | p.K57T |
| MAP2K1 PM_COSM4166150 DEL p.K57_G61del MAP2K1 PM_COSM5031101 DEL p.Q58_E62delQkVGE MAP2K1 PM_COSM5031100 DEL p.Q58_E62delQkVGE MAP2K1 PM_COSM1235479 SNV p.D67N MAP2K1 PM_COSM1235479 SNV p.D67N MAP2K1 PM_COSM404998 DEL p.E102_I103delEI MAP2K1 PM_COSM4066152 DEL p.E102_I103del MAP2K1 PM_COSM4166153 DEL p.E102_I103del MAP2K1 PM_COSM5730253 DEL p.I103_K104delIK MAP2K1 PM_COSM5702512 DEL p.I103_K104del MAP2K1 PM_E3 SNV p.E120Q MAP2K1 PM_E3 SNV p.C1215 MAP2K1 COSM555601 SNV p.C1215 MAP2K1 COSM1315829 SNV p.G128D MAP2K1 PM_E4 SNV p.G128D MAP2K1 COSM23755 SNV p.E203K GNA11 COSM23755 SNV | MAP2K1 | COSM1235478 | SNV | p.K57N |
| MAP2K1 PM_COSM5031101 DEL p.Q58_E62delQkVGE MAP2K1 PM_COSM5031100 DEL p.Q58_E62delQkVGE MAP2K1 PM_COSM1235479 SNV p.D67N MAP2K1 COSM1678546 SNV p.D67N MAP2K1 PM_COSM404998 DEL p.E102_l103delEl MAP2K1 PM_COSM4166152 DEL p.E102_l103del MAP2K1 PM_COSM4166153 DEL p.E102_l103del MAP2K1 PM_COSM5730253 DEL p.I103_K104dellK MAP2K1 PM_COSM5702512 DEL p.I103_K104del MAP2K1 PM_E3 SNV p.E120Q MAP2K1 PM_E3 SNV p.C121S MAP2K1 COSM1315829 SNV p.C121S MAP2K1 COSM1374186 SNV p.G128D MAP2K1 COSM1374186 SNV p.G128D MAP2K1 COSM232755 SNV p.Q209L GNA11 COSM52970 SNV p.Q209P GNAQ COSM28757 SNV p | MAP2K1 | COSM5520914 | SNV | p.K57N |
| MAP2K1 PM_COSM5031100 DEL p.Q58_E62delQKVGE MAP2K1 PM_COSM1235479 SNV p.D67N MAP2K1 COSM1678546 SNV p.D67N MAP2K1 PM_COSM404998 DEL p.E102_l103delEl MAP2K1 PM_COSM4166152 DEL p.E102_l103del MAP2K1 PM_COSM4166153 DEL p.E102_l103del MAP2K1 PM_COSM5730253 DEL p.I103_K104dellK MAP2K1 PM_COSM5702512 DEL p.I103_K104del MAP2K1 PM_E3 SNV p.E120Q MAP2K1 PM_E3 SNV p.C121S MAP2K1 COSM555601 SNV p.C121S MAP2K1 COSM1315829 SNV p.C121S MAP2K1 COSM137486 SNV p.G128D MAP2K1 COSM1374186 SNV p.E203K GNA11 COSM52975 SNV p.Q209L GNA11 COSM52975 SNV p.Q209P GNAQ COSM28758 SNV p.Q209P < | MAP2K1 | PM_COSM4166150 | DEL | p.K57_G61del |
| MAP2K1 PM_COSM1235479 SNV p.D67N MAP2K1 COSM1678546 SNV p.D67N MAP2K1 PM_COSM404998 DEL p.E102_I103del MAP2K1 PM_COSM4166152 DEL p.E102_I103del MAP2K1 PM_COSM5730253 DEL p.I103_K104dellK MAP2K1 PM_COSM57302512 DEL p.I103_K104del MAP2K1 PM_COSM5702512 DEL p.I103_K104del MAP2K1 PM_E3 SNV p.E120Q MAP2K1 COSM5555601 SNV p.C121S MAP2K1 COSM1315829 SNV p.C121S MAP2K1 COSM1315829 SNV p.G128D MAP2K1 PM_E4 SNV p.G128D MAP2K1 COSM1374186 SNV p.G128D MAP2K1 COSM232755 SNV p.Q209L GNA11 COSM52969 SNV p.Q209L GNAQ COSM28758 SNV p.Q209P GNAQ COSM28758 SNV p.Q209P | MAP2K1 | PM_COSM5031101 | DEL | p.Q58_E62delQKVGE |
| MAP2K1 COSM1678546 SNV p.D67N MAP2K1 PM_COSM404998 DEL p.E102_I103del MAP2K1 PM_COSM4166152 DEL p.E102_I103del MAP2K1 PM_COSM5730253 DEL p.I103_K104dellK MAP2K1 PM_COSM57302512 DEL p.I103_K104del MAP2K1 PM_COSM5702512 DEL p.I103_K104del MAP2K1 PM_E3 SNV p.E120Q MAP2K1 COSM555601 SNV p.C121S MAP2K1 COSM555601 SNV p.C121S MAP2K1 COSM1315829 SNV p.C121S MAP2K1 PM_E4 SNV p.G128D MAP2K1 COSM1374186 SNV p.G128D MAP2K1 COSM23755 SNV p.E203K GNA11 COSM52969 SNV p.Q209L GNA11 COSM52970 SNV p.Q209P GNAQ COSM28758 SNV p.Q209P GNAQ COSM28760 SNV p.Q209P | MAP2K1 | PM_COSM5031100 | DEL | p.Q58_E62delQKVGE |
| MAP2K1 PM_COSM404998 DEL p.E102_I103delEI MAP2K1 PM_COSM4166152 DEL p.E102_I103del MAP2K1 PM_COSM4166153 DEL p.E102_I103del MAP2K1 PM_COSM5730253 DEL p.I103_K104delIK MAP2K1 PM_COSM5702512 DEL p.I103_K104del MAP2K1 PM_E3 SNV p.E120Q MAP2K1 COSM555601 SNV p.C121S MAP2K1 COSM1315829 SNV p.C121S MAP2K1 COSM1374186 SNV p.G128D MAP2K1 COSM1374186 SNV p.G128D MAP2K1 COSM232755 SNV p.E203K GNA11 COSM52969 SNV p.Q209L GNA11 COSM52970 SNV p.Q209P GNAQ COSM28757 SNV p.Q209P GNAQ COSM28760 SNV p.Q209P GNAQ COSM52975 SNV p.R183Q TSC1 PM_MCH12 SNV p.Q527* | MAP2K1 | PM_COSM1235479 | SNV | p.D67N |
| MAP2K1 PM_COSM4166152 DEL p.E102_I103del MAP2K1 PM_COSM4166153 DEL p.E102_I103del MAP2K1 PM_COSM5730253 DEL p.I103_K104dellK MAP2K1 PM_COSM5702512 DEL p.I103_K104del MAP2K1 PM_E3 SNV p.E120Q MAP2K1 COSM555601 SNV p.C121S MAP2K1 COSM1315829 SNV p.C121S MAP2K1 COSM1374186 SNV p.G128D MAP2K1 COSM1374186 SNV p.E203K MAP2K1 COSM232755 SNV p.Q209L GNA11 COSM52969 SNV p.Q209L GNA11 COSM52970 SNV p.Q209P GNAQ COSM28757 SNV p.Q209P GNAQ COSM28758 SNV p.Q209P GNAQ COSM52975 SNV p.R183Q TSC1 PM_MCH12 SNV p.Q527* TSC1 PM_COSM1636659 DEL p.E636fs*51 T | MAP2K1 | COSM1678546 | SNV | p.D67N |
| MAP2K1 PM_COSM4166153 DEL p.E102_I103del MAP2K1 PM_COSM5730253 DEL p.I103_K104dellK MAP2K1 PM_COSM5702512 DEL p.I103_K104del MAP2K1 PM_E3 SNV p.E120Q MAP2K1 COSM555601 SNV p.C121S MAP2K1 COSM1315829 SNV p.C121S MAP2K1 PM_E4 SNV p.S123T MAP2K1 COSM1374186 SNV p.G128D MAP2K1 COSM1374186 SNV p.E203K GNA11 COSM52969 SNV p.Q209L GNA11 COSM52970 SNV p.Q209P GNAQ COSM28757 SNV p.Q209P GNAQ COSM28758 SNV p.Q209P GNAQ COSM28760 SNV p.Q209R GNAQ COSM52975 SNV p.R183Q TSC1 PM_MCH12 SNV p.E636fs*51 TSC1 PM_COSM1636659 DEL p.E636fs*51 TSC1 | MAP2K1 | PM_COSM404998 | DEL | p.E102_I103delEI |
| MAP2K1 PM_COSM5730253 DEL p.I103_K104dellK MAP2K1 PM_COSM5702512 DEL p.I103_K104dell MAP2K1 PM_E3 SNV p.E120Q MAP2K1 COSM555601 SNV p.C121S MAP2K1 COSM1315829 SNV p.C121S MAP2K1 PM_E4 SNV p.S123T MAP2K1 COSM1374186 SNV p.G128D MAP2K1 COSM232755 SNV p.E203K GNA11 COSM52969 SNV p.Q209L GNA11 COSM52970 SNV p.Q209P GNAQ COSM28757 SNV p.Q209P GNAQ COSM28758 SNV p.Q209P GNAQ COSM28760 SNV p.Q209R GNAQ COSM52975 SNV p.R183Q TSC1 PM_MCH12 SNV p. E636fs*51 TSC1 PM_COSM1636659 DEL p.E636fs*51 TSC1 PM_MCH11 SNV p. Q781* TSC1 PM_D22< | MAP2K1 | PM_COSM4166152 | DEL | p.E102_l103del |
| MAP2K1 PM_COSM5702512 DEL p.I103_K104del MAP2K1 PM_E3 SNV p.E120Q MAP2K1 COSM555601 SNV p.C121S MAP2K1 COSM1315829 SNV p.C121S MAP2K1 PM_E4 SNV p.S123T MAP2K1 COSM1374186 SNV p.G128D MAP2K1 COSM232755 SNV p.E203K GNA11 COSM52969 SNV p.Q209L GNA11 COSM52970 SNV p.Q209P GNAQ COSM28757 SNV p.Q209P GNAQ COSM28758 SNV p.Q209P GNAQ COSM28760 SNV p.Q209R GNAQ COSM52975 SNV p.R183Q TSC1 PM_MCH12 SNV p.Q527* TSC1 PM_COSM1636659 DEL p.E636fs*51 TSC1 PM_MCH11 SNV p.Q781* TSC1 PM_D22 SNV F158S | MAP2K1 | PM_COSM4166153 | DEL | p.E102_l103del |
| MAP2K1 PM_E3 SNV p.E120Q MAP2K1 COSM555601 SNV p.C121S MAP2K1 COSM1315829 SNV p.C121S MAP2K1 PM_E4 SNV p.S123T MAP2K1 COSM1374186 SNV p.G128D MAP2K1 COSM232755 SNV p.E203K GNA11 COSM52969 SNV p.Q209L GNA11 COSM52970 SNV p.Q209P GNAQ COSM28757 SNV p.Q209L GNAQ COSM28758 SNV p.Q209P GNAQ COSM28760 SNV p.Q209R GNAQ COSM52975 SNV p.R183Q TSC1 PM_MCH12 SNV p. Q527* TSC1 PM_COSM1636659 DEL p.E636fs*51 TSC1 PM_MCH11 SNV p. Q781* TSC1 PM_MCH11 SNV F158S | MAP2K1 | PM_COSM5730253 | DEL | p.I103_K104delIK |
| MAP2K1 COSM555601 SNV p.C121S MAP2K1 COSM1315829 SNV p.C121S MAP2K1 PM_E4 SNV p.S123T MAP2K1 COSM1374186 SNV p.G128D MAP2K1 COSM232755 SNV p.E203K GNA11 COSM52969 SNV p.Q209L GNA11 COSM52970 SNV p.Q209P GNAQ COSM28757 SNV p.Q209L GNAQ COSM28758 SNV p.Q209P GNAQ COSM28760 SNV p.Q209R GNAQ COSM52975 SNV p.R183Q TSC1 PM_MCH12 SNV p. Q527* TSC1 PM_COSM1636659 DEL p.E636fs*51 TSC1 PM_MCH11 SNV p. Q781* TSC1 PM_D22 SNV F158S | MAP2K1 | PM_COSM5702512 | DEL | p.I103_K104del |
| MAP2K1 COSM1315829 SNV p.C121S MAP2K1 PM_E4 SNV p.S123T MAP2K1 COSM1374186 SNV p.G128D MAP2K1 COSM232755 SNV p.E203K GNA11 COSM52969 SNV p.Q209L GNA11 COSM52970 SNV p.Q209P GNAQ COSM28757 SNV p.Q209L GNAQ COSM28758 SNV p.Q209P GNAQ COSM28760 SNV p.Q209R GNAQ COSM52975 SNV p.R183Q TSC1 PM_MCH12 SNV p. Q527* TSC1 PM_COSM1636659 DEL p.E636fs*51 TSC1 PM_MCH11 SNV p. Q781* TSC1 PM_D22 SNV F158S | MAP2K1 | PM_E3 | SNV | p.E120Q |
| MAP2K1 PM_E4 SNV p.S123T MAP2K1 COSM1374186 SNV p.G128D MAP2K1 COSM232755 SNV p.E203K GNA11 COSM52969 SNV p.Q209L GNA11 COSM52970 SNV p.Q209P GNAQ COSM28757 SNV p.Q209L GNAQ COSM28758 SNV p.Q209P GNAQ COSM28760 SNV p.Q209R GNAQ COSM52975 SNV p.R183Q TSC1 PM_MCH12 SNV p.Q527* TSC1 PM_COSM1636659 DEL p.E636fs*51 TSC1 PM_MCH11 SNV p.Q781* TSC1 PM_D22 SNV F158S | MAP2K1 | COSM555601 | SNV | p.C121S |
| MAP2K1 COSM1374186 SNV p.G128D MAP2K1 COSM232755 SNV p.E203K GNA11 COSM52969 SNV p.Q209L GNA11 COSM52970 SNV p.Q209P GNAQ COSM28757 SNV p.Q209L GNAQ COSM28758 SNV p.Q209P GNAQ COSM28760 SNV p.Q209R GNAQ COSM52975 SNV p.R183Q TSC1 PM_MCH12 SNV p.Q527* TSC1 PM_COSM1636659 DEL p.E636fs*51 TSC1 PM_MCH11 SNV p.Q781* TSC1 PM_D22 SNV F158S | MAP2K1 | COSM1315829 | SNV | p.C121S |
| MAP2K1 COSM232755 SNV p.E203K GNA11 COSM52969 SNV p.Q209L GNA11 COSM52970 SNV p.Q209P GNAQ COSM28757 SNV p.Q209L GNAQ COSM28758 SNV p.Q209P GNAQ COSM28760 SNV p.Q209R GNAQ COSM52975 SNV p.R183Q TSC1 PM_MCH12 SNV p.Q527* TSC1 PM_COSM1636659 DEL p.E636fs*51 TSC1 PM_MCH11 SNV p.Q781* TSC1 PM_D22 SNV F158S | MAP2K1 | PM_E4 | SNV | p.S123T |
| GNA11 COSM52969 SNV p.Q209L GNA11 COSM52970 SNV p.Q209P GNAQ COSM28757 SNV p.Q209L GNAQ COSM28758 SNV p.Q209P GNAQ COSM28760 SNV p.Q209R GNAQ COSM52975 SNV p.R183Q TSC1 PM_MCH12 SNV p. Q527* TSC1 PM_COSM1636659 DEL p.E636fs*51 TSC1 PM_MCH11 SNV p. Q781* TSC1 PM_D22 SNV F158S | MAP2K1 | COSM1374186 | SNV | p.G128D |
| GNA11 COSM52970 SNV p.Q209P GNAQ COSM28757 SNV p.Q209L GNAQ COSM28758 SNV p.Q209P GNAQ COSM28760 SNV p.Q209R GNAQ COSM52975 SNV p.R183Q TSC1 PM_MCH12 SNV p. Q527* TSC1 PM_COSM1636659 DEL p.E636fs*51 TSC1 PM_MCH11 SNV p. Q781* TSC1 PM_D22 SNV F158S | MAP2K1 | COSM232755 | SNV | p.E203K |
| GNAQ COSM28757 SNV p.Q209L GNAQ COSM28758 SNV p.Q209P GNAQ COSM28760 SNV p.Q209R GNAQ COSM52975 SNV p.R183Q TSC1 PM_MCH12 SNV p. Q527* TSC1 PM_COSM1636659 DEL p.E636fs*51 TSC1 PM_MCH11 SNV p. Q781* TSC1 PM_D22 SNV F158S | GNA11 | COSM52969 | SNV | p.Q209L |
| GNAQ COSM28758 SNV p.Q209P GNAQ COSM28760 SNV p.Q209R GNAQ COSM52975 SNV p.R183Q TSC1 PM_MCH12 SNV p. Q527* TSC1 PM_COSM1636659 DEL p.E636fs*51 TSC1 PM_MCH11 SNV p. Q781* TSC1 PM_D22 SNV F158S | GNA11 | COSM52970 | SNV | p.Q209P |
| GNAQ COSM28760 SNV p.Q209R GNAQ COSM52975 SNV p.R183Q TSC1 PM_MCH12 SNV p. Q527* TSC1 PM_COSM1636659 DEL p.E636fs*51 TSC1 PM_MCH11 SNV p. Q781* TSC1 PM_D22 SNV F158S | GNAQ | COSM28757 | SNV | p.Q209L |
| GNAQ COSM52975 SNV p.R183Q TSC1 PM_MCH12 SNV p. Q527* TSC1 PM_COSM1636659 DEL p.E636fs*51 TSC1 PM_MCH11 SNV p. Q781* TSC1 PM_D22 SNV F158S | GNAQ | COSM28758 | SNV | p.Q209P |
| TSC1 PM_MCH12 SNV p. Q527* TSC1 PM_COSM1636659 DEL p.E636fs*51 TSC1 PM_MCH11 SNV p. Q781* TSC1 PM_D22 SNV F158S | GNAQ | COSM28760 | SNV | p.Q209R |
| TSC1 PM_COSM1636659 DEL p.E636fs*51 TSC1 PM_MCH11 SNV p. Q781* TSC1 PM_D22 SNV F158S | GNAQ | COSM52975 | SNV | p.R183Q |
| TSC1 PM_MCH11 SNV p. Q781* TSC1 PM_D22 SNV F158S | TSC1 | PM_MCH12 | SNV | p. Q527* |
| TSC1 PM_D22 SNV F158S | TSC1 | PM_COSM1636659 | DEL | p.E636fs*51 |
| | TSC1 | PM_MCH11 | SNV | p. Q781* |
| | TSC1 | PM_D22 | SNV | F158S |
| | TSC1 | PM_D23 | SNV | F216S |



| TSC1 | PM_D24 | SNV | G132D |
|------|----------------|-------|-------------------|
| TSC1 | PM_D25 | SNV | G305R |
| TSC1 | PM_D26 | SNV | G305W |
| TSC1 | PM_D27 | SNV | 176N |
| TSC1 | PM_D28 | SNV | K121R |
| TSC1 | PM_D29 | SNV | L117P |
| TSC1 | PM_D30 | SNV | L180P |
| TSC1 | PM_D31 | SNV | L191H |
| TSC1 | PM_D32 | SNV | L191R |
| TSC1 | PM_D33 | SNV | L50P |
| TSC1 | COSM5013848 | SNV | L61P |
| TSC1 | PM_D34 | SNV | L61R |
| TSC1 | COSM277850 | SNV | L72P |
| TSC1 | PM_D35 | SNV | L93R |
| TSC1 | PM_D36 | SNV | M224R |
| TSC1 | PM_D1 | DEL | p.128delV |
| TSC1 | PM_D2 | INDEL | p.N198F199delinsI |
| TSC1 | COSM1314592 | SNV | R190P |
| TSC1 | PM_D37 | SNV | R204P |
| TSC1 | PM_D38 | SNV | R246K |
| TSC1 | PM_D39 | SNV | R246T |
| TSC1 | PM_D3 | DEL | S201del |
| TSC1 | PM_D40 | SNV | V133F |
| TSC2 | PM_COSM4440414 | SNV | p. Q1178* |
| TSC2 | PM_D41 | SNV | A1141T |
| TSC2 | PM_D42 | SNV | A328P |
| TSC2 | PM_D43 | SNV | A607E |
| TSC2 | PM_D44 | SNV | A614D |
| TSC2 | PM_D45 | SNV | A889P |
| TSC2 | PM_D46 | SNV | A889V |
| TSC2 | PM_D47 | SNV | C244R |
| TSC2 | PM_D48 | SNV | C696Y |
| TSC2 | PM_D49 | SNV | C804R |
| TSC2 | PM_D50 | SNV | D1028N |
| TSC2 | PM_D51 | SNV | D1535A/D1512A |
| TSC2 | PM_D4 | DEL | E1552del/E1529del |
| TSC2 | PM_D52 | SNV | E337K |
| TSC2 | PM_D53 | SNV | E412V |
| TSC2 | PM_D54 | SNV | E75G |
| TSC2 | PM_D55 | SNV | F615S |



| TSC2 | PM_D56 | SNV | F897S |
|------|--------|-------|-----------------------|
| TSC2 | PM_D57 | SNV | G1204E |
| TSC2 | PM_D58 | SNV | G1567D/D1544D |
| TSC2 | PM_D59 | SNV | G1567V/G1544V |
| TSC2 | PM_D60 | SNV | G1579S/G1556S |
| TSC2 | PM_D61 | SNV | G1596V/G1573V |
| TSC2 | PM_D62 | SNV | G1642D/G1619D |
| TSC2 | PM_D5 | SNV | G305V |
| TSC2 | PM_D63 | SNV | H1620R/H1597R |
| TSC2 | PM_D64 | SNV | H1640Y/H1617Y |
| TSC2 | PM_D65 | SNV | H597Y |
| TSC2 | PM_D66 | SNV | L1061P |
| TSC2 | PM_D67 | SNV | L146R |
| TSC2 | PM_D68 | SNV | L1534H/L1511H |
| TSC2 | PM_D69 | SNV | L1548P/L1525P |
| TSC2 | PM_D70 | SNV | L1578P/L1555P |
| TSC2 | PM_D71 | SNV | L1584R/L1561R |
| TSC2 | PM_D6 | INDEL | L1750Afs25/L1727Afs25 |
| TSC2 | PM_D72 | SNV | L219P |
| TSC2 | PM_D73 | SNV | L340P |
| TSC2 | PM_D74 | SNV | L410R |
| TSC2 | PM_D75 | SNV | L448P |
| TSC2 | PM_D76 | SNV | L466P |
| TSC2 | PM_D77 | SNV | L493P |
| TSC2 | PM_D7 | SNV | L612P |
| TSC2 | PM_D78 | SNV | L693P |
| TSC2 | PM_D8 | SNV | L713R |
| TSC2 | PM_D79 | SNV | L737P |
| TSC2 | PM_D80 | SNV | L792R |
| TSC2 | PM_D81 | SNV | L826P |
| TSC2 | PM_D82 | SNV | L830R |
| TSC2 | PM_D83 | SNV | L844R |
| TSC2 | PM_D84 | SNV | L850P |
| TSC2 | PM_D9 | SNV | L916R |
| TSC2 | PM_D85 | SNV | M1I - no start codon |
| TSC2 | PM_D86 | SNV | M788R |
| TSC2 | PM_D87 | SNV | N1643H/N1620H |
| TSC2 | PM_D88 | SNV | N1643I/N1620I |
| TSC2 | PM_D89 | SNV | N1643K/N1620K |
| TSC2 | PM_D90 | SNV | N1643S/N1620S |



| TSC2 | PM_D10 | INS | p.105insALL |
|------|---------|-----|---------------------|
| TSC2 | PM_D12 | DEL | p.1746del6/1723del6 |
| TSC2 | PM_D13 | DEL | p.275delN |
| TSC2 | PM_D14 | DEL | p.412del8 |
| TSC2 | PM_D16 | INS | p.597 ins H |
| TSC2 | PM_D17 | INS | p.609insS |
| TSC2 | PM_D18 | DEL | p.820dell |
| TSC2 | PM_D91 | SNV | P1202H |
| TSC2 | PM_D92 | SNV | P1497R/P1474R |
| TSC2 | PM_D93 | SNV | P1497S/P1474S |
| TSC2 | PM_D94 | SNV | P1497T/P1474T |
| TSC2 | PM_D95 | SNV | P1675L/P1652L |
| TSC2 | PM_D96 | SNV | P1709L/P1686L |
| TSC2 | PM_D97 | SNV | P419S |
| TSC2 | PM_D98 | SNV | Q1503P/Q1480P |
| TSC2 | PM_D99 | SNV | Q1554H/Q1531H |
| TSC2 | PM_D100 | SNV | Q1686P/Q1663P |
| TSC2 | PM_D101 | SNV | Q373P |
| TSC2 | PM_D102 | SNV | R1032P |
| TSC2 | PM_D103 | SNV | R1200W |
| TSC2 | PM_D104 | SNV | R1713H/R1690H |
| TSC2 | PM_D105 | SNV | R1743Q/R1720Q |
| TSC2 | PM_D106 | SNV | R1743W/R1720W |
| TSC2 | PM_D107 | SNV | R261P |
| TSC2 | PM_D108 | SNV | R462C |
| TSC2 | PM_D109 | SNV | R462H |
| TSC2 | PM_D19 | SNV | R462P |
| TSC2 | PM_D110 | SNV | R57H |
| TSC2 | PM_D111 | SNV | R611Q |
| TSC2 | PM_D112 | SNV | R611W |
| TSC2 | PM_D113 | SNV | R622W |
| TSC2 | PM_D114 | SNV | R628G |
| TSC2 | PM_D115 | SNV | R905G |
| TSC2 | PM_D116 | SNV | R905Q |
| TSC2 | PM_D117 | SNV | R905W |
| TSC2 | PM_D118 | SNV | R98W |
| TSC2 | PM_D119 | SNV | S1036P |
| TSC2 | PM_D120 | SNV | S1653F/S1630F |



| TSC2 | PM_D121 | SNV | S1653P/S1630P |
|------|---------|-----|---------------|
| TSC2 | PM_D20 | SNV | T1068I |
| TSC2 | PM_D122 | SNV | T1203K |
| TSC2 | PM_D123 | SNV | T1623I/T1600I |
| TSC2 | PM_D124 | SNV | V1199G |
| TSC2 | PM_D125 | SNV | V1500G/V1477G |
| TSC2 | PM_D126 | SNV | V1646G/V1623G |
| TSC2 | PM_D127 | SNV | V1673D/V1650D |
| TSC2 | PM_D128 | SNV | V1673F/V1650F |
| TSC2 | PM_D21 | DEL | V241del |
| TSC2 | PM_D129 | SNV | V299G |
| TSC2 | PM_D130 | SNV | V334A |
| TSC2 | PM_D131 | SNV | V334G |
| TSC2 | PM_D132 | SNV | V560M |
| TSC2 | PM_D133 | SNV | V705E |
| TSC2 | PM_D134 | SNV | V705M |
| TSC2 | PM_D135 | SNV | V769E |
| TSC2 | PM_D136 | SNV | W1610G/W1587G |
| TSC2 | PM_D137 | SNV | Y1571N/Y1548N |
| TSC2 | PM_D138 | SNV | Y598C |
| TSC2 | PM_D139 | SNV | Y598H |

**Fusions** 

| 1 0310113 | | | |
|-----------|----------------------------|---------|------------------|
| | | Variant | |
| Gene Name | Variant ID | Type | aMOI |
| BRAF | AGAP3-BRAF.A10B11 | Fusion | BRAF Gene Fusion |
| BRAF | AGAP3-BRAF.A9B9 | Fusion | BRAF Gene Fusion |
| BRAF | AGK-BRAF.A2B8 | Fusion | BRAF Gene Fusion |
| BRAF | AGTRAP-BRAF.A5B8.COSF828.1 | Fusion | BRAF Gene Fusion |
| BRAF | AKAP9-BRAF.A21B10 | Fusion | BRAF Gene Fusion |
| BRAF | AKAP9-BRAF.A22B9 | Fusion | BRAF Gene Fusion |
| BRAF | AKAP9-BRAF.A28B9 | Fusion | BRAF Gene Fusion |
| BRAF | AKAP9-BRAF.A7B11 | Fusion | BRAF Gene Fusion |
| BRAF | AKAP9-BRAF.A8B9.COSF1013.1 | Fusion | BRAF Gene Fusion |
| BRAF | AP3B1-BRAF.A22B9 | Fusion | BRAF Gene Fusion |
| BRAF | ARMC10-BRAF.A4B11 | Fusion | BRAF Gene Fusion |
| BRAF | ATG7-BRAF.A18B9 | Fusion | BRAF Gene Fusion |
| BRAF | BAIAP2L1-BRAF.B12B9 | Fusion | BRAF Gene Fusion |
| BRAF | BBS9-BRAF.B19B4 | Fusion | BRAF Gene Fusion |
| BRAF | BCL2L11-BRAF.B3B10 | Fusion | BRAF Gene Fusion |



| BRAF | BRAF-AP3B1.B8A23 | Fusion | <b>BRAF Gene Fusion</b> |
|------|------------------------------|--------|-------------------------|
| BRAF | BRAF-BRAF.B1B11 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | BRAF-BRAF.B1B9 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | BRAF-BRAF.B3B11 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | BRAF-BRAF.B3B9 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | BRAF-CIITA.B9C6 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | BRAF-MACF1.B8M15 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | BRAF-MRPS33.B1M2 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | BRAF-SLC26A4.B3S7 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | BRAF-SUGCT.B1S13 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | BTF3L4-BRAF.B3B11 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | C7orf73-BRAF.C2B9 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | CCDC6-BRAF.C1B9 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | CCDC91-BRAF.C11B9 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | CCNY-BRAF.C1B10 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | CDC27-BRAF.C16B9.1 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | CEP89-BRAF.C16B9 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | CLCN6-BRAF.C2B11.COSF1440 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | CLIP2-BRAF.C6B11 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | CUL1-BRAF.C7B9 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | CUX1-BRAF.C10B9 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | DYNC1I2-BRAF.D7B10 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | EML4-BRAF.E6B10 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | EPS15-BRAF.E22B10 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | ERC1-BRAF.E12B10 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | ERC1-BRAF.E17B8 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | FAM114A2-BRAF.F9B11 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | FAM131B-BRAF.F1B10.COSF1191 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | FAM131B-BRAF.F2B9.COSF1189.1 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | FAM131B-BRAF.F3B9.COSF1193 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | FCHSD1-BRAF.F13B9.COSF403 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | FXR1-BRAF.F13B10 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | GATM-BRAF.G2B11 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | GHR-BRAF.G1B10 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | GNAI1-BRAF.G1B10.COSF1442 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | GTF2I-BRAF.G4B10 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | HERPUD1-BRAF.H4B7 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | KCTD7-BRAF.K3B8 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | KCTD7-BRAF.K4B8 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | KDM7A-BRAF.K11B11 | Fusion | <b>BRAF Gene Fusion</b> |



| 1 | | | |
|------|---------------------------------|--------|-------------------------|
| BRAF | KIAA1549-BRAF.K12B11 | Fusion | BRAF Gene Fusion |
| BRAF | KIAA1549-BRAF.K12B9.COSF1474 | Fusion | BRAF Gene Fusion |
| BRAF | KIAA1549-BRAF.K13B9 | Fusion | BRAF Gene Fusion |
| BRAF | KIAA1549-BRAF.K14B11.COSF1226 | Fusion | BRAF Gene Fusion |
| BRAF | KIAA1549-BRAF.K14B9.COSF483 | Fusion | BRAF Gene Fusion |
| BRAF | KIAA1549-BRAF.K15B10.COSF1283.1 | Fusion | BRAF Gene Fusion |
| BRAF | KIAA1549-BRAF.K15B11.COSF485.1 | Fusion | BRAF Gene Fusion |
| BRAF | KIAA1549-BRAF.K15B9.COSF481.1 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | KIAA1549-BRAF.K16B10 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | KIAA1549-BRAF.K17B10.COSF509 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | KIAA1549-BRAF.K18B9.COSF511 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | KIAA1549-BRAF.K9B9 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | KLHL7-BRAF.K5B9 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | LSM12-BRAF.L3B9 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | LSM14A-BRAF.L9B9 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | MACF1-BRAF.M60B9 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | MAD1L1-BRAF.M16B9 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | MAD1L1-BRAF.M17B10 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | MKRN1-BRAF.M4B11.COSF1444 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | MKRN1-BRAF.M4B9 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | MYRIP-BRAF.M16B9 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | MZT1-BRAF.M2B11 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | NUB1-BRAF.N3B9 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | NUDCD3-BRAF.N4B9 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | NUP214-BRAF.N21B10 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | PAPSS1-BRAF.P5B9.1 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | PLIN3-BRAF.P1B9 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | RAD18-BRAF.R7B10 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | RBMS3-BRAF.R11B11 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | RNF11-BRAF.R1B11 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | RNF130-BRAF.R3B9.COSF1483 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | RP2-BRAF.R3B10 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | SLC12A7-BRAF.S17B11 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | SLC45A3-BRAF.S1B8.COSF871 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | SND1-BRAF.S10B11 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | SND1-BRAF.S10B9 | Fusion | <b>BRAF Gene Fusion</b> |
| BRAF | SND1-BRAF.S11B11 | Fusion | BRAF Gene Fusion |
| BRAF | SND1-BRAF.S14B11 | Fusion | BRAF Gene Fusion |
| BRAF | SND1-BRAF.S14B9 | Fusion | BRAF Gene Fusion |
| BRAF | SND1-BRAF.S16B9.1 | Fusion | <b>BRAF Gene Fusion</b> |



| i . | | | |
|------|----------------------|--------|------------------|
| BRAF | SND1-BRAF.S18B10 | Fusion | BRAF Gene Fusion |
| BRAF | SND1-BRAF.S9B2 | Fusion | BRAF Gene Fusion |
| BRAF | SND1-BRAF.S9B9 | Fusion | BRAF Gene Fusion |
| BRAF | SOX6-BRAF.S5B9 | Fusion | BRAF Gene Fusion |
| BRAF | SOX6-BRAF.S6B9 | Fusion | BRAF Gene Fusion |
| BRAF | STRN3-BRAF.S3B10 | Fusion | BRAF Gene Fusion |
| BRAF | TANK-BRAF.T4B9 | Fusion | BRAF Gene Fusion |
| BRAF | TAX1BP1-BRAF.T8B11.1 | Fusion | BRAF Gene Fusion |
| BRAF | TMEM178B-BRAF.T2B9 | Fusion | BRAF Gene Fusion |
| BRAF | TMPRSS2-BRAF.T3B11 | Fusion | BRAF Gene Fusion |
| BRAF | TRIM24-BRAF.T10B9 | Fusion | BRAF Gene Fusion |
| BRAF | TRIM24-BRAF.T11B2 | Fusion | BRAF Gene Fusion |
| BRAF | TRIM24-BRAF.T3B10 | Fusion | BRAF Gene Fusion |
| BRAF | TRIM24-BRAF.T3B11 | Fusion | BRAF Gene Fusion |
| BRAF | TRIM24-BRAF.T5B8 | Fusion | BRAF Gene Fusion |
| BRAF | TRIM24-BRAF.T9B9.1 | Fusion | BRAF Gene Fusion |
| BRAF | TRIM4-BRAF.T6B10 | Fusion | BRAF Gene Fusion |
| BRAF | UBN2-BRAF.U3B11 | Fusion | BRAF Gene Fusion |
| BRAF | ZC3HAV1-BRAF.Z3B10 | Fusion | BRAF Gene Fusion |
| BRAF | ZC3HAV1-BRAF.Z7B11 | Fusion | BRAF Gene Fusion |
| BRAF | ZKSCAN5-BRAF.Z2B9 | Fusion | BRAF Gene Fusion |
| BRAF | ZSCAN30-BRAF.Z3B10 | Fusion | BRAF Gene Fusion |

| INCLUSION | VARIANTS | | | |
|-----------|-------------|---------|----------|-----|
| Hotspots | | | | |
| | | Variant | | |
| Gene Name | Variant ID | Туре | aMOI | LOE |
| MTOR | COSM51889 | SNV | p.L2220F | 3 |
| MTOR | COSM3965698 | SNV | p.L2216P | 3 |
| MTOR | MCH4 | SNV | p.R2217W | 3 |
| MTOR | COSM1560108 | SNV | p.S2215P | 3 |
| MTOR | COSM20417 | SNV | p.S2215Y | 3 |
| MTOR | COSM1686998 | SNV | p.S2215F | 3 |
| MTOR | COSM462592 | SNV | p.A2210P | 3 |
| MTOR | COSM414183 | SNV | p.L2209V | 3 |
| MTOR | COSM527403 | SNV | p.N2206S | 3 |
| MTOR | COSM893813 | SNV | p.F1888L | 3 |
| MTOR | COSM462604 | SNV | p.F1888L | 3 |
| MTOR | COSM3358968 | SNV | p.F1888I | 3 |



| MTOR | COSM3358967 | SNV | p.F1888L | 3 |
|--------|-------------|-----|----------|---|
| MTOR | PM_D142 | SNV | p.E1799K | 3 |
| MTOR | COSM180789 | SNV | p.E1799K | 3 |
| MTOR | OM9 | SNV | p.C1483W | 3 |
| MTOR | COSM462615 | SNV | p.C1483Y | 3 |
| MTOR | COSM462616 | SNV | p.C1483F | 3 |
| MTOR | COSM3747775 | SNV | p.C1483R | 3 |
| MTOR | COSM462618 | SNV | p.L1460P | 3 |
| MTOR | COSM462619 | SNV | p.A1459P | 3 |
| PIK3CA | COSM746 | SNV | p.R88Q | 2 |
| PIK3CA | COSM27493 | SNV | p.R93W | 3 |
| PIK3CA | COSM748 | SNV | p.G106V | 3 |
| PIK3CA | COSM13570 | SNV | p.K111E | 3 |
| PIK3CA | COSM751 | SNV | p.G118D | 3 |
| PIK3CA | COSM754 | SNV | p.N345K | 2 |
| PIK3CA | COSM757 | SNV | p.C420R | 3 |
| PIK3CA | COSM759 | SNV | p.P539R | 3 |
| PIK3CA | COSM760 | SNV | p.E542K | 3 |
| PIK3CA | COSM763 | SNV | p.E545K | 3 |
| PIK3CA | COSM764 | SNV | p.E545G | 3 |
| PIK3CA | COSM12458 | SNV | p.E545A | 3 |
| PIK3CA | COSM765 | SNV | p.E545D | 2 |
| PIK3CA | COSM766 | SNV | p.Q546K | 3 |
| PIK3CA | COSM767 | SNV | p.Q546P | 3 |
| PIK3CA | COSM12590 | SNV | p.T1025S | 3 |
| PIK3CA | COSM12591 | SNV | p.M1043V | 3 |
| PIK3CA | COSM773 | SNV | p.M1043I | 3 |
| PIK3CA | COSM94984 | SNV | p.M1043I | 3 |
| PIK3CA | COSM29313 | SNV | p.M1043I | 3 |
| PIK3CA | COSM774 | SNV | p.H1047Y | 3 |
| PIK3CA | COSM775 | SNV | p.H1047R | 2 |
| PIK3CA | COSM776 | SNV | p.H1047L | 3 |
| PTEN | COSM5133 | SNV | p.Y16C | 3 |
| PTEN | COSM5247 | SNV | p.Y27S | 3 |
| PTEN | COSM86058 | SNV | p.A34D | 3 |
| PTEN | OM1539 | SNV | p.N48K | 3 |
| PTEN | COSM5223 | SNV | p.M35R | 3 |
| PTEN | MCH13 | SNV | p.H61D | 3 |
| PTEN | COSM5042 | SNV | p.H61R | 3 |
| PTEN | COSM5036 | SNV | p.Y68H | 3 |



| PTEN | MCH14 | SNV | p.Y68D | 3 |
|------|------------|-----|---------|---|
| PTEN | COSM5102 | SNV | p.C71Y | 3 |
| PTEN | COSM23566 | SNV | p.D92H | 3 |
| PTEN | COSM5099 | SNV | p.D92G | 3 |
| PTEN | COSM5264 | SNV | p.D92A | 3 |
| PTEN | COSM5236 | SNV | p.D92V | 3 |
| PTEN | COSM35759 | SNV | p.D92E | 3 |
| PTEN | COSM125653 | SNV | p.D92E | 3 |
| PTEN | COSM5043 | SNV | p.H93Y | 3 |
| PTEN | COSM5283 | SNV | p.H93D | 3 |
| PTEN | COSM5265 | SNV | p.P96Q | 3 |
| PTEN | COSM5266 | SNV | p.C105F | 3 |
| PTEN | COSM5212 | SNV | p.D107Y | 3 |
| PTEN | COSM5106 | SNV | p.L112P | 3 |
| PTEN | MCH15 | SNV | p.L112R | 3 |
| PTEN | COSM5214 | SNV | p.A121P | 3 |
| PTEN | COSM5273 | SNV | p.A121E | 3 |
| PTEN | COSM5234 | SNV | p.l122S | 3 |
| PTEN | COSM921088 | SNV | p.H123D | 3 |
| PTEN | COSM921089 | SNV | p.C124R | 3 |
| PTEN | COSM5224 | SNV | p.C124S | 3 |
| PTEN | COSM5082 | SNV | p.K125E | 3 |
| PTEN | COSM5041 | SNV | p.A126V | 3 |
| PTEN | COSM5143 | SNV | p.G127E | 3 |
| PTEN | COSM246853 | SNV | p.G129R | 3 |
| PTEN | COSM28917 | SNV | p.G129E | 3 |
| PTEN | COSM5276 | SNV | p.G129V | 3 |
| PTEN | COSM5219 | SNV | p.R130G | 3 |
| PTEN | COSM5216 | SNV | p.R130L | 3 |
| PTEN | COSM5033 | SNV | p.R130Q | 3 |
| PTEN | COSM5104 | SNV | p.T131I | 3 |
| PTEN | COSM5044 | SNV | p.V133I | 3 |
| PTEN | COSM12734 | SNV | p.C136Y | 3 |
| PTEN | COSM5144 | SNV | p.Y155C | 3 |
| PTEN | COSM5091 | SNV | p.G165R | 3 |
| PTEN | COSM5114 | SNV | p.G165E | 3 |
| PTEN | COSM249877 | SNV | p.G165V | 3 |
| PTEN | MCH20 | SNV | p.S170R | 3 |
| PTEN | COSM5045 | SNV | p.S170N | 3 |



| | PTEN | MCH21 | SNV | p.S170R 3 | |
|---|--------|-----------|-----|--------------------|---|
| | PTEN | COSM5089 | SNV | p.R173C 3 | |
| | PTEN | COSM5039 | SNV | p.R173H 3 | |
| | PTEN | MCH16 | SNV | p.R173P 3 | |
| | PTEN | COSM5221 | SNV | p.Y174N 3 | |
| | PTEN | MCH17 | SNV | p.L181P 3 | |
| | PTEN | COSM5220 | SNV | p.G251C 3 | |
| | PTEN | COSM5255 | SNV | p.F341V 3 | |
| | PTEN | MCH18 | SNV | p.V343E 3 | |
| | PTEN | SM5213 | SNV | p.L345Q 3 | |
| i | | | | | ı |
| | PIK3R1 | PM_D147 | DEL | p.KS459delN | 3 |
| | PIK3R1 | PM_D150 | DEL | p.QY579_580H | 3 |
| | PIK3R1 | PM_D153 | DEL | p.QYL579L | 3 |
| | PIK3R1 | PM_D157 | DEL | p.DKRMNS560del | 3 |
| | PIK3R1 | PM_D158 | DEL | p.NSIKPDLIQL564del | 3 |
| | PIK3R1 | PM_D159 | SNV | p.N564D | 3 |
| | PIK3R1 | COSM35808 | SNV | p.N564DK | 3 |
| | PIK3R1 | COSM35765 | SNV | p.D560Y | 3 |

| IHC | RESULTS |
|-------|------------|
| GENE: | STATUS: |
| PTEN | NEGATIVE * |

<sup>\*</sup>Patients who have PTEN loss by IHC but a technical sequencing failure will be eligible for Cohort B of this sub-protocol.



#### APPENDIX VIII: TARGET HISTOLOGIES FOR APEC1621D EXPANSION COHORTS

Target tumor types considered for biomarker-positive expansion cohorts and biomarker-negative cohorts in the event of agent activity in a specific tumor type.

# **Tumor type**

- 1. Ependymoma
- 2. Ewing Sarcoma/Peripheral PNET
- 3. Hepatoblastoma
- 4. Glioma, high grade
- 5. Glioma, low grade
- 6. Langerhans Cell Histiocytosis
- 7. Malignant Germ Cell Tumor
- 8. Medulloblastoma
- 9. Neuroblastoma
- 10. Non-Hodgkin Lymphoma
- 11. Non-RMS Soft Tissue Sarcoma
- 12. Osteosarcoma
- 13. Rhabdoid Malignancy
- 14. Rhabdomyosarcoma
- 15. Wilms Tumor
- 16. Other Histology (based on COG/NCI-CTEP approval)



#### APPENDIX IX: YOUTH INFORMATION SHEETS

# INFORMATION SHEET REGARDING RESEARCH STUDY APEC1621D (for children from 7 through 13 years of age)

We want to tell you all about this study. You and your family can decide if you want to be in it. Ask questions if you don't understand.

- 1. What is the name of the study? A study of Molecular Analysis for Therapy Choice (MATCH) in children with a cancer that has come back after treatment or is difficult to treat
- 2. Who is in charge of the study? The study is being done by Children's Oncology Group and is being done at other hospitals.
- 3. What is the study about? We are asking you to take part in a research study because you have a cancer that has come back after treatment or is difficult to treat. A research study is when doctors work together to try out new ways to help people who are sick. In this study, we are trying to learn more about how to treat the kind of cancer that you have.
- 4. What will happen to me on the study? Children who are a part of this study will be given LY3023414 that could "match" your tumor. The doctors want to see if LY3023414 will help children with your type of cancer get better. We don't know if LY3023414 will work well to get rid of your cancer. That is why we are doing the study. You will have some tests and check-ups done more often than if you weren't part of this study. Some of these tests will require extra needle sticks for blood collection. We will follow your health after you finish the study treatment.

Sometimes good things can happen to people when they are in a research study. These good things are called "benefits." We hope that a benefit to you of being part of this study is that LY3023414 may cause your cancer to stop growing or to shrink for a period of time but we don't know for sure if there is any benefit of being part of this study.

Sometimes bad things can happen to people when they are in a research study. These bad things are called "risks." The risks to you from this study are that you may have problems, or side effects from LY3023414. Your doctor will talk to you about the risks we know about from LY3023414. Other things may happen to you that we don't yet know about.

- 5. Do I have to be in the study? You and Your family can choose to be part of this study or not. You and your family can also decide to stop being in this study at any time once you start. The doctors and nurses will still take care of you. There may be other treatments for your illness that your doctor can tell you about. If you have any questions or don't like what is happening, please tell your parent, the doctor or nurse.
- 6. We are asking your permission to collect additional blood. We want to see if there are ways to tell how the cancer will respond to treatment. You can still take part in this study even if you don't allow us to collect the extra blood samples for research.



# INFORMATION SHEET REGARDING RESEARCH STUDY APEC1621D (for teens from 14 through 17 years of age)

We want to tell you all about this study. You and your family can decide if you want to be in it. Ask questions if you don't understand.

- 1. What is the name of the study? A study of Molecular Analysis for Therapy Choice (MATCH) in children with a cancer that has come back after treatment or is difficult to treat
- 2. Who is in charge of the study? The study is being done by Children's Oncology Group and is being done at other hospitals.
- 3. What is the study about? We are asking you to take part in a research study because you have a cancer that has come back after treatment or is difficult to treat. A research study is when doctors work together to try out new ways to help people who are sick. In this study, we are trying to learn more about how to treat the kind of cancer that you have.
- 4. What will happen to me in the study? Children and teens who are part of this study will be given LY3023414 that could "match" your tumor. The doctors want to see if LY3023414 will help children with your type of cancer get better. We don't know if LY3023414 will work well to get rid of your cancer. That is why we are doing the study. You will have some tests and check-ups done more often than if you weren't part of this study. Some of these tests will require extra needle sticks for blood collection. We will collect information about your health after you finish the study treatment.

Sometimes good things can happen to people when they are in a research study. These good things are called "benefits." We hope that a benefit to you of being part of this study is that LY3023414 may cause your cancer to stop growing or to shrink for a period of time but we don't know for sure if there is any benefit of being part of this study.

Sometimes bad things can happen to people when they are in a research study. These bad things are called "risks." The risks to you from this study are that you may have side effects from LY3023414. Your doctor will talk to you about the risks we know about from LY3023414. Other things may happen to you that we don't yet know about.

- 5. Will I be paid to be in this study? You will not be paid for being in this study.
- 6. <u>Do I have to be in the study?</u> You and your family can choose to be part of this study or not. You and your family can also decide to stop being in this study at any time once you start. The doctors and nurses will still take care of you. There may be other treatments for your illness that your doctor can tell you about. If you have any questions or don't like what is happening, tell your parent, the doctor or nurse.
- 7. We are asking your permission to collect additional blood. We want to see if there are ways to tell how the cancer will respond to treatment. You can still take part in this study even if you don't allow us to collect the extra blood samples for research.



#### APPENDIX X: CTEP AND CTSU REGISTRATION PROCEDURES

Food and Drug Administration (FDA) regulations and National Cancer Institute (NCI) policy require all individuals contributing to NCI-sponsored trials to register and to renew their registration annually. To register, all individuals must obtain a Cancer Therapy Evaluation Program (CTEP) Identity and Access Management (IAM) account at <a href="https://ctepcore.nci.nih.gov/iam">https://ctepcore.nci.nih.gov/iam</a>. In addition, persons with a registration type of Investigator (IVR), Non-Physician Investigator (NPIVR), or Associate Plus (AP) must complete their annual registration using CTEP's web-based Registration and Credential Repository (RCR) at <a href="https://ctepcore.nci.nih.gov/rcr">https://ctepcore.nci.nih.gov/rcr</a>.

RCR utilizes five person registration types.

- IVR MD, DO, or international equivalent;
- NPIVR advanced practice providers (e.g., NP or PA) or graduate level researchers (e.g., PhD);
- AP clinical site staff (e.g., RN or CRA) with data entry access to CTSU applications such as the Roster Update Management System (RUMS), OPEN, Rave, acting as a primary site contact, or with consenting privileges;
- Associate (A) other clinical site staff involved in the conduct of NCI-sponsored trials; and
- Associate Basic (AB) individuals (e.g., pharmaceutical company employees) with limited access to NCI-supported systems.

RCR requires the following registration documents:

| <b>Documentation Required</b> | IVR | NPIVR | AP | A | AB |
|---|---|---|---|---|---|
| FDA Form 1572 | <b>✓</b> | <b>√</b> | | | |
| Financial Disclosure Form | ✓ | ✓ | ✓ | | |
| NCI Biosketch (education, training, employment, license, and certification) | <b>√</b> | ✓ | <b>√</b> | | |
| GCP training | ✓ | <b>✓</b> | ✓ | | |
| Agent Shipment Form (if applicable) | <b>√</b> | | | | |
| CV (optional) | <b>✓</b> | ✓ | ✓ | | |

An active CTEP-IAM user account and appropriate RCR registration is required to access all CTEP and Cancer Trials Support Unit (CTSU) websites and applications. In addition, IVRs and NPIVRs must list all clinical practice sites and Institutional Review Boards (IRBs) covering their practice sites on the FDA Form 1572 in RCR to allow the following:

- Addition to a site roster;
- Assign the treating, credit, consenting, or drug shipment (IVR only) tasks in OPEN;
- Act as the site-protocol Principal Investigator (PI) on the IRB approval; and
- Assign the Clinical Investigator (CI) role on the Delegation of Tasks Log (DTL).



In addition, all investigators acting as the Site-Protocol PI (investigator listed on the IRB approval), consenting/treating/drug shipment investigator in OPEN, or as the CI on the DTL must be rostered at the enrolling site with a participating organization.

Additional information is located on the CTEP website at <a href="https://ctep.cancer.gov/investigatorResources/default.htm">https://ctep.cancer.gov/investigatorResources/default.htm</a>. For questions, please contact the RCR <a href="https://ctep.cancer.gov/investigatorResources/default.htm">https://ctep.cancer.gov/investigatorResources/default.htm</a>. For questions, please contact the RCR <a href="https://ctep.cancer.gov/investigatorResources/default.htm">https://ctep.cancer.gov/investigatorResources/default.htm</a>. For questions, please contact the RCR <a href="https://ctep.cancer.gov/investigatorResources/default.htm">https://ctep.cancer.gov/investigatorResources/default.htm</a>. For questions, please contact the RCR <a href="https://ctep.cancer.gov/investigatorResources/default.htm">https://ctep.cancer.gov/investigatorResources/default.htm</a>. For questions, please contact the RCR <a href="https://ctep.cancer.gov/investigatorResources/default.htm">https://ctep.cancer.gov/investigatorResources/default.htm</a>.

#### CTSU REGISTRATION PROCEDURES

This study is supported by the NCI Cancer Trials Support Unit (CTSU).

#### **Protocol-Specific Requirements For Site Registration:**

• IRB approval (For sites not participating via the NCI CIRB; local IRB documentation, an IRB-signed CTSU IRB Certification Form, Protocol of Human Subjects Assurance Identification/IRB Certification/Declaration of Exemption Form, or combination is accepted)

### **Submitting Regulatory Documents:**

Submit required forms and documents to the CTSU Regulatory Office using the Regulatory Submission Portal on the CTSU website.

To access the Regulatory Submission Portal log in to the CTSU members' website, go to the Regulatory section and select Regulatory Submission.

Institutions with patients waiting that are unable to use the Regulatory Submission Portal should alert the CTSU Regulatory Office immediately at 1-866-651-2878 in order to receive further instruction and support.

#### **Checking Your Site's Registration Status**

Site registration status may be verified on the CTSU members' website.

- Click on Regulatory at the top of the screen;
- Click on Site Registration; and
- Enter the site's 5-character CTEP Institution Code and click on Go.
  - o Additional filters are available to sort by Protocol, Registration Status, Protocol Status, and/or IRB Type.

Note: The status shown only reflects institutional compliance with site registration requirements as outlined within the protocol. It does not reflect compliance with protocol requirements for individuals participating on the protocol or the enrolling investigator's status with NCI or their affiliated networks.

### **Data Submission / Data Reporting**

Medidata Rave is a clinical data management system being used for data collection for this trial/study. Access to the trial in Rave is controlled through the CTEP-IAM system and role assignments.

Requirements to access Rave via iMedidata:



- A valid CTEP-IAM account: and
- Assigned a Rave role on the LPO or PO roster at the enrolling site of: Rave CRA, Rave Read Only, Rave CRA (LabAdmin), Rave SLA, or Rave Investigator.

# Rave role requirements:

- Rave CRA or Rave CRA (Lab Admin) role must have a minimum of an Associate Plus (AP) registration type;
- Rave Investigator role must be registered as an Non-Physician Investigator (NPIVR) or Investigator (IVR); and
- o Rave Read Only role must have at a minimum an Associates (A) registration type.

Refer to <a href="https://ctep.cancer.gov/investigatorResources/default.htm">https://ctep.cancer.gov/investigatorResources/default.htm</a> for registration types and documentation required.

Upon initial site registration approval for the study in Regulatory Support System (RSS), all persons with Rave roles assigned on the appropriate roster will be sent a study invitation e-mail from iMedidata. To accept the invitation, site staff must log in to the Select Login (https://login.imedidata.com/selectlogin) using their CTEP-IAM username and password and click on the *accept* link in the upper right-corner of the iMedidata page. Site staff will not be able to access the study in Rave until all required Medidata and study specific trainings are completed. Trainings will be in the form of electronic learnings (eLearnings) and can be accessed by clicking on the link in the upper right pane of the iMedidata screen. If an eLearning is required and has not yet been taken, the link to the eLearning will appear under the study name in iMedidata instead of the *Rave EDC* link; once the successful completion of the eLearning has been recorded, access to the study in Rave will be granted, and a *Rave EDC* link will display under the study name.

Site staff that have not previously activated their iMedidata/Rave account at the time of initial site registration approval for the study in RSS will receive a separate invitation from iMedidata to activate their account. Account activation instructions are located on the CTSU website in the Data Management section under the Rave resource materials (Medidata Account Activation and Study Invitation Acceptance). Additional information on iMedidata/Rave is available on the CTSU members' website in the Data Management > Rave section at <a href="www.ctsu.org/RAVE/">www.ctsu.org/RAVE/</a> or by contacting the CTSU Help Desk at 1-888-823-5923 or by e-mail at <a href="test-account-action-contact-account-action-contact-account-accou

#### **Data Quality Portal**

The Data Quality Portal (DQP) provides a central location for site staff to manage unanswered queries and form delinquencies, monitor data quality and timeliness, generate reports, and review metrics.

The DQP is located on the CTSU members' website under Data Management. The Rave Home section displays a table providing summary counts of Total Delinquencies and Total Queries. DQP Queries, DQP Delinquent Forms and the DQP Reports modules are available to access details and reports of unanswered queries, delinquent forms, and timeliness reports. Review the DQP modules on a regular basis to manage specified queries and delinquent forms.

The DQP is accessible by site staff that are rostered to a site and have access to the CTSU website. Staff that have Rave study access can access the Rave study data using a direct link on the DQP.

To learn more about DQP use and access, click on the Help icon displayed on the Rave Home, DQP Queries, and DQP Delinquent Forms modules.



Note: Some Rave protocols may not have delinquent form details or reports specified on the DQP. A protocol must have the Calendar functionality implemented in Rave by the Lead Protocol Organization for delinquent form details and reports to be available on the DQP. Site staff should contact the LPO Data Manager for their protocol regarding questions about Rave Calendaring functionality.



# APPENDIX XI: TOXICITY-SPECIFIC GRADING

# Bilirubin

| Grade 1: | $\leq$ 1.5 x ULN |
|----------|--------------------|
| Grade 2: | > 1.5 x - 3 x ULN |
| Grade 3: | > 3 x - 10 x ULN |
| Grade 4: | > 10 x ULN |

ALT: For the purpose of this study, the ULN for SGPT is 45 U/L regardless of baseline.

| Grade 1: | ≤ 135 |
|----------|----------|
| Grade 2: | 136- 225 |
| Grade 3: | 226- 900 |
| Grade 4: | > 900 |

AST: For the purpose of this study, the ULN for SGPT is 50 U/L regardless of baseline.

| Grade 1: | ≤ 150 |
|----------|----------|
| Grade 2: | 151-250 |
| Grade 3: | 251-1000 |
| Grade 4: | > 1000 |

# GGT:

| Grade 1: | > ULN- 2.5 x ULN |
|----------|----------------------|
| Grade 2: | > 2.5 x ULN- 5 x ULN |
| Grade 3: | > 5 x ULN-20 x ULN |
| Grade 4: | > 20 x ULN |